Sponsor: APGD EUCT 2024-511648-16-00: EudraCT number 2018-000519-26


A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus CAPOX Compared with Placebo Plus CAPOX as First-line Treatment of Subjects with Claudin (CLDN) 18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma

## **GLOW**

# ISN/Protocol 8951-CL-0302 Version 8.0

# **Incorporating Substantial Amendment 7**

06 Dec 2024

IND 129598

EUCT 2024-511648-16-00

EudraCT 2018-000519-26

Sponsor:

## Astellas Pharma Global Development, Inc. (APGD)

Northbrook, IL 60062

## Protocol History

Version 1.0 [26 Apr 2018]

Version 2.0 [29 Jun 2018] Incorporating Substantial Amendment 1

Version 3.0 [06 Aug 2019] Incorporating Substantial Amendment 2

Version 3.1 [06 Jan 2021] Incorporating Nonsubstantial Amendment 1

Version 4.0 [29 Aug 2019] Incorporating Country-specific Substantial Amendment 3 for China

Version 4.1 [11 Jan 2021] Incorporating Country-specific Nonsubstantial Amendment 2 for China

Version 5.0 [18 Oct 2021] Incorporating Substantial Amendment 4

Version 6.0 [CN] [18 Oct 2021] Incorporating Country-specific Substantial Amendment 5 for China

Version 6.1 [JP] [04 Oct 2023] Incorporating Country-specific Nonsubstantial Amendment 3 for Japan

Version 7.0 [04 Mar 2024] Incorporating Substantial Amendment 6

The information contained in this document is supplied as a background for clinical investigations. This document contains confidential information which is the intellectual property of Astellas. By accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others or use it for unauthorized purposes except (1) as otherwise agreed to in writing; (2) where required by applicable law; (3) where disclosure is directly related to the care and safety of the research participant; and (4) where disclosure of such information is made to a member of the investigator's team who agrees to hold this information in confidence.


## **Table of Contents**

| I. | | SIG | NATURES | 9 |
|---|---|---|---|---|
| II. | • | CO | NTACT DETAILS OF KEY SPONSOR'S PERSONNEL | 12 |
| III. | | LIS | T OF ABBREVIATIONS AND DEFINITION OF KEY TERMS | 13 |
| IV | 7. | PRO | PROTOCOL AMENDMENT SUMMARY OF CHANGES 18 | |
| V. | | SYN | NOPSIS | 20 |
| V] | [ <b>.</b> | FLO | OW CHART, STUDY SCHEMATICS AND SCHEDULE OF | |
| | | | | 36 |
| 1 | | INT | TRODUCTION | <b>48</b> |
| | 1.1 | | Background ····· | 49 |
| | 1.2 | | Nonclinical and Clinical Data | 50 |
| | 1 | .2.1 | Nonclinical Data······ | 50 |
| | 1 | .2.2 | Clinical Data ····· | 51 |
| | 1.3 | | Summary of Key Safety Information for Study Drugs ···································· | 52 |
| | 1.4 | | Efficacy | 53 |
| | 1 | .4.1 | Efficacy Results from Study GM-IMAB-001-02 (MONO) | 53 |
| | 1 | .4.2 | Efficacy Results from Study GM-IMAB-001-03 (FAST)······ | 53 |
| | 1 | .4.3 | Efficacy of CAPOX ···································· | 54 |
| | 1.5 | | Risk Benefit Assessment | 54 |
| 2 | | STU | JDY OBJECTIVE(S), DESIGN AND ENDPOINTS | 55 |
| | 2.1 | | Study Objective(s) ······ | 55 |
| | 2 | 2.1.1 | Primary Objectives ····· | 55 |
| | 2 | 2.1.2 | Secondary Objectives ···································· | 55 |
| | 2 | 2.1.3 | Exploratory Objectives ······· | 56 |
| | 2.2 | | Study Design and Dose Rationale | 56 |
| | 2 | 2.2.1 | , , | 56 |
| | 2 | 2.2.2 | | 60 |
| | 2.3 | | Endpoints | 61 |
| | 2 | 2.3.1 | | 61 |
| | 2 | 2.3.2 | Secondary Endpoints | 61 |
| | 2 | 2.3.3 | | 62 |
| 3 | | STU | | <b>62</b> |
| | 3.1 | | Selection of Study Population · | 62 |

| | 3.2 | Inclusion Criteria | 62 |
|---|---|---|---|
| | 3.3 | Exclusion Criteria ····· | 64 |
| 4 | IDE | NTIFICATION OF STUDY TREATMENT(S) | 66 |
| | 4.1 | Zolbetuximab (Investigational Product)······ | 66 |
| | 4.2 | 0.9% Sodium Chloride Injection ······ | 67 |
| | 4.3 | Comparative Drug (Placebo) | 67 |
| | 4.4 | CAPOX (Backbone Treatment) | 67 |
| | 4.5 | Other Drug(s) ······ | 68 |
| | 4.5.1 | Antiemetic Premedication ······ | 68 |
| | 4.6 | Study Drug Handling | 68 |
| | 4.7 | Blinding | 69 |
| | 4.7.1 | Blinding Method····· | 69 |
| | 4.7.2 | Confirmation of the Indistinguishability of the Study Drugs | 69 |
| | 4.7.3 | Retention of the Assignment Schedule and Procedures for Treatment Code | |
| | | Breaking ····· | 69 |
| | 4.7.4 | Breaking the Treatment Code for Emergency | |
| | 4.7.5 | Breaking the Treatment Code by the Sponsor | 70 |
| | 4.8 | Assignment and Allocation ······ | • 70 |
| 5 | TRI | EATMENTS AND EVALUATION | <b>70</b> |
| | 5.1 | Dosing and Administration of Study Drug(s) and Other Medication(s) ······ | 70 |
| | 5.1.1 | Dose/Dose Regimen and Administration Period ······ ···· | · 70 |
| | 5.1 | .1.1 Zolbetuximab/Placebo ······ | 70 |
| | 5.1 | .1.2 Antiemetics | 71 |
| | 5.1 | 1.1.3 CAPOX | 72 |
| | 5.1.2 | Study Treatment Dose Modifications, Delays And Interruptions | 72 |
| | 5.1 | .2.1 Increase or Reduction of zolbetuximab/Placebo ····· | 72 |
| | 5.1 | .2.2 Zolbetuximab/Placebo Interruption or Permanent Discontinuation | 72 |
| | 5.1 | .2.3 Guidelines for Infusion-related Reactions for Zolbetuximab/Placebo ······ | 76 |
| | 5.1 | .2.4 CAPOX Dose Modification | 77 |
| | 5.1 | .2.5 CAPOX: Dose Modifications for Hematologic Toxicity | <del>7</del> 9 |
| | 5.1 | .2.6 CAPOX: Dose Modification for Non-hematologic Toxicity | 81 |
| | 5.1 | .2.7 Guidelines for Infusion-related Reactions for Oxaliplatin | 83 |
| | 5.1 | .2.8 Oxaliplatin-induced Neurotoxicity | 83 |
| | | .2.9 Oxaliplatin-induced Laryngopharyngeal Dysesthesia | 84 |
| 06 | Dec 2024 | Astellas Page 3 | of? |

| 5.1.2.1 | O Allergic Reaction to Oxaliplatin | 85 |
|---|---|---|
| 5.1.2.1 | 1 Extravasation of Oxaliplatin | 86 |
| 5.1.3 | Treatment Compliance · | · 86 |
| 5.1.4 | Criteria for Continuation of Treatment | 86 |
| 5.1.4.1 | \ | |
| | Zolbetuximab/Placebo ······ | 86 |
| 5.1.4.2 | | |
| | CAPOX (One or Both Components) | 87 |
| 5.1.4.3 | If Both Zolbetuximab/Placebo and CAPOX (Both Components) are Discontinued | 87 |
| 5.1.5 | Previous and Concomitant Treatment (Medication and Non-Medication | |
| | Therapy) ····· | 87 |
| 5.2 Der | mographics and Baseline Characteristics | 89 |
| 5.2.1 | Demographics | 89 |
| 5.2.2 | Medical History | 89 |
| 5.2.3 | Diagnosis of the Target Disease, Severity, and Duration of Disease | 89 |
| 5.3 Effi | cacy Assessments | 89 |
| 5.4 Safe | ety Assessment ······ | 90 |
| 5.4.1 | Vital Signs····· | 90 |
| 5.4.2 | Observation Period Following Zolbetuximab/Placebo Infusion ······ | 90 |
| 5.4.3 | Laboratory Assessments | 90 |
| 5.4.4 | Physical Examination ······ | 93 |
| 5.4.5 | Electrocardiogram | 93 |
| 5.4.6 | Performance Status | 93 |
| 5.5 Adv | verse Events and Other Safety Aspects ······ | 93 |
| 5.5.1 | Definition of Adverse Events | 94 |
| 5.5.1.1 | Abnormal Laboratory Findings ······· | 94 |
| 5.5.1.2 | Potential Cases of Drug-Induced Liver Injury | .94 |
| 5.5.1.3 | | 95 |
| 5.5.2 | Definition of Serious Adverse Events····· | 95 |
| 5.5.2.1 | Important Medical Events | 96 |
| 5.5.3 | Criteria for Causal Relationship to Study Treatment | 96 |
| 5.5.4 | Criteria for Defining the Severity of an Adverse Event | 97 |
| 5.5.5 | Reporting of Serious Adverse Events | 97 |
| 5.5.6 | Follow-up of Adverse Events ····· | 99 |
| 5.5.7 | Monitoring of Common Serious Adverse Events | 100 |
| Dec 2024 | | of 175 |

| 5.5.8 | Adverse Events of Special Interest | 100 |
|---|---|---|
| 5.5.9 | Special Situations | 100 |
| 5.5.9.1 | Pregnancy | 101 |
| 5.5.9.2 | Medication Error, Overdose and "Off-Label Use" | 101 |
| 5.5.9.3 | | 102 |
| 5.5.9.4 | 1 1 | 102 |
| 5.5.9.5 | Suspected Drug-Drug Interaction | 102 |
| 5.5.10 | Supply of New Information Affecting the Conduct of the Study | 102 |
| 5.5.11 | Urgent Safety Measures ····· | 103 |
| 5.5.12 | Reporting Urgent Safety Measures | 103 |
| 5.6 Tes | t Drug Concentration | 104 |
| 5.7 Oth | er Measurements, Assessments or Methods ······ | 104 |
| 5.7.1 | Biomarkers ····· | 104 |
| 5.7.2 | Blood, Serum and Plasma Samples | 104 |
| 5.7.3 | Tumor Tissue Samples | 105 |
| 5.7.4 | Immunogenicity Assessment (Anti-drug Antibody) ······ | 106 |
| 5.7.5 | Optional Samples for Banked Pharmacogenomics Sample Analysis ········ | 106 |
| 5.7.6 | Electronic Clinical Outcome Assessments | 107 |
| 5.7.6.1 | Quality of Life Questionnaire C30 ······ | 107 |
| 5.7.6.2 | Oesophago-Gastric Module 25 plus STO22 Belching Subscale ········ 1 | |
| 5.7.6.3 | Global Pain ····· | 108 |
| 5.7.6.4 | EuroQOL Five Dimensions Questionnaire ···································· | 108 |
| 5.7.6.5 | Health Resource Utilization ······ | 108 |
| 5.8 Tot | al Amount of Blood··································· | 108 |
| DISCO | NTINUATION | 108 |
| 6.1 Dis | continuation of Individual Subject(s) From Study Treatment | 108 |
| 6.1.1 | Lost to Follow Up ······ | 110 |
| 6.2 Dis | continuation of the Site · | 110 |
| 6.3 Dis | continuation of the Study | 110 |
| STATIS | STICAL METHODOLOGY | 111 |
| 7.1 San | nple Size······ | 111 |
| | alysis Sets······ | 111 |
| 7.2.1 | Full Analysis Set ······ | 111 |
| 7.2.2 | | 112 |

6

7

| 7.2.3 | Pharmacokinetic Analysis Set (PKAS) ······· | 112 |
|---|---|---|
| 7.3 De | emographics and Baseline Characteristics | 112 |
| 7.3.1 | Subject Disposition | 112 |
| 7.3.2 | Previous and Concomitant Medications | 112 |
| 7.3.3 | Medical History | 112 |
| 7.4 Ar | nalysis of Efficacy ······· | 112 |
| 7.4.1 | Analysis of Primary Endpoint | 112 |
| 7.4.1. | 1 Primary Analysis ······ | 112 |
| 7.4.1. | 2 Sensitivity Analysis ······ | 113 |
| 7.4.1. | | 113 |
| 7.4.2 | Analysis of Secondary Endpoints | 113 |
| 7.4.2. | | 113 |
| 7.4.2. | | 114 |
| 7.4.2. | 3 1 | 115 |
| 7.4.2. | 1 | 115 |
| 7.4.2. | | 115 |
| 7.4.3 | Analysis of Exploratory Endpoints | 115 |
| 7.4.3. | 1 Time to Progression ····· | 115 |
| 7.4.3. | | 115 |
| 7.4.3. | | 116 |
| 7.4.3. | | 116 |
| 7.4.3. | | 116 |
| 7.5 Ar | nalysis of Safety | 116 |
| 7.5.1 | Adverse Events ····· | 116 |
| 7.5.2 | Laboratory Assessments ····· | 117 |
| 7.5.3 | Vital Signs······ | 117 |
| 7.5.4 | Routine 12-lead Electrocardiograms ······ | 117 |
| 7.5.5 | Eastern Cooperative Oncology Group Performance Status | 117 |
| 7.6 Ar | nalysis of Pharmacokinetics | 117 |
| 7.6.1 | | 117 |
| 7.6.2 | Immunogenicity ···································· | 117 |
| 7.7 M | ajor Protocol Deviations and Other Analyses ······ | 118 |
| 7.8 Int | terim Analysis (and Early Discontinuation of the Clinical Study)······ | 118 |
| 7.9 Ha | andling of Missing Data, Outliers, Visit Windows, and Other Information | 118 |
| OPER | ATIONAL CONSIDERATIONS | <b>119</b> |

8

| | 8.1 Pro | ocedure for Clinical Study Quality Control | 119 |
|---|---|---|---|
| | 8.1.1 | Data Collection ····· | 119 |
| | 8.1.1.1 | Collection of Data Via Electronic Source | 119 |
| | 8.1.1.2 | Electronic Clinical Outcomes Assessment ···································· | 120 |
| | 8.2 Ma | jor Protocol Deviations ···································· | 120 |
| 9 | END O | F TRIAL | 121 |
| 10 | STUDY | ORGANIZATION | 121 |
| | 10.1 Ind | ependent Data Monitoring Committee | 121 |
| | 10.2 Oth | ner Study Organization ···································· | 121 |
| 11 | REFER | RENCES | 122 |
| 12 | APPEN | DICES | 125 |
| | 12.1 Eth | nical, Regulatory, and Study Oversight Considerations | 125 |
| | 12.1.1 | Ethical Conduct of the Study | 125 |
| | 12.1.2 | Institutional Review Board (IRB)/Independent Ethics Committee | |
| | | (IEC)/Competent Authorities (CA) ···································· | 125 |
| | 12.1.3 | Protocol Amendment and/or Revision ······ | 125 |
| | 12.1.4 | Informed Consent of Subjects ······ | 126 |
| | 12.1.4 | .1 Subject Information and Consent ······ | 126 |
| | 12.1.4 | | |
| | | Consent and Revision of the Written Information | 126 |
| | 12.1.5 | | 127 |
| | 12.1.6 | Record Retention | 127 |
| | 12.1.7 | Subject Confidentiality and Privacy | 128 |
| | 12.1.8 | Arrangement for Use of Information and Publication of the Clinical Study $\cdots$ | 128 |
| | 12.1.9 | Insurance of Subjects and Others (UNIQUE TO JAPAN REGION/STUDIES ENROLLING SUBJECTS IN EU) | 129 |
| | 12.1.10 | Signatory Investigator for Clinical Study Report | 129 |
| | 12.2 Pro | ocedures for Clinical Study Quality Control | 130 |
| | 12.2.1 | Clinical Study Monitoring | 130 |
| | 12.2.2 | Direct Access to Source Data/Documents | 130 |
| | 12.2.3 | Data Management ······ | 130 |
| | 12.2.4 | QUALITY ASSURANCE | 130 |
| | 12.3 Con | ntraception Requirements | 132 |
| | | ncomitant Medication Restrictions or Requirements | 134 |

| - | _ | | | | | | | | | |
|------------|---|----|----|---|---|----|----|---|----|---|
| <br>$\sim$ | 7 | NΠ | El | Т | 1 | E. | NΓ | Г | ſΑ | T |

| 12.5 | Liver Safety Monitoring and Assessment ······ | 136 |
|---|---|---|
| 12.6 | Common Serious Adverse Events····· | 139 |
| 12.7 | Pharmacogenomic Analysis with Banked Sample | 140 |
| 12.8 | Eastern Cooperative Oncology Group Performance Status Scale | 142 |
| 12.9 | Clinical Study Continuity ···································· | 143 |
| 12.10 | Unblinding Procedures Following Final Overall Survival Database Lock | 145 |
| LA | OTOCOL VERSION 7.0 (SUBSTANTIAL AMENDMENT 6) AND TER: FLOW CHART AND SCHEDULE OF ASSESSMENTS | 161<br>174 |
| | | 174<br>175 |
| 15 SPC | UNSUR'S SIGNATURES | 1/3 |
| | List of In-text Tables | |
| Table 1 | Up Through Protocol 6.1 (Original Protocol Version 1 Through 6.1): Schedule of Assessments | 40 |
| Table 2 | Guidelines for Zolbetuximab/Placebo Treatment Modification Due to Non-hematologic Toxicity | |
| Table 3 | Guidelines for Zolbetuximab/Placebo Treatment Modification Due to Hematologic Toxicity | |
| Table 4 | | 77 |
| Table 5 | Recommended Dose Adjustment Levels for Oxaliplatin and Capecitabine | 78 |
| Table 6 | CAPOX Dose Modification Due to Hematologic Toxicity | 79 |
| Table 7 | CAPOX Dose Modification Due to Non-hematologic Toxicity······ | 82 |
| Table 8 | Oxaliplatin Dose Modification for Associated Neurotoxicity | 84 |
| Table 9 | Comparison of the Symptoms and Treatment of Laryngopharyngeal Dysesthesia and Platinum Hypersensitivity Reactions | 85 |
| Table 10 | Up Through Protocol Version 6.1 or Earlier (Original Protocol Version 1 through 6.1): Alternative Schedule of Assessments in Response to a Crisis | 146 |
| Table 11 | Protocol Version 7.0 (Substantial Amendment 6) and Later: Schedule of Assessments | 162 |
| Table 12 | Protocol Version 7.0 (Substantial Amendment 6) and Later: Alternate Schedule of Assessments in Response to a Crisis | 167 |

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


## I. SIGNATURES

## 1. SPONSOR'S SIGNATURES

Required signatures (e.g., Protocol authors and contributors, etc.) are located in [Section 15 Sponsor's Signatures].

**Sponsor: APGD** EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


## 2. COORDINATING INVESTIGATOR'S SIGNATURE

The Coordinating Investigator's signature can be found in [Section 14 Coordinating Investigator's Signature]; located at the end of this document.

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

## 3. INVESTIGATOR'S SIGNATURE

A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus CAPOX Compared with Placebo Plus CAPOX as First-line Treatment of Subjects with Claudin (CLDN)18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma

ISN/Protocol 8951-CL-0302

**Version 8.0 Incorporating Substantial Amendment 7** 

06 Dec 2024

I have read all pages of this clinical study protocol for which Astellas is the sponsor. I agree to conduct the study as outlined in the protocol and to comply with all the terms and conditions set out therein. I confirm that I will conduct the study in accordance with International Council for Harmonisation (ICH) Good Clinical Practice (GCP) guidelines and applicable local regulations. I will also ensure that subinvestigator(s) and other relevant members of my staff have access to copies of this protocol and the ICH GCP guidelines to enable them to work in accordance with the provisions of these documents.

| Principal Investigator: | |
|-------------------------|--------------------|
| Signature: | Date (DD Mmm YYYY) |
| Printed Name: | |
| Address: | |


## II. CONTACT DETAILS OF KEY SPONSOR'S PERSONNEL

| 24h-Contact for Serious<br>Adverse Events (SAEs) | Please fax or email the SAE Worksheet to: Astellas Pharma Global Development, Inc. Global Pharmacovigilance |
|---|---|
| See [Section 5.5.5] Reporting of Serious Adverse Events] for SAE | North America Fax number: +1-888-396-3750<br>North America Alternate Fax number: +1-847-317-1241 |
| Fax Number and Email | International Fax Number: +44-800-471-5263<br>Email: safety-us@us.astellas.com |
| | Japan investigational sites: PAREXEL International Global Monitoring Operations Fax: 03-6888-5798 |
| Medical Monitor/Study<br>Physician: | Astellas Pharma China 27th Floor, Beijing IFC Tower, NO.8 Jianguomenwai Avenue, Chaoyang District, Beijing 100022, P.R.C. PPD PPD |


## III. LIST OF ABBREVIATIONS AND DEFINITION OF KEY TERMS

## **List of Abbreviations**

| Abbreviations | Description of abbreviations |
|---------------|------------------------------------------------------------|
| 5-FU | fluorouracil |
| ADA | anti-drug antibody |
| ADCC | antibody-dependent cellular cytotoxicity |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| APEBV | Astellas Pharma Europe B.V. |
| AST | aspartate aminotransferase |
| βhCG | beta human chorionic gonadotropin |
| C1D1 | Cycle 1 Day 1 |
| CA | Competent Authorities |
| CAPOX | capecitabine and oxaliplatin |
| CDC | complement-dependent cytotoxicity |
| CE | Conformité Européenne |
| CI | confidence interval |
| CLDN | claudin |
| СМН | Cochran-Mantel-Haenszel |
| CR | complete response |
| CRO | contract research organization |
| CT | computerized tomography |
| CTCAE | Common Terminology Criteria For Adverse Events |
| DCR | disease control rate |
| DOR | duration of response |
| DPD | dihydropyrimidine dehydrogenase |
| ECG | electrocardiogram |
| ECL | electrochemiluminescense |
| eCOA | Electronic Clinical Outcomes Assessment |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EEA | European Economic Area |
| EORTC | European Organization for Research and Treatment of Cancer |
| EOX | epirubicin, oxaliplatin and capecitabine |
| EQ5D-5L | EuroQOL Five Dimensions Questionnaire 5L |

| Abbreviations | Description of abbreviations |
|---|---|
| EU | European Union |
| FAS full analysis set | |
| FIM | first-in-human |
| FFPE | formalin-fixed paraffin embedded |
| GCP | Good Clinical Practices |
| GE | gastroesophageal |
| GEJ | gastroesophageal junction |
| GHS/QoL | Global Health Status/Quality of Life |
| GMP | Good Manufacturing Practices |
| GP | Global Pain |
| Hgb | hemoglobin |
| HEOR | health economics and outcomes research |
| HER2 | human epidermal growth factor receptor 2 |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HRQoL | health-related quality of life |
| HRU | Health Resource Utilization |
| HSR | hypersensitivity reactions |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| IDMC | independent data monitoring committee |
| IEC | independent ethics committee |
| IND | investigational new drug |
| IHC | immunohistochemistry |
| IMAB | ideal monoclonal antibody |
| INR | international normalized ratio |
| IRB | institutional review board |
| IRC | independent review committee |
| IRR | infusion-related reaction |
| IRT | interactive response technology |
| ISN | international study number |
| LA-CRF | liver abnormality case report form |
| LFT | liver function tests |
| mAbs | monoclonal antibodies |
| МСН | Mean Corpuscular Hemoglobin |

| Abbreviations | Description of abbreviations |
|---|---|
| MRI | magnetic resonance imaging |
| NCCN | National Comprehensive Cancer Network |
| NCI | National Cancer Institute |
| NSAID | nonsteroidal anti-inflammatory drugs |
| OG25-Pain | oesophago-gastric questionnaire (OG25) on abdominal pain and discomfort |
| ORR | objective response rate |
| OS | overall survival |
| PD | progressive disease |
| PF | physical function |
| PFS | progression free survival |
| PFS2 | progression free survival following subsequent anticancer treatment |
| PGx | pharmacogenomics |
| PKAS | pharmacokinetic analysis set |
| PR | partial response |
| PRES | posterior reversible encephalopathy syndrome |
| PT | preferred term |
| QLQ-C30 | Quality of Life Questionnaire - Core Questionnaire |
| QLQ-OG25 | Quality of Life Questionnaire - Oesophago-Gastric Module 25 |
| QTc | QT corrected |
| RBC | red blood cell |
| RECIST | Response Evaluation Criteria In Solid Tumors |
| RSI | reference safety information |
| (S)AE | serious adverse event and/or adverse event |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SD | stable disease |
| SOP | standard operating procedure |
| SPC | summary of product characteristics |
| SUSAR | suspected unexpected serious adverse reactions |
| T4 | thyroxine |
| TEAE | treatment-emergent adverse event |
| TSH | thyroid stimulating hormone |
| TTCD | time to confirmed deterioration |
| TTP | time to progression |
| ULN | upper limit of normal |
| USM | urgent safety measure |

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


| Abbreviations | Description of abbreviations |
|---------------|------------------------------------|
| VEGF | vascular endothelial growth factor |
| WBC | white blood cell |
| WOCBP | woman of childbearing potential |

## **Definition of Key Study Terms**

| Terms | Definition of terms |
|---|---|
| Baseline | Assessments of subjects as they enter a study before they receive any treatment. |
| Endpoint | Variable that pertains to the efficacy or safety evaluations of a study. |
| Enroll | To register or enter a subject into a clinical study. NOTE: Once a subject has received the study drug or placebo, the clinical study protocol applies to the subject. |
| Intervention | The drug, device, therapy or process under investigation in a clinical study that is believed to have an effect on outcomes of interest in a study. (e.g., health-related quality of life, efficacy, safety and pharmacoeconomics). |
| Investigational period | Period of time where major interests of protocol objectives are observed, and where the test drug or comparative drug (sometimes without randomization) is usually given to a subject, and continues until the last assessment after completing administration of the test drug or comparative drug. |
| Post investigational period | Period of time after the last assessment of the protocol. Follow-up observations for sustained adverse events and/or survival are done in this period. |
| Randomization | The process of assigning study subjects to treatment or control groups using an element of chance to determine assignments in order to reduce bias. |
| Screening | A process of active consideration of potential subjects for enrollment in a study. |
| Screen failure | Potential subject who did not meet 1 or more criteria required for participation in a study. |
| Screening period | Period of time before entering the investigational period, usually from the time when a subject signs the consent until just before the test drug or comparative drug (sometimes without randomization) is given to a subject. |
| Study period | Period of time from the first site initiation date to the last site completing the study. |
| Study Treatment | Includes zolbetuximab/placebo and both components of CAPOX |
| Variable | Any entity that varies; any attribute, phenomenon or event that can have different qualitative or quantitative values. |


## IV. PROTOCOL AMENDMENT SUMMARY OF CHANGES

| DOCUMENT HISTORY | | |
|---|---|---|
| Document | Global | <b>Country Specific</b> |
| Initial Protocol | Version 1.0 | N/A |
| First Global Substantial Amendment | Version 2.0 | N/A |
| Second Global Substantial Amendment | Version 3.0 | N/A |
| First Global Nonsubstantial Amendment | Version 3.1 | N/A |
| Third China Country-specific Substantial Amendment | N/A | 4.0 [CN] |
| Second China Country-specific Nonsubstantial Amendment | N/A | 4.1 [CN] |
| Fourth Global Substantial Amendment | Version 5.0 | N/A |
| Fifth China Country-specific Substantial Amendment | N/A | 6.0 [CN] |
| Third Japan Country-specific Nonsubstantial Amendment | N/A | 6.1 [JP] |
| Fifth Global Substantial Amendment | Version 7.0 | N/A |

## Amendment 7 [Substantial] 06 Dec 2024

This amendment is considered to be substantial based on the criteria set forth in Regulation (EU) No 536/2014 of the European Parliament. The changes in this amendment do not include any change in study conduct that would affect participant outcomes.

## **Overall Rationale for the Amendment:**

The amendment updates the following:

- Description of the investigational product vial to match the drug label update.
- Clarifications are made to existing study procedures and guidance is provided on transitioning participants to commercially marketed and locally accessible product supply.

## **Summary of Changes**

## **Substantial Changes**

| Section | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| Number | | |
| V, 2.2.1, | Added study discontinuation criterion | Zolbetuximab is available |
| 5.1.1.1, 6.1, | to conclude study once participants | outside of clinical trials in some |
| 6.3 | have transitioned to commercially | regions. |
| | marketed and locally accessible | |
| | product supply. | |

# **Nonsubstantial Changes**

| Section<br>Number | Description of Change | Brief Rationale |
|---|---|---|
| II | Update Medical Monitor and contact information. | Change in personnel. |
| II | Remove contact information for Sponsor's individual clinical research personnel (while retaining Medical Monitor). | Prevents additional future protocol amendments due to future personnel changes. |
| V, 2.2.1,<br>5.1.1.1, 5.1.4,<br>5.1.4.1,<br>5.1.4.2, 6.1 | Add a guidance to transition participants to commercially marketed and locally accessible product supply. | Zolbetuximab is available outside of clinical trials in some regions. |
| V, 2.2.1, 5.5, 5.5.5, 5.5.6, 13 | Specify requirements for safety reporting for participants continuing treatment on commercially marketed and locally accessible product supply. | Define safety reporting requirements once a participant transitions to commercially marketed and locally accessible product supply and is no longer participating in the clinical trial. |
| V, 4.1 | Add description of amount of zolbetuximab extractable from the investigational product vial. | Update vial description in protocol to match drug label update. |
| 1.1, 1.2.1 | Clarify and update nonclinical background information. | Additional relevant information for nonclinical background. |
| 13 | Specify that the section and schedules of assessments (Tables 11 and 12) apply for Protocol Versions 7.0 and later. | Clarify the continued applicability of the section. |
| Throughout | Minor administrative-type changes were made, e.g., typos, formatting, section and footnote numbering and other continuity throughout the protocol. | To provide clarification and consistency. |

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

## V. SYNOPSIS

| Date and Version No of Protocol Synopsis: | 06 Dec 2024, Version 8.0 |
|---|---|
| Sponsor: Astellas Pharma Global Development Inc. (APGD) | Protocol Number:<br>8951-CL-0302 |
| Name of Study Drug:<br>Zolbetuximab (IMAB362) | Phase of Development:<br>Phase 3 |

## Title of Study:

A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus CAPOX Compared with Placebo Plus CAPOX as First-line Treatment of Subjects with Claudin (CLDN)18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma

## **Planned Study Period:**

From 4Q2018 to 3Q2025

## **Study Objective(s):**

## **Primary**

• To evaluate the efficacy of zolbetuximab plus capecitabine and oxaliplatin (CAPOX) compared with placebo plus CAPOX (as first-line treatment) as measured by Progression Free Survival (PFS) in subjects with Claudin (CLDN) 18.2-positive, human epidermal growth factor receptor 2 (HER2)-negative locally advanced unresectable or metastatic gastric and gastroesophageal junction (GEJ) adenocarcinoma

#### Secondary

- To evaluate efficacy as measured by Overall Survival (OS) as a key secondary objective
- To evaluate the physical function (PF), OG25-Pain and GHS/QoL scores as measured by European Organization for Research and Treatment of Cancer (EORTC) as a key secondary objective
- To evaluate efficacy as measured by Objective Response Rate (ORR)
- To evaluate efficacy as measured by Duration of Response (DOR)
- To evaluate safety and tolerability of zolbetuximab
- To further evaluate other health related quality of life (HRQoL) using additional parameters as measured by EORTC QLQ-C30 and QLQ-OG25 plus STO22 Belching subscale, Global Pain (GP) and the EuroQOL Five Dimensions Questionnaire 5L (EQ5D-5L) questionnaires
- To evaluate the pharmacokinetics of zolbetuximab
- To evaluate the immunogenicity profile of zolbetuximab

#### **Exploratory**

- To evaluate efficacy as measured by Time to Progression (TTP)
- To evaluate PFS following subsequent anticancer treatment (PFS2)
- To evaluate Disease Control Rate (DCR)
- To evaluate potential genomic and/or other biomarkers that may correlate with treatment outcome to zolbetuximab and CAPOX. (NOTE: Genomic and exploratory biomarker testing will not be performed on samples from subjects in China.)
- To evaluate Health Resource Utilization (HRU)

## Planned Total Number of Study Centers and Location(s):

Approximately 175 centers globally

## **Study Population:**


Subjects with locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma whose tumors are CLDN18.2-positive, HER2-negative and who have not been previously treated for metastatic disease with chemotherapy (first-line).

For the purpose of this study, CLDN18.2-positive is defined as CLDN18.2 expression in  $\geq$  75% of tumor cells demonstrating moderate to strong membranous staining as determined by central immunohistochemistry (IHC) testing.

## Number of Subjects to be Enrolled/Randomized:

Approximately 500 subjects

## **Study Design Overview:**

This global, multicenter, double-blind, 1:1 randomized, phase 3 study will evaluate efficacy of zolbetuximab plus CAPOX versus placebo plus CAPOX as first-line treatment in subjects with CLDN18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric and GEJ adenocarcinoma.

PFS as assessed by the Independent Review Committee (IRC) is the primary outcome. Secondary outcomes include OS, ORR, DOR, safety and tolerability, HRQoL, pharmacokinetics and the immunogenicity profile of zolbetuximab. Exploratory outcomes include TTP, PFS2, DCR, biomarkers, and HRU.

Approximately 500 subjects will be randomized 1:1 into 1 of 2 treatment arms:

- Arm A (zolbetuximab in combination with CAPOX chemotherapy)
- Arm B (placebo in combination with CAPOX chemotherapy)

Randomization of subjects will be stratified by the following factors:

- Region (Asia vs Non-Asia)
- Number of Organs with Metastatic Sites (0 to 2 vs  $\geq$  3)
- Prior Gastrectomy (Yes or No)

## Screening:

The Screening period is 45 days from full main informed consent form (ICF) signature. Retesting of lab values is allowed within the 45-day Screening period. Re-screening outside the 45-day window under a new subject number may be allowed once and upon discussion with the Medical Monitor. Computerized tomography (CT) scans and magnetic resonance imaging (MRI) conducted as part of a subject's routine clinical management (i.e., standard of care) obtained before signing the ICF may be utilized for screening or baseline purposes, provided the procedures met the protocol-specified criteria and were performed within the Screening period.

Formalin fixed paraffin embedded (FFPE) tumor tissue will be collected for central testing to determine CLDN18.2 and HER2 status. (*UNIQUE TO CHINA*: FFPE tumor tissue will be collected for central testing to determine CLDN18.2 status.)

An optional partial screening ICF may be available to allow central testing of tissue for CLDN18.2 and HER2 only. (*UNIQUE TO CHINA*: An optional partial screening ICF may be available to allow central testing of tissue for CLDN18.2. only)

- Archival tumor tissue is preferred.
  - A minimum of 1 FFPE tumor tissue block (preferred) OR a minimum\* of 15 FFPE unstained slides are required as allowed per local policy. If slides are submitted, the slides should be freshly cut from the FFPE block within the time frame described in the laboratory manual.

- If local HER2 results are already available from local testing, a <u>minimum\* of 12</u> FFPE unstained slides are required to be submitted to the central laboratory as allowed per local policy.
- \*If the required minimum number of slides is not able to be submitted, sponsor notification and approval is required.
- If the specimen is insufficient or unavailable, a biopsy may be performed to obtain tumor sample.
  - Sponsor pre-approval is required when the sole purpose of the biopsy procedure is to assess eligibility for this study.
  - o If the required number of slides cannot be provided, the sponsor or designee should be contacted for further guidance.
  - o (*UNIQUE TO CHINA*: Five FFPE unstained slides are required, as allowed per local policy. The slides should be freshly cut from the FFPE block within the time frame described in the laboratory manual.)

#### Treatment Period:

Subjects will be treated with either zolbetuximab (Arm A) or placebo (Arm B) on day 1 of each cycle (for all study treatments, a cycle is defined as approximately 21 days) until the subject meets study treatment discontinuation criteria or zolbetuximab is commercially marketed and locally accessible. Once the product is commercially marketed and locally accessible, participants should complete the study, transition to commercial supply and follow the local label for treatment. Astellas is planning to close the clinical study when zolbetuximab (Vyloy) is commercially marketed in all countries with active participants and all participants have successfully transitioned to an alternative means of drug supply.

During treatment on study protocol, subjects will receive up to 8 treatments of CAPOX treatment. Oxaliplatin is administered on day 1 of each cycle, whereas capecitabine is taken twice daily on days 1 through 14. After a maximum of 8 treatments of oxaliplatin, subjects may continue to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the subject meets study treatment discontinuation criteria. (NOTE: An ECG is required to be performed and assessed locally prior to every oxaliplatin infusion [before any antiemetic treatment] and following completion of every oxaliplatin infusion. ECG should be performed up to 48 hours *prior* to and up to 6 hours *following* every oxaliplatin infusion. Oxaliplatin administration and electrolyte levels should be managed according to investigator judgment for subjects with grade 1 or 2 hypokalemia, hypomagnesemia and/or hypocalcemia.) Participants who discontinue zolbetuximab and continue to receive CAPOX or components of CAPOX should complete procedures on the study and transition to commercially marketed and locally accessible product(s) (CAPOX or its applicable components).

Radiologic imaging will be evaluated every 9 weeks ( $\pm$  7 days) counting from cycle 1/day 1 (C1D1) for the first 54 weeks and every 12 weeks ( $\pm$  7 days) thereafter until subject develops radiological disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 locally or by IRC or starts other systemic anticancer treatment, whichever occurs earlier. If a subject discontinues CAPOX (or oxaliplatin only) due to any reason other than disease progression as confirmed locally or by IRC, they may continue on zolbetuximab/placebo at the discretion of the investigator provided that all of the following have been met:

- the subject completed at least 2 cycles of CAPOX treatment;
- the subject will not receive another systemic chemotherapy, immunotherapy, radiotherapy or other treatment intended for antitumor activity; and
- in the investigator's opinion, the subject continues to derive clinical benefit with acceptable toxicity. Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), radiological disease progression will be determined locally and subjects should continue to follow the Study Treatment Period see the Schedule of Assessments [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), radiological disease progression was

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

determined by IRC and subjects should continue to follow the Study Treatment Period Schedule of Assessments [Table 1].

## Safety Assessments:

Safety will be evaluated based on adverse events (AEs), vital signs, ECGs, physical exams, Eastern Cooperative Oncology Group (ECOG) performance status and laboratory assessments. Severity of AEs and laboratory abnormalities will be assessed based on National Cancer Institute-Common Terminology Criteria For Adverse Events (NCI-CTCAE) v4.03.

## Radiologic Imaging and Independent Review Committee:

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), radiologic imaging will be evaluated locally [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), radiographic imaging was evaluated centrally by IRC.

Radiologic imaging will be evaluated at Screening (within 28 days prior to randomization) and every 9 weeks (±7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (±7 days) thereafter until subject develops radiological disease progression per RECIST 1.1 by local confirmation or IRC or starts other systemic anticancer treatment, whichever comes earlier.

All radiologically evaluable disease (measurable and/or non-measurable), per local assessment, must be documented at Screening and re-assessed at each subsequent radiologic evaluation. Imaging will include CT scans with contrast of the thorax, abdomen, and pelvis. If CT scan with contrast is medically not feasible, magnetic resonance imaging (MRI) may be used for imaging. Bone scans (or focal X-ray) or brain imaging should be performed if metastatic disease in bone or brain is suspected, respectively. The same mode of imaging should be utilized throughout the study unless medical necessity requires a change. For randomized subjects, screening imaging should be sent to the central imaging vendor no later than at the time of submission of the first on-treatment imaging. All imaging acquired post randomization will be sent to the local or central imaging vendor within 7 days of scanning for the blinded IRC assessment of radiological tumor response based on RECIST 1.1 [Eisenhauer et al, 2009]. The investigator should make every effort to immediately submit radiologic assessments for local or IRC review when progressive disease (PD) is suspected.

## Study Treatment Discontinuation and Safety Follow-up Visits:

Following discontinuation from zolbetuximab/placebo, subjects will have a zolbetuximab/placebo Study Treatment Discontinuation Visit within 7 days after the decision to discontinue, and 30-day and 90-day Safety Follow-up Visits after their last dose of zolbetuximab/placebo. If a participant transitions to commercially marketed zolbetuximab and has discontinued from the study, the 30-and 90-day safety follow up visits are not required. Once participants have transitioned to commercially marketed zolbetuximab, safety assessment and reporting should continue as per post-marketing product requirements.

Additionally, if CAPOX (both components) is discontinued on a different day than zolbetuximab/placebo, subjects will also have a Study Treatment Discontinuation Visit within 7 days after the decision to discontinue, and 30-day and 90-day Safety Follow-up Visits after the last dose of CAPOX (both components). The CAPOX 30-day and 90-day Safety Follow-up Visits may be conducted by telephone if the subject is unable to visit the study site and will require contact for AE/SAE collection only. If a participant transitions to commercially marketed CAPOX and has discontinued from the study, the 30- and 90-day safety follow up visits are not required. Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the 90-day Safety Follow-up Visit will be conducted by phone; see the Schedule of Assessments [Table 11] in [Section 13].

Post-treatment Follow-up Period (for PFS):

Note: Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the Post

Treatment Follow-up Period (for PFS) is discontinued; see the Schedule of Assessments [Table 11] in [Section 13].

Subjects that completed the 90-Day Safety Follow up Visit(s) treatment period under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) were eligible for the Post Treatment Follow up Period (for PFS) with radiological disease progression determined by IRC as outlined in Protocol Version 6.1 [Table 1].

If a subject discontinues all study treatments (zolbetuximab/placebo and both components of CAPOX) prior to IRC-confirmed radiological disease progression, the subject will enter the Post-treatment Follow-up Period and continue to undergo scheduled imaging assessments every 9 weeks (±7 days) (or every 12 weeks [±7 days] if subject has been on study over 54 weeks) until radiologic disease progression (i.e., PFS event) per IRC, or until the subject starts any other anticancer treatment, whichever occurs earlier.

If study treatments (zolbetuximab/placebo and both components of CAPOX) are discontinued due to disease progression (PFS event), the subject will enter the Long-term and Survival Follow-up Period.

## <u>Long-term Follow-up Period (for PFS2) and Survival Follow-up (for OS) Period:</u>

Note: Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the Long Term Follow-up Period (for PFS2) and Survival Follow-up (for OS) Period is discontinued; see the Schedule of Assessments [Table 11] in [Section 13].

Subjects that completed the Post-Treatment Follow-up Period (for PFS) under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) were eligible for the Long Term Follow-up Period (for PFS2) and Survival Follow-up (for OS) Period and were followed as outlined in Protocol Version 6.1 as outlined in [Table 1].

Following disease progression on first-line treatment or start of any other anticancer treatment, subjects will be followed in the Long-term and Survival Follow-up Period per institutional guidelines, but not less than every 12 weeks. Subsequent anticancer treatment details, progression status and survival status will be collected until PD following subsequent anticancer therapy (PFS2) is documented, or the subject starts another systemic anticancer treatment, whichever occurs earlier. Radiologic imaging for PFS2 will be done per local standard of care and read locally. Subjects will continue to be followed for survival status (OS) in the Survival Follow-up Period until death (from any cause).

All post-progression details including subsequent anticancer treatment and date and site of progression will be recorded on the electronic case report form (eCRF). Subject contact by phone or other remote method is sufficient during Long-term and Survival Follow-up. Additional follow-up contacts may be required per sponsor request for analysis purposes.

## Biomarkers and Other Sampling:

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), samples for pharmacokinetics, immunogenicity and biomarkers, as well as FFPE tumor tissue specimens will be collected as outlined in [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), samples for pharmacokinetics, immunogenicity and biomarkers, as well as FFPE tumor tissue specimens will be collected. Optional pharmacogenomics and post-progression tumor samples may be collected for those subjects who sign a separate informed consent form (ICF).

## Electronic Clinical Outcomes Assessments (HRQoL and HRU):

HRQoL and HRU should be assessed during the visit (or up to 48 hours) before any antiemetic or drug treatment and before the disease status is discussed with the subject. Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), assessments are discontinued [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), HRQoL and HRU were assessed at Screening (except for HRU), every 3 weeks, at study treatment

discontinuation and 30 and 90 days post zolbetuximab/placebo treatment in [Table 1]. HRQoL will be measured by EORTC QLQ-C30, QLQ-OG25 plus STO22 Belching subscale, GP and the EQ5D-5L.

## Independent Data Monitoring Committee and Independent Data Analysis Center:

An Independent Data Monitoring Committee (IDMC) will be established and will monitor the ongoing benefit-risk status of study treatment in an unblinded fashion per a pre-defined IDMC charter. The first IDMC meeting will be approximately 6 weeks after the 40th subject enrolled has completed or discontinued cycle 2 (6 weeks) and meetings will be conducted thereafter, as defined in the IDMC charter.

An Independent Data Analysis Center will conduct an interim analysis of OS at the same time as the final PFS analysis, which will occur when approximately 300 PFS events have occurred. This analysis will be utilized by the IDMC to recommend whether the study should be stopped earlier than planned if zolbetuximab in combination with CAPOX has a favorable outcome compared with placebo in combination with CAPOX. If the OS interim analysis demonstrates a highly more favorable outcome for zolbetuximab in combination with CAPOX, the study may be stopped for success. However, any subject continuing to derive clinical benefit from zolbetuximab/placebo in combination with CAPOX, as assessed by the investigator, will be allowed to continue treatment.

(UNIQUE to JP): In case that zolbetuximab is approved for marketing authorization in Japan, the study will continue as a "phase 4 post-marketing study" in accordance with Good Post-marketing Study Practice on and after the day of marketing authorization. In this case, "Study" in the protocol is read as "Post-marketing study."

#### **Inclusion/Exclusion Criteria:**

#### Inclusion Criteria:

Waivers to the inclusion criteria will **NOT** be allowed.

## **General Criteria**:

- 1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] Authorization for US sites) must be obtained from the subject or legally authorized representative (if applicable) prior to any study-related procedures.
- 2. Subject is considered an adult (e.g.,  $\geq$  18 years of age in the US) according to local regulation at the time of signing the informed consent.
- 3. A female subject is eligible to participate if she is not pregnant (negative serum pregnancy test at screening; female subjects with elevated serum beta human chorionic gonadotropin (βhCG) and a demonstrated non-pregnant status through additional testing are eligible) and at least 1 of the following conditions applies:
  - Not a woman of childbearing potential (WOCBP) as defined in [Appendix 12.3 Contraception Requirements]

#### OR

- WOCBP who agrees to follow the contraceptive guidance as defined in [Appendix 12.3 Contraception Requirements] throughout the treatment period and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
- 4. Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study treatment administration.

- 5. Female subject must not donate ova starting at screening and throughout the study period, and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
- 6. A male subject with female partner(s) of childbearing potential:
  - must agree to use contraception as detailed in [Appendix 12.3 Contraception Requirements] during the treatment period and for 6 months after the final study treatment administration.
- 7. A male subject must not donate sperm during the treatment period and for 6 months after the final study treatment administration.
- 8. Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study treatment administration.
- 9. Subject agrees not to participate in another interventional study while receiving study drug in present study.

## Disease Specific Criteria:

- 10. Subject has histologically confirmed diagnosis of Gastric or GEJ adenocarcinoma.
- 11. Subject has radiologically confirmed locally advanced unresectable or metastatic disease within 28 days prior to randomization.
- 12. Subject has radiologically evaluable disease (measurable and/or non-measurable) according to RECIST 1.1, per local assessment,  $\leq 28$  days prior to randomization. For subjects with only 1 evaluable lesion and prior radiotherapy  $\leq 3$  months before randomization, the lesion must either be outside the field of prior radiotherapy or have documented progression following radiation therapy.
- 13. Subject's tumor expresses CLDN18.2 in ≥ 75% of tumor cells demonstrating moderate to strong membranous staining as determined by central IHC testing.
- 14. Subject has a HER2-negative tumor as determined by local or central testing on a gastric or GEJ tumor specimen. (*UNIQUE TO CHINA*: Subject has a known HER2-negative gastric or GEJ tumor).

#### Physical or Laboratory Findings:

- 15. Subject has ECOG performance status 0 or 1.
- 16. Subject has predicted life expectancy  $\geq 12$  weeks in the opinion of the investigator.
- 17. Subject must meet all of the following criteria based on the centrally or locally analyzed laboratory tests collected within 14 days prior to randomization. In the case of multiple sample collections within this period, the most recent sample collection with available results should be used to determine eligibility.
  - a. Hemoglobin (Hgb)  $\geq$  9 g/dL. Subjects requiring transfusions are eligible if they have a post-transfusion Hgb  $\geq$  9 g/dL.
  - b. Absolute Neutrophil Count (ANC)  $\geq 1.5 \times 10^9 / L$
  - c. Platelets  $\geq 100 \times 10^9 / L$
  - d. Albumin  $\geq 2.5 \text{ g/dL}$
  - e. Total bilirubin  $\leq$  1.5 x upper limit of normal (ULN) without liver metastases (or < 3.0 x ULN if liver metastases are present)
  - f. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)  $\leq$  2.5 x ULN without liver metastases (or  $\leq$  5 x ULN if liver metastases are present)
  - g. Estimated creatinine clearance ≥ 30 mL/min
  - h. Prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time (PTT)  $\leq$  1.5 x ULN (except for subjects receiving anticoagulation therapy)

#### Exclusion Criteria:

Waivers to the exclusion criteria will **NOT** be allowed.

Subject who meets any of the following exclusion criteria prior to enrollment is not eligible for enrollment:

## Prohibited Treatment or Therapies:

- 1. Subject has received prior systemic chemotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma. However, subject may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies as long as it was completed at least 6 months prior to randomization.
- 2. Subject has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days prior to randomization and has not recovered from any related toxicity.
- 3. Subject has received treatment with herbal medications or other treatments that have known antitumor activity within 28 days prior to randomization.
- 4. Subject has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to randomization. Subject using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single dose of systemic corticosteroids, or receiving systemic corticosteroids as premedication for radiologic imaging contrast use is eligible.
- 5. Subject has received other investigational agents or devices within 28 days prior to randomization.

#### Medical History or Concurrent Disease:

- 6. Subject has prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibodies, including humanized or chimeric antibodies.
- 7. Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment.
- 8. Subject has prior severe allergic reaction or intolerance to any component of CAPOX.
- 9. Subject has known dihydropyrimidine dehydrogenase (DPD) deficiency. (NOTE: Screening for DPD deficiency should be conducted per local requirements.)
- 10. Subject has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
- 11. Per investigator judgment, subject has significant gastric bleeding and/or untreated gastric ulcers that exclude the subject from participation.
- 12. Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection or known active hepatitis B (positive HBs Ag) or C infection. NOTE: Screening for these infections should be conducted per local requirements.
  - a. For subjects who are negative for HBs Ag, but HBc Ab positive, an HB DNA test will be performed and if positive, the subject will be excluded.
  - b. Subjects with positive hepatitis C virus (HCV) serology but negative HCV RNA test are eligible.
  - c. Subjects treated for HCV with undetectable viral load results are eligible.
- 13. Subject has an active autoimmune disease that has required systemic treatment within the past 3 months prior to randomization.
- 14. Subject has active infection requiring systemic therapy that has not completely resolved within 7 days prior to randomization.

- 15. Subject has significant cardiovascular disease, including any of the following:
  - a. Congestive heart failure (defined as New York Heart Association [NYHA] Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, coronary artery bypass graft, cerebrovascular accident (CVA), or hypertensive crisis within 6 months prior to randomization;
  - b. History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes);
  - QTc interval > 450 msec for male subjects; QTc interval > 470 msec for female subjects;
  - d. History or family history of congenital long QT syndrome
  - e. Cardiac arrhythmias requiring anti-arrhythmic medications (Subjects with rate controlled atrial fibrillation for > 1 month prior to randomization are eligible.)
- 16. Subject has a history of central nervous system (CNS) metastases and/or carcinomatous meningitis from gastric/GEJ cancer.
- 17. Subject has known peripheral sensory neuropathy > grade 1 unless the absence of deep tendon reflexes is the sole neurological abnormality.
- 18. Subject has had a major surgical procedure  $\leq$  28 days prior to randomization.
  - a. Subject is without complete recovery from a major surgical procedure  $\leq$  14 days prior to randomization.
- Subject has psychiatric illness or social situations that would preclude study compliance, per investigator judgment.
- Subject has another malignancy for which treatment is required per investigator's clinical judgment
- 21. Subject has any concurrent disease, infection, or co-morbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data in the opinion of the investigator.

#### Investigational Product(s):

| Zolbetuximab/<br>Placebo: | Zolbetuximab: The investigational product, zolbetuximab, is a sterile lyophilized powder preparation with the chimeric monoclonal antibody zolbetuximab as the active pharmaceutical ingredient. Each vial contains 105 mg of zolbetuximab and has to be reconstituted with 5.0 mL sterile water for injection (WFI), to a concentration of 20 mg/mL. Further dilution with sterile 0.9% Sodium Chloride Injection, to a final concentration of 2 mg/mL is required. The extractable amount of zolbetuximab from each vial is 100 mg. Placebo: Placebo will not be manufactured or provided by the sponsor. 0.9% Sodium Chloride Injection will be used for placebo treatment arm as a placebo infusion solution. |
|---|---|
| Dose(s): | 800 mg/m² loading dose of zolbetuximab at C1D1 followed by subsequent doses of 600 mg/m² every 3 weeks. |
| Dosing Schedule: | Subjects will be treated with either zolbetuximab (Arm A) or placebo (Arm B) on day 1 of each cycle until the subject meets study treatment discontinuation criteria. Zolbetuximab/placebo should be administered after antiemetic premedication but <u>prior to CAPOX</u> . |
| Mode of<br>Administration: | Intravenous infusion of zolbetuximab/placebo as a minimum 2-hour infusion. Intravenous infusion may be slowed or interrupted to manage toxicity. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information. |


| 0.9% Sodium Chloride<br>Injection | 0.9% Sodium Chloride Injection will be used for infusion solution in this study for both zolbetuximab arm and placebo arm. Details of preparation of infusion solution are provided in the Pharmacy Manual and Infusion Guidelines UNIQUE TO JAPAN: In this study, 0.9% Sodium Chloride Injection is not considered an 'investigational product' as defined in J-GCP. |
|---|---|
| CAPOX: | Subjects will receive CAPOX treatment until local or IRC confirmed disease progression or a total of 8 treatments over 8 or more cycles (each cycle is defined as approximately 3 weeks = approximately 21 days). Oxaliplatin is administered on day 1 of each cycle, whereas capecitabine is taken twice daily on days 1 through 14. After 8 treatments of CAPOX, subjects may continue to receive capecitabine twice daily on days 1 through 14 of each cycle at the investigator's discretion until the subject meets study treatment discontinuation criteria. CAPOX should be administered after zolbetuximab/placebo infusion. |
| Oxaliplatin: | 130 mg/m² intravenous infusion on day 1 of each cycle over 2 hours (or longer per institutional standard of care) for a maximum of 8 treatments. (NOTE: ECG is required to be performed and assessed locally prior to every oxaliplatin infusion [before any antiemetic treatment] and following completion of every oxaliplatin infusion. ECG should be performed up to 48 hours <i>prior</i> to and up to 6 hours <i>following</i> every oxaliplatin infusion. Oxaliplatin administration and electrolyte levels should be managed according to investigator judgment for subjects with grade 1 or 2 hypokalemia, hypomagnesemia, and/or hypocalcemia). |
| Capecitabine | Administered orally at 1000 mg/m <sup>2</sup> twice daily (bid) (total daily dose is 2000 mg/m <sup>2</sup> ) on days 1 through 14 of each cycle |
| Antiemetic Pre-medications | Antiemetic premedication (prophylactic antiemetics) should be administered prior to each study treatment. (NOTE: Subjects receiving zolbetuximab do not need to be premedicated for prevention of infusion-related reactions [IRRs]; however, subjects should be closely monitored for IRRs to facilitate early identification and management.) |
| | <ul> <li>Antiemetic premedication</li> <li>IV antiemetic premedication should be initiated prior to treatment, or</li> <li>Oral antiemetic premedication should be initiated at a minimum of 30 minutes prior to zolbetuximab/placebo treatment.</li> <li>It is recommended that the prophylactic antiemetic regimen include (but is not limited to) the following agents: <ul> <li>NK-1 receptor blockers</li> <li>5-HT3 receptor blockers*</li> </ul> </li> <li>*To minimize the risk of Torsades de Pointes, administer 5-HT3 receptor blockers with caution to subjects who have or may develop QTc prolongation.</li> <li>Antiemetic premedication should be administered according to institutional standard of care, published guidelines and the respective product package insert(s).</li> <li>Corticosteroids: <ul> <li>The impact of corticosteroids on the potential efficacy of zolbetuximab is not known. Therefore, consideration should be given to avoid or minimize the use of corticosteroids as a prophylactic antiemetic if possible.</li> </ul> </li> </ul> |
| | <ul> <li>corticosteroids as a prophylactic antiemetic, if possible.</li> <li>For a subject's <u>first dose</u> of zolbetuximab/placebo, it is recommended that the prophylactic use of corticosteroids <u>be avoided</u>.</li> </ul> |

## **Concomitant Medication Restrictions or Requirements:**

## Prohibited Concomitant Treatment

The following are <u>strictly prohibited</u>:

- Sorivudine or analogs (during capecitabine treatment)
- Concurrent nonsteroid systemic immunosuppressive agents (for systemic corticosteroids see cautionary concomitant treatment below).
- Live vaccines should be avoided during the treatment period in which subject is receiving oxaliplatin or capecitabine and up to 6 months after final oxaliplatin or capecitabine dose. In cases where a live vaccine is needed for COVID-19 prevention and allowed per local regulations, please contact the Medical Monitor for discussion.
- Other systemic chemotherapy, immunotherapy, radiotherapy, herbal medications or other treatments intended for antitumor activity.
  - o Palliative radiotherapy for peripheral bone metastases is allowed.
  - o For gastric bleeding, palliative radiotherapy is prohibited, but esophagogastroduodenoscopy with epinephrine injection is allowed.
- Investigational products or therapy other than zolbetuximab.

## Cautionary Concomitant Treatment

Considerations should be given to avoid or minimize the use of the following concomitant medications, if possible, during <u>zolbetuximab/placebo</u> treatment:

- Systemic corticosteroids, because their impact on the potential efficacy of zolbetuximab is not known.
  - Systemic corticosteroids should be avoided or minimized while subject is on study treatment unless required for management of an emergent medical condition (e.g., severe nausea/vomiting or hypersensitivity reaction).
  - o For a subject's <u>first dose</u> of zolbetuximab/placebo, it is recommended that the prophylactic use of corticosteroids be avoided.
  - o Inhaled, intranasal, ophthalmic, otic and topically applied steroids are allowed.
  - Subjects are allowed to use a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg/day of hydrocortisone or up to 10 mg/day of prednisone), receive a single dose of systemic corticosteroids or receive systemic corticosteroids as pre-medication for radiologic imaging contrast use.
- Administer 5-HT3 blockers with caution in subjects who have or may develop QTc prolongation.
- Nonsteroidal anti-inflammatory drugs (NSAIDs) because of the potential to cause gastric
  ulcers and covert bleeding.
  - In such cases where NSAID use is necessary, the use of NSAIDs with lower gastric
    ulcerogenic potential is preferred and concomitant gastric protection with proton pump
    inhibitors is recommended.

The following should be avoided or used with caution and closely monitored during <u>capecitabine</u> administration:

- CytochromeP450 (CYP) 2C9 substrates (Subjects taking coumarin-derivative anticoagulants concomitantly with capecitabine should have PT/INR monitored regularly and anticoagulant dose adjusted accordingly).
- Anti-epileptic medications (e.g. phenobarbital, phenytoin and primidone)
  The following should be avoided or used with caution and closely monitored during <u>oxaliplatin</u> administration:

• Medications known to prolong the QT or QTc interval (refer to https://www.crediblemeds.org for a list of these medications)

Prohibited and cautionary concomitant treatments are described in Appendix 12.4.

#### **Duration of Treatment:**

Subjects will receive zolbetuximab/placebo until locally or IRC confirmed disease progression, toxicity requiring study treatment cessation, start of another anticancer treatment, or other treatment discontinuation criteria are met.

Subjects will also receive up to 8 treatments of CAPOX followed by continued use of capecitabine (based on investigator's judgment) beyond 8 treatments until treatment discontinuation criteria are met.

## **Study Treatment Discontinuation Criteria:**

A subject who enrolled in the study and for whom study treatment (zolbetuximab/placebo and <u>both</u> components of CAPOX) is permanently discontinued for any reason will be assessed as having met study treatment discontinuation criteria.

As overall survival is the key secondary end-point of the study, all subjects will be followed for survival after meeting study treatment discontinuation criteria unless the subject withdraws consent or is considered lost to follow-up after repeated attempts to contact or if the sponsor discontinues the study.

A subject is free to withdraw from the study treatment and/or study for any reason and at any time without giving reason for doing so and without penalty or prejudice. The investigator is also free to terminate a subject's involvement in the study at any time if the subject's clinical condition warrants it.

The subject will be discontinued from study treatment (zolbetuximab/placebo and both components of CAPOX) if any of the following occur:

- Investigator determines it is in the subject's best interest to discontinue study treatment.
- Subject develops radiological disease progression per RECIST 1.1 criteria based on assessment locally or by IRC.
  - o If the investigator believes that the subject is continuing to derive clinical benefit (asymptomatic and/or without worsening of performance status or overall health) from study treatment, and an increase in tumor burden is not likely to affect vital organ function, the subject may remain on study treatment until an additional radiologic assessment is completed (≤ 9 weeks from previous radiologic assessment).
    - If the additional radiologic assessment locally or by IRC indicates PD per RECIST 1.1, then the subject must be discontinued from study treatment.
    - If the additional radiologic assessment locally or by IRC does not confirm the initial assessment of PD, the subject may continue to receive study treatment.
- Subject develops clinical progression per investigator assessment and radiologic assessment is not medically feasible to confirm radiologic progression due to the subject's condition.
- Subject starts another systemic chemotherapy, immunotherapy, radiotherapy or other treatment intended for antitumor activity.

- Subject starts another investigational agent or device.
- Subject develops unacceptable toxicity.
- Subject has a delay of zolbetuximab/placebo <u>and</u> both components of CAPOX for > 28 days from when the next zolbetuximab/placebo <u>and</u> both components of CAPOX treatment was scheduled to be begin (> 49 days from when the last dose of zolbetuximab/placebo and both components of CAPOX treatment began).
- Any clinical AE, laboratory abnormality, or inter-current illness, in the opinion of the investigator, indicates continued treatment is not in the best interest of the subject
- Female subject becomes pregnant.
- Significant deviation from the protocol or eligibility criteria as determined by the sponsor.
- Subject declines further treatment.
- Subject is lost to follow-up despite reasonable efforts by the investigator to locate the subject.
- Subject is noncompliant with the protocol based on investigator or Medical Monitor assessment.

Note, if a subject discontinues both components of CAPOX and zolbetuximab/placebo due to any reason other than locally confirmed or IRC confirmed disease progression (and is not receiving any other anticancer therapy), the subject must be followed according to the protocol-specified radiologic assessment schedule until radiological disease progression per RECIST 1.1 criteria is confirmed locally or by IRC assessment.

#### **Study Discontinuation Criteria**

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6) [Flow Chart] all subjects should remain in the study through the 90 Day Safety Follow-up and the Post Treatment Follow-up Period (for PFS) is no longer applicable; see the Schedule of Assessments [Table 11] in [Section 13].

Participation in the study will end when subjects transition to commercially marketed and locally accessible product(s) (both zolbetuximab and CAPOX). Astellas is planning to close the study when zolbetuximab (Vylov) is commercially marketed in all countries with active participants.

Subjects that completed the 90-Day Safety Follow up Visit(s) treatment period under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) were eligible for the Post Treatment Follow up Period (for PFS) and were to remain in the study through Survival Follow-up Period (OS is a key secondary study endpoint) [Flow Chart] and followed as outlined in Protocol Version 6.1 [Table 1]. A subject will be discontinued from the Post-treatment, Long-term and Survival Follow-up Periods if any of the following occur:

- Subject specifically withdraws consent for any further contact with him/her or persons previously authorized by the participant to provide this information
- Subject is lost to follow-up despite reasonable efforts by the investigator to locate the subject
- Death (from any cause)
- Study termination by the sponsor

### **Endpoints for Evaluation:**

## **Primary:**

 PFS, defined as the time from the date of randomization until the date of radiological PD (by IRC per RECIST 1.1) or death from any cause, whichever is earliest

#### **Secondary:**

• OS, defined as the time from the date of randomization until the date of death from any cause

- Time to confirmed deterioration (TTCD) using the PF, OG25-Pain and GHS/QoL scores as measured by EORTC QLQ-C30 and QLQ-OG25 plus STO22 Belching subscale. TTCD is defined as time to first confirmed deterioration, i.e., time from randomization to first clinically meaningful deterioration that is confirmed at the next scheduled visit.
- ORR, defined as the proportion of subjects who have a best overall response of complete response (CR) or partial response (PR) as assessed by IRC per RECIST 1.1
- DOR, defined as the time from the date of the first response (CR/PR) until the date of PD as assessed by IRC per RECIST 1.1 or date of death from any cause, whichever is earliest
- Safety and tolerability, as measured by AEs, laboratory test results, vital signs, ECGs and ECOG performance status
- HRQoL, using the additional parameters as measured by EORTC QLQ-C30, QLQ-OG25 plus STO22 Belching subscale, GP, and EQ5D-5L questionnaires
- Pharmacokinetics of zolbetuximab, C<sub>trough</sub>
- Immunogenicity of zolbetuximab as measured by the frequency of antidrug-antibody (ADA) positive subjects

## **Exploratory:**

- TTP, defined as the time from the date of randomization until the date of PD as assessed by IRC per RECIST 1.1.
- PFS2, defined as the time from the date of randomization until the date of PD (per investigator) following subsequent anticancer therapy, death from any cause or start of any other anticancer therapy, whichever is earliest
- DCR, defined as the proportion of subjects who have a best overall response of CR, PR or SD as assessed by IRC per RECIST 1.1
- Potential genomic and/or other exploratory biomarkers that may be related to treatment outcome of zolbetuximab. (NOTE: Genomic and exploratory biomarker testing will not be performed on samples from subjects in China.)
- HRU

## **Statistical Methods:**

#### **Sample Size Justification:**

One interim analysis and 1 final analysis are planned for OS, while only 1 final analysis is planned for PFS. The OS interim analysis will occur at the same time of final PFS analysis (after pre-specified number of PFS events) and final OS analysis will be performed after the pre-specified number of OS events are observed. The O'Brien-Fleming boundaries as implemented by Lan-DeMets (1983) alpha spending method (East®) will be used for the OS interim and OS final analyses. All statistical tests of treatment effects will be conducted at the 1-sided 0.025 level of significance unless otherwise specified.

Approximately 500 subjects will be randomized in a 1:1 ratio to receive zolbetuximab in combination with CAPOX chemotherapy (Arm A) or placebo in combination with CAPOX chemotherapy (Arm B).

The planned 300 PFS events during the study will provide 93.4% power to detect a difference in PFS between Arm A (zolbetuximab+CAPOX) with the assumption of 9 months median PFS time and Arm B (placebo+CAPOX) with the assumption of 6 months median PFS time (hazard ratio = 0.67) at the overall 1-sided 0.025 significance level. Similarly, the planned 386 OS events during the study will provide 80% power to detect a difference in OS between Arm A (zolbetuximab+CAPOX) with the assumption of 14.7 months median survival time and Arm B (placebo+CAPOX) with the assumption of 11 months median OS time (hazard ratio = 0.75) at the overall 1-sided 0.025 significance level.

## **Analysis Populations:**

- The full analysis set (FAS) will include all subjects who are randomized to 1 of the treatment arms. Subjects will be analyzed according to the treatment arm to which they were randomized to. The FAS will be used for description of baseline characteristics and all efficacy analyses.
- The safety analysis set (SAF) will contain all subjects who received at least 1 dose of any study drug (zolbetuximab/placebo/CAPOX). The SAF will be used for all safety analyses. Subjects will be analyzed according to the actual treatment they received.
- The pharmacokinetic analysis set (PKAS) will consist of the subset of the SAF for which at least one zolbetuximab concentration measurement is available. Additional subjects may be excluded from the PKAS at the discretion of the pharmacokineticist. The PKAS will be used for description of pharmacokinetic data.

## **Efficacy Analyses:**

All efficacy analyses will be performed using FAS.

## **Primary Efficacy Endpoint:**

The primary efficacy endpoint of PFS will be analyzed using the stratified Log Rank Test with stratification factors to be specified in the SAP.

The hypothesis testing on the primary analysis will be performed at an overall 1-sided 0.025 significance level to test the null hypothesis that PFS is not prolonged in Arm A compared to Arm B versus the alternative hypothesis that PFS is prolonged in Arm A compared to Arm B.

Estimates of the treatment effect will be expressed as Hazard Ratio using a stratified Cox model, including 95% Confidence Interval.

The sensitivity analysis for the primary efficacy endpoint will also be performed.

## **Secondary Endpoints:**

The key secondary efficacy endpoint of OS will be analyzed using the stratified Log Rank Test with the same strata used in the analysis of PFS. To maintain the overall Type I error rate at the 0.025 significance level, the hypothesis testing on OS will be performed only if the null hypothesis on the primary analysis is rejected at the overall 1-sided 0.025 significance level. The key secondary TTCD endpoints of PF, OG25 Pain, and GHS/QoL will be analyzed using the same method as OS and PFS.

The secondary efficacy endpoint of ORR will be analyzed using the Cochran-Mantel-Haenszel test to control for the same strata used in the analysis of PFS and OS. The secondary efficacy endpoint of DOR will be analyzed similarly to PFS and OS.

The secondary HRQoL endpoints collected via the EORTC QLQ-C30 and QLQ-OG25 plus STO22 Belching subscale, GP and EQ-5D-5L will be analyzed with summary of change from baseline over time through the end of CAPOX treatment and inferential methods. Detailed analysis of HRQoL endpoints will be provided in the statistical analysis plan.

## **Exploratory Endpoints:**

TTP and PFS2 will be analyzed in a similar way as PFS. However, in TTP analysis, deaths are not counted as events; rather, deaths are censored. DCR will be analyzed similarly as ORR. The HRU variables will be summarized by treatment arm.

## **Safety Analyses:**

The safety evaluation will be based on AEs, clinical laboratory tests, vital signs, ECG and ECOG status. Descriptive statistics will be used to summarize safety data. All safety data will be summarized by treatment received (SAF).

All summaries of AEs will include only treatment-emergent events unless otherwise stated. AEs will be categorized by SOC and preferred term using MedDRA and will be graded for severity according to the NCI-CTCAE v4.03.

#### **Pharmacokinetics:**

Descriptive statistics will be used to summarize serum concentrations of zolbetuximab. The potential relationship between zolbetuximab immunogenicity and zolbetuximab pharmacokinetics, efficacy, and safety profile may be assessed. Additional model-based analyses may be performed and reported separately.

#### **Biomarkers:**

Biomarkers will be summarized graphically or descriptively, and summary statistics may be tabulated. Associations between biomarkers and clinical (e.g., efficacy, safety or pharmacodynamics, or pharmacokinetics) measures may be performed on subjects who have sufficient baseline and on-study treatment measurements to provide interpretable results for specific parameters.

#### **Interim Analyses:**

To evaluate whether zolbetuximab + CAPOX (Arm A) is beneficial compared to placebo + CAPOX (Arm B) while the study is ongoing, a formal OS interim analysis is planned when the final PFS analysis occurs with the pre-specified number of PFS events. A group sequential design using the O'Brien-Fleming type alpha-spending function [Lan & DeMets, 1983] for efficacy will be utilized to control the overall 1-sided 0.025 significance level (East®) for the OS analyses.

The IDMC may recommend terminating the study for favorable results at the formal efficacy interim analysis using OS. In the case of favorable results, the 1-sided significance level for superiority is 0.0074, assuming about 70% of the target number of OS events is obtained, for the interim OS analysis and 0.0228 for the final OS analysis. (Note: The OS significance level will be adjusted depending on the number of OS event at the time of interim analysis). If the 1-sided P value of the interim analysis is less than the significance level (and PFS is also significant at 1-sided 0.025 alpha), the IDMC may recommend terminating the study for success. If the study is not stopped after the interim analysis, a final OS analysis will occur after 100% of the planned death events have been observed.

Details for the interim analyses, monitoring subject safety, enrollment rates and event (PFS/death) rates will be contained in the IDMC Charter. Recommendations regarding study conduct will be made by the IDMC based on their assessment of these rates.

## VI. FLOW CHART, STUDY SCHEMATICS AND SCHEDULE OF ASSESSMENTS

## a. Up Through Protocol Version 6.1: Flow Chart



CAPOX: capecitabine and oxaliplatin; CLDN: claudin; HER2: human epidermal growth factor receptor 2; IRC: independent review committee; OS: overall survival; PFS: progression free survival; PFS2: progression free survival following subsequent anticancer treatment; RECIST: Response Evaluation Criteria In Solid Tumors

†This assessment at this timepoint has been changed with implementation of Protocol Version 7.0. Please refer to [Table 11] for the Protocol Version 7.0 and later Schedule of Assessments.
## b. Study Treatment Period Dosing Schedule (1 Cycle = approximately 21 Days)

| | Cycles 1-8 | | Cycle 9+ | | |
|---|---|---|---|---|---|
| Day 1 | Days 2-14 | Days 15-21 | Day 1 | Days 2-14 | Days 15-21 |
| Z/P | | | Z/P | | |
| OX | | No<br>Treatment | | | No<br>Treatment |
| \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | | ireacinent | | | ireacinent |
| CAP | CAP | | (CAP) | CAP | |

Cycles 9+: Subjects may continue on Capecitabine at Investigator's discretion



Sponsor: APGD

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


## **Dosing Schematics:**

a. Combination Zolbetuximab/Placebo and CAPOX Dosing (Cycle 1 to Cycle 8)



**Note**: Standard timeframes described above may be modified as per Section 5.1.2, Study Treatment Dose Modifications, Delays and Interruptions

tx: treatment.


## b. Zolbetuximab/Placebo Only Dosing (Cycle 9 and onwards)\*



**Note**: Standard timeframes described above may be modified as per Section 5.1.2, Study Treatment Dose Modifications, Delays and Interruptions

\*Cycles 9+: Subjects may continue on Capecitabine at Investigator's discretion

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


Table 1 Up Through Protocol 6.1 (Original Protocol Version 1 Through 6.1): Schedule of Assessments

| | | Study Treatment Period (Each Cycle = approximately 21 Days) | | | | | | | Follow-up Period | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISIT† | Screening <sup>1</sup> | <u>Cvcles 1-8</u> Zolbetuximab/Placebo + CAPOX | | | Cvcle 9+ Zolbetuximab/Placebo + Capecitabine (at investigator discretion) | | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21, 31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Visit Window (calendar days) | -45 to -1 | +7* | (no visit) | (no visit) | +7 | (no visit) | (no visit) | +7 | ±7 | ±7 | ±7 | ±14 |
| Informed Consent | X | | | | | | | | | | | |
| CLDN18.2 Tumor Sample <sup>2</sup> | X | | | | | | | | | | | |
| HER2 Tumor Sample <sup>2</sup> | X | | | | | | | | | | | |
| Biopsy (if applicable) <sup>2</sup> | X | | | | | | | | | | | |
| Medical and Disease History | X | | | | | | | | | | | |
| Confirmation of Inclusion/Exclusion Criteria <sup>3</sup> | X | | | | | | | | | | | J |
| Randomization <sup>4</sup> | | X | | | | | | | | | | |
| Treatments | | | | | | | | | | | | |
| Antiemetic Pretreatment <sup>5</sup> | | X | | | X | | | | | | | |
| Zolbetuximab/Placebo <sup>6</sup> | | X | | | X | | | | | | | |
| Post-infusion Observation Period <sup>7</sup> | | X | | | X | | | | | | | |
| Oxaliplatin CAPOX8 | | X | | | | | | | | | | |
| Capecitabine | | X | X | | X | X | | | | | | |
| Safety Assessments | ** | ** | | | ** | | | I | | | | |
| Physical Examination <sup>9</sup> | X | X | | | X | | | X | X | | | |
| Weight <sup>9</sup> | X | X | | | X | | | X | X | | | |
| Vital Signs <sup>10</sup> | X | X | | | X | | | X | X | | | |
| ECOG Performance Status <sup>9</sup> 12-lead ECG <sup>11</sup> | X | X<br>X | TC 1 | i i 11 i 11 | X | 11 | | X | X <sup>31</sup> | | | |
| | X<br>X <sup>1</sup> | | | | | | | | | | | |
| Image Assessment <sup>12</sup> | X <sup>1</sup> | Every 9 weeks ±7 days from C1D1 for the first 54 weeks and then every 12 weeks ±7 days thereafter <sup>31</sup> | | | | | | | | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


| | | Study Treatment Period (Each Cycle = approximately 21 Days) | | | | | | | Follow-up Period | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISIT† | Screening <sup>1</sup> | Cycles 1-8 Zolbetuximab/Placebo + CAPOX | | | Cycle 9+ Zolbetuximab/Placebo + Capecitabine (at investigator discretion) | | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21,31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Visit Window (calendar days) | -45 to -1 | +7* | (no visit) | (no visit) | +7 | (no visit) | (no visit) | +7 | ±7 | ±7 | ±7 | ±14 |
| Subject Contact | | | | | | | | | | | | X <sup>31</sup> |
| Laboratory Tests | | | • | | | | | | | | | |
| Biochemistry <sup>13</sup> | X | X | | | X | | | X | X | | | |
| TSH and Free T4 <sup>13</sup> | X | | | If clinicall | y indicated | | | X | | | | |
| Hematology <sup>13</sup> | X | X | | | X | | | X | X | | | |
| Coagulation Parameters (PT, PTT and INR) <sup>14</sup> | X | | | If clinicall | | | | | | | | |
| Urinalysis <sup>13</sup> | X | X | | | $X^{31}$ | | | X <sup>31</sup> | $X^{31}$ | | | |
| Serum Pregnancy Test <sup>15</sup> | X | | If clinically | y indicated and | or per local re | quirements | | | | | | |
| Urine Pregnancy Test <sup>16</sup> | | X | | | X | | | X | X | | | |
| DPD testing per local requirements | X | | | | | | | | | | | |
| Cytokine/Chemokine and/or Tryptase | | If clinically indicated | | | | | | | | | | |
| Electronic Clinical Outcomes Assessments (eCOA) | | | | | | | | | | | | |
| HRQoL <sup>17</sup> | X | X | | | $X^{31}$ | | | $X^{31}$ | X <sup>31</sup> | $X^{31}$ | | |
| Health Resource Utilization (HRU) <sup>17</sup> | | X | | | X <sup>31</sup> | | | X <sup>31</sup> | X <sup>31</sup> | X <sup>31</sup> | | |
| Sampling | | | | | | | | | | | | |
| Pharmacokinetics of Zolbetuximab (Serum) <sup>23</sup> | | X | | | X | | | | X <sup>31</sup> | $X^{31}$ | | |
| Antidrug-Antibodies (ADA) for Immunogenicity <sup>24</sup> | | X | | | X | | | | X <sup>31</sup> | X <sup>31</sup> | | |
| Genetic Immune Polymorphisms (Whole Blood) <sup>25</sup> | | X | | | | | | | | | | |
| Exploratory Biomarkers (Serum) <sup>26</sup> | | X | | | | | | $X^{31}$ | | | | |
| Exploratory Biomarkers (Plasma) <sup>26</sup> | | X | | | | | | X <sup>31</sup> | | | | |
| Whole Blood Sample for PGx (optional) <sup>27</sup> | | X | | | | | | | | | | |
| Post-progression Tumor Sample (optional) <sup>28</sup> | | | | | | | | X | | | | |
| Concomitant Medication <sup>29</sup> | X | X | | | X | | | X | X | $X^{31}$ | | |
| AE/SAE <sup>30</sup> | X | X | | | X | | | X | X | $X^{31}$ | | |

Footnotes appear on next page

06 Dec 2024


ADA: antidrug antibody; AE: adverse event; βhCG: beta human chorionic gonadotropin; C1D1: Cycle 1 Day 1; CAPOX: capecitabine and oxaliplatin; CLDN: claudin; CT: computerized tomography; DPD: dihydropyrimidine dehydrogenase; ECG: electrocardiogram; eCOA: electronic Clinical Outcomes Assessment; ECOG: Eastern Cooperative Oncology Group; eCRF: electronic case report form; FFPE: formalin fixed paraffin embedded; HER2: human epidermal growth factor receptor 2; HRQoL: health-related quality of life; HRU: Health Resource Utilization; ICF: informed consent form: INR: international normalized ratio; IRC: independent review committee; IRR: infusion-related reaction; IRT: interactive response technology; IV: intravenous; MRI: magnetic resonance imaging; OS: overall survival; PD: progressive disease; PFS: progression free survival; PFS2: progression free survival following subsequent anticancer treatment; PGx: pharmacogenomics; PT: prothrombin time; PTT: partial thromboplastin time; RECIST: Response Evaluation Criteria In Solid Tumors; SAE: serious adverse event; T4: thyroxine; TSH: thyroid stimulating hormone

†Local and/or regional protocols or precautions for COVID-19 management should be followed as applicable.

\*+7 calendar day visit window does not apply to C1D1.

- 1. <u>Screening</u>: The Screening period is 45 days from full main ICF signature. Retesting of lab values is allowed within the 45-day Screening period. Re-screening outside the 45-day window under a new subject number may be allowed once and upon discussion with the Medical Monitor. CT scans and MRIs conducted as part of a subject's routine clinical management (i.e., standard of care) obtained before signing the ICF may be utilized for screening or baseline purposes, provided the procedures met the protocol-specified criteria and were performed within the Screening period.
  - Optional partial screening: A partial screening ICF may be available for central testing of tissue for CLDN18.2 and HER2 only. (UNIQUE TO CHINA: A partial screening ICF may be available for central testing of tissue for CLDN18.2 only.)
  - Laboratory testing:
    - Eligibility can be determined based on central and/or local laboratory testing; however:
      - o The most recent laboratory tests with available results must be used to confirm the subject's eligibility.
      - o Central labs must be collected and submitted to the central laboratory during the Screening period.
      - o If retesting of lab values is necessary to confirm eligibility, local labs can be used without requiring additional sample collection for central laboratory submission.
    - The screening labs used to determine eligibility should be collected within 14 days prior to randomization.
  - Radiologic imaging used to confirm eligibility must be conducted within 28 days prior to randomization.
- 2. <u>CLDN18.2 and HER2 Testing</u>: FFPE tumor tissue will be collected for central testing to determine CLDN18.2 and HER2 status. (*UNIQUE TO CHINA*: FFPE tumor tissue will be collected for central testing to determine CLDN18.2 status.) Archival tumor tissue from the primary tumor (gastric or GEJ) is preferred. If primary tumor tissue is not available, tumor tissue from a metastatic site (excluding bone metastasis) may be used. A minimum of 1 FFPE tumor tissue block (preferred) OR a minimum of 15 FFPE unstained slides are required as allowed per local policy. If slides are submitted, the slides should be freshly cut from the FFPE block within the time frame described in the laboratory manual. If local HER2 results are already available from local testing, a minimum of 12 FFPE unstained slides are required to be submitted to the central lab as allowed per local policy. If the specimen is insufficient or unavailable, a biopsy may be performed to obtain primary tumor tissue (preferred) or tumor tissue from metastatic site (excluding bone metastasis). Sponsor pre-approval is required when the sole purpose of the biopsy procedure Tumor Tissue Samples]. (*UNIQUE TO CHINA*: Five FFPE unstained slides are required, as allowed per local policy.)
- 3. Confirmation of Inclusion/Exclusion Criteria must be completed prior to randomization. is to assess eligibility for this study. If the required number of slides cannot be provided, the sponsor or designee should be contacted for further guidance. See [Section 5.7.3]


4. <u>Randomization</u>: After confirmation of eligibility, the blinded site user will perform the randomization IRT transaction. The unblinded pharmacist/designee will be notified by the IRT system about the randomly assigned treatment. Randomization may be performed prior to C1D1. If C1D1 cannot be performed within 5 calendar days from Randomization, please contact the Medical Monitor for discussion. Details of infusion preparation and storage requirements are defined in the Pharmacy Manual and Infusion Guidelines.

- 5. <u>Antiemetic Pretreatment</u>: Antiemetic premedication (prophylactic antiemetics) should be administered prior to each study treatment. IV antiemetic premedication should be initiated prior to treatment, or oral antiemetic premedication should be initiated at a <u>minimum of 30 minutes</u> prior to treatment. Antiemetic premedication should be given according to institutional standard of care, published guidelines and the respective product package insert(s). For further details, see [Section 5.1.1.2 Antiemetics].
- 6. <u>Zolbetuximab/placebo</u> will be administered as a minimum 2-hour intravenous infusion every 3 weeks starting on C1D1. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information. Zolbetuximab/placebo should be administered prior to CAPOX. For further details, see [Section 5.1.1.1 Zolbetuximab/Placebo].
- 7. Post-infusion Observation Period: Following the first dose of zolbetuximab/placebo on C1D1, the subject must be observed for 2 hours post zolbetuximab/placebo infusion. The post-infusion observation period can be conducted during the CAPOX administration. If any ≥ grade 2 AEs are observed during infusion or during the post-infusion observation period, subsequent zolbetuximab/placebo infusion times should be extended and subjects should continue to be observed for 2 hours post zolbetuximab/placebo infusion. If the subject does not develop any grade ≥ 2 AEs, the subject should be observed for 1 hour post-infusion for their subsequent zolbetuximab/placebo infusions. The subject should be instructed to notify site personnel if they develop any AEs during this observation time period. In the event of an IRR with features of anaphylaxis (regardless of grade) or grade 3 or 4 IRR, blood samples for cytokine/chemokine panel and serum total tryptase level (levels typically peak within 3 hours after the onset of symptoms) should be collected once the subject has stabilized, for shipment to the central laboratory. See Observation Period following zolbetuximab/placebo infusion [Section 5.4.2] for further details.
- 8. CAPOX is a combination of oxaliplatin intravenous infusion and capecitabine tablets and will be administered starting at C1D1 for up to 8 treatments. See [Section 5.1.1.3].
- 9. Physical Exam: should include height (at Screening only), weight and ECOG performance status. A full physical exam is required at Screening. The physical exam only needs to be repeated on C1D1 if clinically significant changes from screening are observed (in the opinion of the investigator). For all cycles, the physical examination, weight and ECOG performance status assessments can be completed up to 48 hours prior to zolbetuximab/placebo administration. Targeted (symptom driven) physical exams should be conducted every 3 weeks on day 1 of each cycle. For further details, see [Section 5.4.4 Physical Examination]
- 10. <u>Vital signs</u> (pulse, blood pressure, temperature) should be taken during every visit at the following time points (see [Section 5.4.1 Vital Signs]):
  - o Predose at every visit
  - o C1D1: Every 30 (±10) minutes during zolbetuximab/placebo infusion
    - o If the subject did not develop any ≥ grade 2 AEs during the C1D1 zolbetuximab/placebo infusion or Post-infusion Observation Period, the site may do the following for subsequent zolbetuximab/placebo infusions:
    - The post-infusion observation period can be 1 hour for subsequent visits after C1D1
    - The vital signs can be assessed every 60 minutes for subsequent visits after C1D1
  - o Every 60 (±10) minutes post zolbetuximab/placebo infusion during the Post-infusion Observation Period (for 1 or 2 hours. See footnote 7)
  - o Unscheduled if clinically indicated

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

- 11. <u>ECGs</u>: ECGs will be locally assessed. When collected on the same day, ECG should be collected prior to pharmacokinetic samples. For further details, see [Section 5.4.5 Electrocardiogram]. A single ECG will be performed at the following time points:
  - o Screening
  - o Up to 48 hours prior to every oxaliplatin infusion (before any antiemetic treatment administration)
  - o Up to 6 hours following completion of every oxaliplatin infusion
  - o Zolbetuximab/placebo Discontinuation Visit
  - o Zolbetuximab/placebo 30-day Follow-up Visit
  - o If clinically indicated or per local requirements
- 12. Imaging Assessments: Radiologic imaging will be evaluated at Screening (must be conducted within 28 days prior to randomization) and every 9 weeks (± 7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (± 7 days) thereafter until subject develops radiological disease progression per RECIST 1.1 by IRC or starts other systemic anticancer treatment, whichever comes earlier. Imaging schedule should be maintained regardless of treatment delay. Imaging will include CT scans with contrast of the thorax, abdomen, and pelvis. If CT scan with contrast is medically not feasible, MRI may be used for imaging. Bone scans (or focal X-ray) or brain imaging should be performed if metastatic disease in bone or brain is suspected, respectively. The same mode of imaging should be utilized throughout the study unless medical necessity requires a change. For randomized subjects, screening imaging should be sent to the central imaging vendor no later than at the time of submission of the first on-treatment imaging. All imaging acquired post randomization will be sent to the central imaging vendor within 7 days of scanning for the blinded independent central assessment of radiological tumor response based on RECIST 1.1. The investigator should make every effort to immediately submit radiologic assessments for IRC review when PD is suspected. See [Section 5.3 Efficacy Assessments]. Refer to Imaging Acquisition Guidelines for further detail on scan modality and contrast options.
- 13. <u>Laboratory Assessments</u>: See [Section 5.4.3 Laboratory Assessments] for list of laboratory assessments. Laboratory tests must be sent to the central laboratory for analysis. For screening/eligibility laboratory assessments, see footnote number 1.
  - <u>Laboratory test results (central or local) will be reviewed by the investigator prior to any study treatment</u>. Clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician.
  - Local laboratory results may be used for treatment decisions; however, central laboratory samples must also be drawn per protocol and sent to the central laboratory. (*UNIQUE TO CHINA*: Local laboratory results may be used for treatment decisions; however, central laboratory samples should also be drawn per protocol and sent to the central laboratory unless otherwise approved by the sponsor.)
  - Central and local labs may be collected up to 48 hours prior to study treatment.
  - <u>Holidays</u> and weekends should be taken into account when scheduling these sample collections.
  - Additional assessments may be done centrally or locally to monitor AEs or as clinically indicated.
- 14. <u>Coagulation</u> (PT, PTT and INR): Coagulation tests should be done at Screening and during study treatment period if clinically indicated. Local or central lab results may be used to confirm eligibility. Ongoing evaluation should be continued for subjects who are receiving therapeutic anticoagulation according to local standard of care. See [Section 5.4.3 Laboratory Assessments].
- 15. Serum Pregnancy Test: Serum pregnancy tests will be collected for female subjects of childbearing potential only. Serum pregnancy tests collected at Screening, during study treatment period and if clinically indicated or per local requirements. Serum pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. (Note: For Screening, subjects with elevated serum βHCG and a demonstrated non-pregnant status through additional testing are eligible.) Local or central laboratory results may be used to confirm eligibility.


16. <u>Urine Pregnancy Test</u>: Urine pregnancy tests will be collected for female subjects of childbearing potential only. Local urine pregnancy tests to be performed during the treatment period every 3 weeks on day 1 of each cycle and at the zolbetuximab/placebo Study Treatment Discontinuation and 30-day Safety Follow-up Visits. Urine pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. Additional urine pregnancy testing for up to 9 months after the final study treatment administration may be conducted based on local requirements.

- 17. <u>HRQoL and HRU questionnaires</u>: eCOA questionnaires should be completed by the subject at Screening (except for HRU), on day 1 of each cycle (or up to 48 hours) before any antiemetic or drug treatment and before the disease status is discussed with the subject, using the electronic tablet device provided. When completion by the subject is not possible, the questionnaires may be administered to the subject by site personnel using the electronic tablet device. For subjects with low literacy, situations where translations are unavailable or other circumstances preventing the screening questionnaires to be completed, please contact the sponsor for further guidance.
- 18. <u>Study Treatment Discontinuation Visit (End of Study Treatment):</u> The Study Treatment Discontinuation Visit will take place ≤ 7 days following the decision to discontinue study treatment (zolbetuximab/placebo and CAPOX [both components]). If zolbetuximab/placebo and CAPOX (both components) are discontinued on a different day, subjects will have separate Study Treatment Discontinuation Visits following each treatment's discontinuation. Laboratory tests must be sent to the central laboratory for analysis. HRQoL and HRU questionnaires are not required at CAPOX treatment discontinuation visit. A combined visit can be completed if zolbetuximab/placebo are discontinued on the same day.
- 19. 30-day Safety Follow-up Visit: A 30-day Safety Follow-up Visit should occur 30 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 30-day Safety Follow-up Visit should occur 30 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. HRQoL and HRU questionnaires are not required at CAPOX 30-day safety follow up visit. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day and HRQoL and HRU questionnaires should be completed for a combined visit.
- 20. 90-day Safety Follow-up Visits: A 90-day Safety Follow-up Visit should occur 90 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 90-day Safety Follow-up Visit should occur 90 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. HRQoL and HRU questionnaires are not required at CAPOX 90-day safety follow up visit. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day and HRQoL and HRU questionnaires should be completed for a combined visit.
- 21. <u>Post-treatment Follow-up</u>: if a subject discontinues all study treatments (zolbetuximab/placebo and both components of CAPOX) prior to IRC-confirmed radiological disease progression, the subject will enter the Post-treatment Follow-up Period and continue to undergo imaging assessments every 9 weeks (±7 days) (or every 12 weeks [±7 days] if subject has been on study over 54 weeks) until radiologic disease progression (i.e., PFS) or the subject starts subsequent anticancer treatment, whichever occurs earlier. If study treatments (zolbetuximab/placebo and both components of CAPOX) are discontinued due to PD, the subject will enter the Long-term and Survival Follow-up Period.
- 22. <u>Long-term and Survival Follow-up Period</u>: Following disease progression on first-line treatment or start of subsequent anticancer treatment, subjects will be followed in the Long-term and Survival Follow-up Period per institutional guidelines, but at least every 12 weeks. Radiologic imaging will be done per standard of care and read locally until PFS2 is documented. Survival Follow-up Period will continue until death (from any cause). All post-progression details including subsequent anticancer treatment and date and site of progression will be recorded on the eCRF. Subject contact by phone or other remote methods is sufficient during Long-term and Survival Follow-up.

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

- 23. <u>Pharmacokinetics</u>: Serum samples for zolbetuximab/placebo will be taken at the below time points and sent to the central laboratory. The date and time of each blood sample collection will be recorded to the nearest minute.
  - o Cycle 1 Day 1: End of zolbetuximab/placebo infusion
  - o Cycle 2 Day 1: Predose
  - o Cycle 3 Day 1: End of zolbetuximab/placebo infusion
  - o Predose on Day 1 of Cycles 5, 9, 13 and 17
  - Zolbetuximab/placebo 30-Day Safety Follow-up visit
  - Zolbetuximab/placebo 90-Day Safety Follow-up visit
  - o Unscheduled pharmacokinetic blood samples may be taken at any time during the study to evaluate drug exposure following a safety event

## Pharmacokinetic Sampling Window:

- o Predose: within 60 minutes prior to dosing
- o End of Infusion: within 10 minutes after the end of the infusion
- 24. ADA: Blood samples (Serum) for ADA will be taken at the below time points and sent to the central laboratory.
  - o Cycle 1 Day 1: Predose
  - o Cycle 2 Day 1: Predose
  - o Predose on Day 1 of Cycles 5, 9, 13 and 17
  - o Zolbetuximab/placebo 30-Day Safety Follow-up visit
  - o Zolbetuximab/placebo 90-Day Safety Follow-up visit

ADA Sampling Window: Predose: within 60 minutes prior to dosing

- 25. <u>Genetic Immune Polymorphism</u>: To be collected per local policy. Whole blood sample taken at C1D1 will be sent to the central laboratory. Samples may be collected up to 48 hours prior to study treatment. (*UNIQUE TO CHINA*: Genomic biomarker testing will not be performed on samples from subjects in China.)
- 26. Exploratory Biomarker (Serum and Plasma): To be collected per local policy. Samples should be taken at the below time points and sent to the central laboratory:
  - o Cycle 1 Day 1: Predose
  - o Cycle 2 Day 1: Predose
  - o Cycle 3 Day 1: Predose
  - o Cycle 4 Day 1: Predose
  - o Cycle 5 Day 1: Predose
  - o Cycle 6 Day 1: Predose
  - o Cycle 8 Day 1: Predose
  - o Zolbetuximab/placebo Study Treatment Discontinuation Visit

Exploratory Biomarker samples may be collected up to 48 hours prior to study treatment.

27. (*UNIQUE TO CHINA*: Exploratory biomarker testing will not be performed on samples from subjects in China.) Optional PGx: For subjects who signed a separate ICF, an optional whole blood sample for PGx for exploratory biomarker analysis may be collected up to 48 hours prior to first study drug administration. Sample collection is optional and only collected as allowed per local policy. (*UNIQUE TO CHINA*: Genomic testing will not be performed on samples from subjects in China.)


- 28. Optional Post-Progression Tumor Sample: For subjects who signed a separate ICF, an optional post-progression tumor sample for exploratory biomarker analysis may be collected following IRC confirmation of disease progression and prior to initiation of subsequent anticancer therapy. Sample collection is optional and only collected as allowed per local policy. (UNIQUE TO CHINA: Optional post-progression tumor sample is not applicable for China.)
- 29. Concomitant medications will be collected from the time of full main informed consent through 90 days following the last dose of study treatment.
- 30. <u>AEs/SAEs</u>: AEs and SAEs (regardless of causality) will be collected from the time of full main informed consent through 90 days following the last dose of study treatment. See [Section 5.5.5 Reporting of Serious Adverse Events].
- 31. With implementation of Protocol Version 7.0, please refer to [Table 11] for the Protocol Version 7.0 and later Schedule of Assessments.

#### 1 INTRODUCTION

Gastric and gastroesophageal junction (GEJ) cancers are among the malignancies with the highest unmet medical need. Gastric cancer-related mortality is the fourth leading cause of cancer death worldwide, even if its incidence has decreased over the last 50 years in different regions of the world [Cancer Fact Sheet, 2018; Amiri et al, 2011]. On the other hand, the incidence of subjects with GEJ adenocarcinoma has increased in recent decades, coinciding with a shift in histological type and primary tumor location [Waddell et al, 2013; Sahin et al, 2008].

In 2017, an estimated 723100 people died worldwide from gastric cancer [Lederman, 2017]. The overall 5-year survival rate for gastric and GEJ cancers is averaging 20% in the US and Europe, despite aggressive standard treatments, which are also associated with substantial side effects [Pennathur et al, 2013; Sahin et al, 2008].

There is no single standard, globally accepted first-line reference chemotherapeutic regimen for advanced gastric cancer. In the US and Europe, the current standard of care cytotoxic chemotherapy regimen consists of fluoropyrimidine with platinum-based combination chemotherapy regimens with or without a third agent such as docetaxel or epirubicin [National Comprehensive Cancer Network (NCCN), 2017; Waddell et al, 2013; Pasini et al, 2011]. Subjects in this study will receive CAPOX (a combination of capecitabine and oxaliplatin), which is a globally accepted standard-of-care treatment for subjects with locally advanced unresectable or metastatic gastric or gastroesophageal (GE) cancer. The safety of this combination regimen is well-documented [Kim et al, 2012].

The lack of a major benefit from the various newer generation combination chemotherapy regimens for these cancers has stimulated research into the use of targeted agents such as monoclonal antibodies (mAbs). Two mAbs, trastuzumab and ramucirumab, have received approval for treatment of gastric cancer. Trastuzumab selectively binds the extracellular domain of human epidermal growth factor receptor 2 (HER2), which is overexpressed in approximately 20% to 30% of gastric tumors [Bang et al, 2009], and ramucirumab specifically binds vascular endothelial growth factor (VEGF) receptor 2 and blocks binding of VEGF receptor ligands VEGF-A, VEGF-C and VEGF-D. Trastuzumab is approved for treatment of HER2 overexpressing metastatic gastric or GEJ adenocarcinoma while ramucirumab is approved as a single agent or in combination with paclitaxel, for treatment of advanced gastric or GEJ adenocarcinoma, with disease progression on or after prior fluoropyrimidine-or platinum-containing chemotherapy [CYRAMZA Prescribing Information, 2017; HERCEPTIN Prescribing Information, 2016]. These agents prolonged median overall survival (OS) by 4 or fewer months when given alone or in combination with chemotherapy compared with standard of care cytotoxic chemotherapy [Fuchs et al, 2014; Wilke et al, 2014; Ohtsu et al, 2011; Bang et al, 2010].

Approximately 70% to 80% of patients with metastatic or advanced unresectable gastric and GEJ adenocarcinoma in the first line setting have tumors that are HER2 negative and are not treatable with trastuzumab. These patients have an expected median survival of approximately 1 year [Shah et al, 2017]. Therefore, a significant unmet medical need exists 06 Dec 2024 Astellas

for the first-line treatment of patients with HER2 negative locally advanced or metastatic unresectable gastric and GEJ cancers. Zolbetuximab is being developed with the goal of addressing this unmet medical need.

# 1.1 Background

Zolbetuximab is a genetically engineered, highly purified chimeric (mouse/human IgG1) antibody directed against the tight junction molecule Claudin 18.2 (CLDN18.2). The target is a member of the claudin family of more than 20 structurally related proteins that are involved in the formation of tight junctions in epithelia and endothelia [Niimi et al, 2001]. Tight junctions, together with adherens junctions and desmosomes, form the apical junctional complex in epithelial and endothelial cellular sheets. Adherens junctions and desmosomes are responsible for the mechanical adhesion between adjacent cells, whereas tight junctions are essential for the tight sealing of the cellular sheets forming a luminary barrier and controlling the paracellular ion flux.

CLDN18.2 is a 27.7 kDa protein with 4 membrane-spanning domains and 2 small extracellular loops [Gunzel & Yu, 2013; Sahin et al, 2008]. Zolbetuximab recognizes the first extracellular domain of CLDN18.2 with high affinity and specificity. Zolbetuximab does not bind to any other claudin family member including the closely related splice variant 1 of Claudin 18 (CLDN18.1).

CLDN18.2 is a highly cell type specific differentiation antigen that is expressed by differentiated gastric mucosa cells in the pit and base regions of gastric glands. Moreover, CLDN18.2 is not detectable in any other normal cell type of the human body either at transcript level or as protein. This highly selective tissue distribution pattern results in CLDN18.2 expression being strictly confined to a subpopulation of gastric epithelial cells in normal tissue [Sahin et al, 2008].

CLDN18.2 is expressed in a diversity of human cancers and is the dominant isoform in GE and pancreatic cancer [Lee et al, 2011]. The expression of CLDN18.2 is retained upon malignant transformation of gastric epithelia and is present in 81% of primary gastric adenocarcinomas. CLDN18.2 expression is frequently detected in diffuse and in intestinal gastric cancers. The CLDN18.2 protein is also localized in lymph node metastases of gastric cancer adenocarcinomas and in distant metastases into the bile duct, lung and especially into the ovary (so-called Krukenberg tumors). Furthermore, over 42% of esophageal adenocarcinomas and 50% to 70% of pancreatic cancers display significant expression of CLDN18.2 [Wöll et al, 2014; Lee et al, 2011; Sanada et al, 2010; Karanjawala et al, 2008; Sahin et al, 2008].

Zolbetuximab is being developed for the first-line treatment of adult subjects with locally advanced unresectable or metastatic CLDN18.2-positive, HER2-negative gastric or GEJ adenocarcinoma in combination with platinum- and fluoropyrimidine-based chemotherapy. For this study, a subject's tumor must express CLDN18.2 in  $\geq 75\%$  of tumor cells demonstrating moderate to strong membranous staining as determined by central immunohistochemistry (IHC) testing.

### 1.2 Nonclinical and Clinical Data

#### 1.2.1 Nonclinical Data

In vitro studies with CLDN18.2-positive and negative cancer cell lines showed that zolbetuximab binds to the extracellular domain 1 of CLDN18.2 on human gastric cancer cell lines with high relative affinity and selectivity. In vitro assays demonstrated that zolbetuximab mediated an efficient lysis of CLDN18.2-positive cells through antibody-dependent cellular cytotoxicity (ADCC) and complement-dependent cytotoxicity (CDC).

All zolbetuximab-mediated effects are strictly CLDN18.2 antigen-specific.

In bio-distribution studies in nude mice with human tumor xenografts, intravenously administered zolbetuximab was retained, as well as specifically and strongly enriched in CLDN18.2-positive human xenografts. No or little in vivo binding of zolbetuximab to any other mouse tissues including stomach tissue was observed.

Administration of repeated doses of zolbetuximab to mice bearing CLDN18.2-positive tumors resulted in retardation of tumor growth kinetics in tumor models.

A series of in vitro experiments were conducted with CLDN18.2-expressing cell lines derived from NUGC-4 and KATO-III to investigate the effects of combining these chemotherapy agents with zolbetuximab. Combinations of chemotherapy agents used in the treatment of gastric and esophageal cancers, including 5-FU, oxaliplatin and epirubicin (e.g., 5-FU/oxaliplatin, 5-FU/oxaliplatin/epirubicin) augmented zolbetuximab activity. In vitro pre-sensitization of human gastric cancer cells with chemotherapy resulted in an increase in the amount of cell surface CLDN18.2 and thus improved zolbetuximab-mediated ADCC and CDC.

In immunocompetent mice, zolbetuximab in combination with chemotherapy resulted in a pronounced T cell infiltration into the tumors and significant long-term survival benefit over zolbetuximab alone. In the same animal model, the combination treatment of zolbetuximab with oxaliplatin and 5-FU significantly inhibited tumor growth compared with each monotherapy of zolbetuximab or the chemotherapeutic agents, along with an increase in tumor-infiltrating CD8+ T cells. These effects might be mediated by induction of adaptive T cell immunity, which may have led to the antitumor effect and immune surveillance.

CLDN18.2 is highly conserved across species, and the epitope of zolbetuximab is identical between humans, mice and cynomolgus monkeys. In addition, the binding affinity of zolbetuximab to CLDN18.2 orthologs from mice, humans and cynomolgus monkeys was shown to be comparable, providing sufficient evidence that testing in mice and monkeys covers the potential on-target effects and toxicities of zolbetuximab.

The nonclinical pharmacology studies conducted with zolbetuximab provide sufficient experimental evidence that zolbetuximab depletes CLDN18.2-positive cells via ADCC and CDC. Cytotoxic drugs were shown to increase CLDN18.2 expression on human cancer cells

and to improve the activity of the major mechanism of action (ADCC and CDC). Hence, the combination of zolbetuximab with first-line chemotherapy is being investigated in the clinic.

Safety pharmacology and toxicity of zolbetuximab were assessed in mice and cynomolgus monkeys. In mice, the maximum exposure tested was 300 mg/kg weekly over 13 weeks, and in cynomolgus monkeys, the maximum exposure tested was 100 mg/kg weekly over 4 weeks.

In both species, no target organs of toxicity were identified; however, in monkeys, emesis was observed in a non-dose-related manner. The emesis that was observed in monkeys was not severe and spontaneously resolved despite continued dosing. The emetic potential of zolbetuximab was confirmed in an investigational study in ferrets. This effect is considered to be related to the binding of zolbetuximab to junctional protein, CLDN18.2, in the gastric epithelium. A human tissue cross-reactivity study of zolbetuximab showed that the gastric mucosa was the only tissue with strong membrane staining. However, histological assessment of the gastric tissue in monkeys failed to identify any histopathological lesions.

Besides the findings listed previously, no other zolbetuximab-related adverse effects were observed in any organ, neither clinically, nor macroscopically or histologically upon postmortem analysis.

In summary, the nonclinical data outlined above supports the clinical development of zolbetuximab in combination with standard chemotherapy for the treatment of CLDN18.2-positive gastric or GEJ adenocarcinoma.

Please refer to the current IB for most recent nonclinical data.

#### 1.2.2 Clinical Data

CLAUDETECT<sup>TM</sup>18.2.

Zolbetuximab has been evaluated in clinical studies as a single agent and in combination with epirubicin, oxaliplatin and capecitabine (EOX) chemotherapy or in combination with immunomodulation therapy (zoledronic acid [ZA] with or without interleukin-2 [IL-2]) for the treatment of adult subjects with CLDN18.2-positive advanced adenocarcinoma of the stomach, esophagus or GEJ.

CLDN18.2 expression was immunohistochemically determined for all subjects enrolled in the clinical studies. Several studies had an enrichment type of design meaning that only subjects above a certain threshold of CLDN18.2 positivity in their tumors were eligible for treatment. Eligibility for enrollment in the GM-IMAB-001-03 (EudraCT No. 2011-005285-38) and GM-IMAB-001-04 (EudraCT No. 2011-005509-64) studies, hereafter referred to as FAST and PILOT, respectively, was determined using the analytically validated and Conformité Européene (CE)-marked diagnostic kit,

To date, 4 clinical studies have been completed and include GM-IMAB-001 (EudraCT No. 2008-004719-37, referred to as first-in-human [FIM]), PILOT, FAST and GM-IMAB-001-02 (EudraCT No. 2009-017365-36) referred to as MONO.

Zolbetuximab has been granted orphan drug designation for the treatment of stomach cancer by the EMA and FDA.

Clinical data from the studies described above supports the clinical development of zolbetuximab in combination with standard chemotherapy for the treatment of CLDN18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric or GEJ adenocarcinomas.

Please refer to the current IB for most recent clinical data.

# 1.3 Summary of Key Safety Information for Study Drugs

As of 06 May 2019, zolbetuximab has been administered to 306 subjects including 259 subjects in the following 4 completed clinical studies:

- FIM study as a single monotherapy dose (up to 1000 mg/m<sup>2</sup>) in 15 subjects;
- MONO study as repeated monotherapy doses up to 600 mg/m<sup>2</sup> once every 2 weeks in 54 subjects (maximum exposure was 72 infusions);
- FAST study as repeated doses of zolbetuximab in combination with EOX chemotherapy (up to 1000 mg/m<sup>2</sup> once every 3 weeks) in 162 subjects (maximum exposure greater than 40 infusions); and
- PILOT study in combination with immunomodulation therapy (up to 600 mg/m<sup>2</sup> once every 3 weeks) in 28 subjects.

And 2 ongoing open-label clinical studies:

- 8951-CL-0103 (ILUSTRO) as monotherapy or in combination with mFOLFOX6 in 32 subjects
- 8951-CL-0104 as monotherapy in 15 Japanese subjects

Current phase 1/2 study status and enrollment are available in the zolbetuximab Investigator's Brochure (IB) (see Table 13 in the IB).

Nausea and vomiting have been confirmed as important identified risks as has hypersensitivity reactions (HSRs), including infusion-related reactions (IRRs). Anemia and neutropenia are considered important potential risks. These important identified risks along with important potential risks, based on observations from the clinical studies, are described in Section 5.2 of the IB. Expected adverse drug reactions, including reference safety information (RSI) used for expedited health authority reporting are described in Appendix 1 of the IB.

One patient from an ongoing Phase 2 study (monotherapy arm) experienced grade 4 acute coronary syndrome, grade 4 cardiac arrest, and grade 4 posterior reversible encephalopathy syndrome (PRES), and grade 3 pulmonary embolism, 22 days after the first infusion of zolbetuximab monotherapy. The patient had a medical history significant for uncontrolled hypertension, asthenia and anemia. The patient recovered from these events, which were deemed serious, and a possible causal relationship to zolbetuximab could not be excluded. Refer to the IB for additional details.

In clinical studies, adverse reactions with nausea and/or vomiting and HSRs up to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade 3 were reported. Subjects receiving zolbetuximab should receive prophylactic antiemetic

06 Dec 2024 Astellas 

medications, but do not need to be premedicated for prevention of HSRs and IRRs; however, subjects should be closely monitored for IRRs to facilitate early identification and management. In the case of zolbetuximab-induced nausea, vomiting or hypersensitivity including IRRs, the infusion rate of zolbetuximab may be reduced or the infusion may be paused or discontinued based on investigator's clinical judgment about severity of toxicity and local standard of care.

Detailed information on the toxicities associated with CAPOX can be found within Section 4.8 of the EU summary of product characteristics (SPC) or local product information for each component.

Potential overlapping toxicities during treatment with zolbetuximab in combination with CAPOX include nausea, vomiting, abdominal pain, constipation, diarrhea, fatigue, HSR, infusion reactions, weight loss and edema.

# 1.4 Efficacy

## 1.4.1 Efficacy Results from Study GM-IMAB-001-02 (MONO)

In the MONO study, efficacy analyses included subjects who received zolbetuximab at least once (Full Analysis Set [FAS]) at doses of 300 mg/m² (3 subjects) and 600 mg/m² (40 subjects). The best overall confirmed response for FAS subjects in the zolbetuximab 600 mg/m² dose group was partial response [PR] in 4 subjects (10.0%) that ranged in duration from 43 through 1037 days (GM-IMAB-001, Listing 13.2.6.4). The best overall confirmed response was stable disease (SD) in 6 subjects (15.0%) and progressive disease (PD) in 28 subjects (70.0%) in the 600 mg/m² group (GM-IMAB-001-02, Table 12.3.7.1). No subject achieved complete response (CR). Median progression free survival (PFS) in the FAS was 10 weeks (95% confidence interval [CI]: 8.6, 10.1 weeks) in the 600 mg/m² group (GM-IMAB-001-02, Table 12.3.3.1).

### 1.4.2 Efficacy Results from Study GM-IMAB-001-03 (FAST)

Treatment groups in the FAST study are referred to as EOX, EOX + IMAB600 (EOX plus zolbetuximab 600 mg/m<sup>2</sup> once every 3 weeks, with a loading dose of 800 mg/m<sup>2</sup> in cycle 1) and EOX + IMAB1000 (EOX plus zolbetuximab 1000 mg/m<sup>2</sup> once every 3 weeks).

In the FAST study, efficacy analyses of all randomized subjects were included in the intent-to-treat set and included subjects randomized to EOX only (85 subjects), EOX + IMAB600 (79 subjects) and EOX + IMAB1000 (88 subjects). Additional analyses were completed for the FAS, defined as randomized subjects who received at least 1 dose of any study drug (E, Ox, capecitabine or zolbetuximab). The FAS differed from the intent-to-treat set (all randomized subjects) by 6 subjects all of whom discontinued the study early without death or post-baseline tumor assessment. The reasons for early discontinuation of these subjects included protocol violation (1 subject), physician decision (1 subject), withdrawal by subject (2 subjects) and adverse event (AE) (1 subject was anemic and another had a deep vein thrombosis) (GM-IMAB-001-03, Listing 13.2.1).

### PFS Based on Central Independent Review (Kaplan-Meier Model, Intent-to-Treat)

The addition of zolbetuximab to EOX led to a statistically significant prolongation of PFS, both for the lower zolbetuximab dose (hazard ratio [HR] 0.45, P < 0.0005) and the higher zolbetuximab dose (HR 0.57, P = 0.0114). Median PFS was 7.5 months in the EOX + IMAB600 arm and 7.1 months in the EOX + IMAB1000 arm vs 5.3 months in the EOX arm, representing a median PFS prolongation by 2.2 and 1.8 months, respectively [IB, Table 17].

#### Overall Survival (Kaplan-Meier, Intent-to-Treat)

The addition of zolbetuximab  $600 \text{ mg/m}^2$  led to a statistically significant prolongation in OS (HR 0.52, P < 0.0005). Median OS was 13 months in the EOX + IMAB600 arm vs 8.3 months in the EOX arm, representing an increase in median OS by 4.7 months. In the EOX + IMAB1000 arm, median OS was 9.6 months and hence, numerically longer than in the EOX arm [IB, Table 18]. However, the difference between the groups did not reach statistical significance. The difference in OS between the 2 zolbetuximab doses was statistically significant (P = 0.0406) (GM-IMAB-001-03, Table 12.3.2.1.5.3).

No major imbalances were seen between the treatment groups in the subsequent use of any anticancer therapy (EOX: 38.1%; EOX + IMAB600: 40.3%; EOX + IMAB1000: 34.1%) and any chemotherapy (EOX: 34.5%; EOX + IMAB600: 39.0%; EOX + IMAB1000: 29.4%) (GM-IMAB-001-03, Tables 12.2.1.1.5.1 and 12.2.1.5 [Safety-evaluable Set]).

#### Best Objective Tumor Response by Independent Review Committee

Based on confirmed responses, the ORR was 38.0% in the EOX + IMAB600 arm, 29.5% in the EOX + IMAB1000 arm and 24.7% in the EOX arm [IB, Table 21]. This included 10.1% of subjects with a CR in the EOX + IMAB600 arm, 4.5% in the EOX + IMAB1000 arm and 3.5% in the EOX arm (GM-IMAB-001-03, Table 12.3.3.1.3).

## 1.4.3 Efficacy of CAPOX

The results from Study GM-IMAB-001-03 (FAST) using EOX support the use of CAPOX in this study, as CAPOX is similar to EOX except that CAPOX does not include epirubicin. Subjects in this study will receive CAPOX, which is an accepted standard-of-care treatment for subjects with locally advanced unresectable metastatic gastric or GE cancer [NCCN, 2017].

#### 1.5 Risk Benefit Assessment

Zolbetuximab is an investigational agent for the treatment of CLDN18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma in combination with standard of care oxaliplatin and fluoropyrimidine-based combination chemotherapy as first-line treatment.

Based on clinical efficacy and safety data from the MONO study, preliminary data from the FAST study and supportive preclinical pharmacological studies, there is potential of achieving clinically relevant benefit in combination with oxaliplatin and

fluoropyrimidine-based chemotherapy in a first-line setting and as a single agent in the later line setting.

Based on currently available clinical data, zolbetuximab was tolerated from a safety perspective and most observed AEs have been considered manageable. Nonclinical toxicity data were supportive of the clinical findings.

Important <u>identified</u> risks of zolbetuximab are:

- Nausea
- Vomiting
- HSRs (including IRRs)

Important potential risks of zolbetuximab include:

- Neutropenia
- Anemia

Management of the important identified risks associated with zolbetuximab includes antiemetic pretreatment, reduction of the initial zolbetuximab infusion rate, and pausing or discontinuing the infusion based on patient tolerability and investigator's clinical judgment about severity of toxicity and local standard of care. Subjects receiving zolbetuximab do not need to be premedicated for prevention of HSRs and IRRs; however, subjects should be closely monitored for IRRs to facilitate early identification and management.

Overall, the risks, both identified and potential, associated with zolbetuximab in combination with CAPOX are balanced by the anticipated benefits to subjects with CLDN18.2-positive, HER2 negative locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma.

As described in [Section 10.1], an Independent Data Monitoring Committee (IDMC) will be responsible for reviewing the unblinded data from the study to ensure the safety of the subjects.

# 2 STUDY OBJECTIVE(S), DESIGN AND ENDPOINTS

# 2.1 Study Objective(s)

#### 2.1.1 Primary Objectives

The primary objective is to evaluate the efficacy of zolbetuximab plus CAPOX compared with placebo plus CAPOX (as first-line treatment) as measured by Progression Free Survival (PFS) in subjects with Claudin (CLDN) 18.2-positive, human epidermal growth factor receptor 2 (HER2)-negative locally advanced unresectable or metastatic gastric and gastroesophageal junction (GEJ) adenocarcinoma.

#### 2.1.2 Secondary Objectives

The secondary objectives are:

• To evaluate efficacy as measured by Overall Survival (OS) as a key secondary objective

- To evaluate the physical function (PF), OG25-Pain and GHS/QoL scores as measured by European Organization for Research and Treatment of Cancer (EORTC) as a key secondary objective
- To evaluate efficacy as measured by Objective Response Rate (ORR)
- To evaluate efficacy as measured by Duration of Response (DOR)
- To evaluate safety and tolerability of zolbetuximab
- To further evaluate other health related quality of life (HRQoL) using additional parameters as measured by EORTC QLQ-C30 and QLQ-OG25 plus STO22 Belching subscale, Global Pain (GP) and the EuroQOL Five Dimensions Questionnaire 5L (EQ5D-5L) questionnaires
- To evaluate the pharmacokinetics of zolbetuximab
- To evaluate the immunogenicity profile of zolbetuximab

### 2.1.3 Exploratory Objectives

The exploratory objectives are:

- To evaluate efficacy as measured by Time to Progression (TTP)
- To evaluate PFS following subsequent anticancer treatment (PFS2)
- To evaluate Disease Control Rate (DCR)
- To evaluate potential genomic and/or other biomarkers that may correlate with treatment outcome to zolbetuximab and CAPOX. (NOTE: Genomic and exploratory biomarker testing will not be performed on samples from subjects in China.)
- To evaluate Health Resource Utilization (HRU)

# 2.2 Study Design and Dose Rationale

#### 2.2.1 Study Design

This global, multicenter, double-blind, 1:1 randomized, phase 3 study will evaluate efficacy of zolbetuximab plus CAPOX versus placebo plus CAPOX as first-line treatment in subjects with CLDN18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric and GEJ adenocarcinoma.

PFS as assessed by the Independent Review Committee (IRC) is the primary outcome. Secondary outcomes include OS, ORR, DOR, safety and tolerability, HRQoL, pharmacokinetics and the immunogenicity profile of zolbetuximab. Exploratory outcomes include TTP, PFS2, DCR, biomarkers, and HRU.

Approximately 500 subjects will be randomized 1:1 into 1 of 2 treatment arms:

- Arm A (zolbetuximab in combination with CAPOX chemotherapy)
- Arm B (placebo in combination with CAPOX chemotherapy)

Randomization of subjects will be stratified by the following factors:

- Region (Asia vs Non-Asia)
- Number of Organs with Metastatic Sites (0 to 2 vs  $\geq$  3)
- Prior Gastrectomy (Yes or No)

#### Screening:

The Screening period is 45 days from full main informed consent form (ICF) signature. Retesting of lab values is allowed within the 45-day Screening period. Re-screening outside the 45-day window under a new subject number may be allowed once and upon discussion with the Medical Monitor (see Re-Screening below). Computerized tomography (CT) scans and magnetic resonance imaging (MRI) conducted as part of a subject's routine clinical management (i.e., standard of care) obtained before signing the ICF may be utilized for screening or baseline purposes, provided the procedures met the protocol-specified criteria and were performed within the Screening period.

An optional partial screening ICF may be available to allow central testing of tissue for CLDN18.2 and HER2 only. (*UNIQUE TO CHINA*: An optional partial screening ICF may be available to allow central testing of tissue for CLDN18.2. only)

Formalin fixed paraffin embedded (FFPE) tumor tissue will be collected for central testing to determine CLDN18.2 and HER2 status. (*UNIQUE TO CHINA*: FFPE tumor tissue will be collected for central testing to determine CLDN18.2 status.)

Archival tumor tissue is preferred.

- A minimum of 1 FFPE tumor tissue block (preferred) OR a <u>minimum\* of 15</u> FFPE unstained slides are required as allowed per local policy. If slides are submitted, the slides should be freshly cut from the FFPE block within the time frame described in the laboratory manual.
- If local HER2 results are already available from local testing, a <u>minimum\* of 12 FFPE</u> unstained slides are required to be submitted to the central laboratory as allowed per local policy.
  - \*If the required minimum number of slides is not able to be submitted, sponsor notification and approval is required.
- If the specimen is insufficient or unavailable, a biopsy may be performed to obtain tumor sample.
  - Sponsor pre-approval is required when the sole purpose of the biopsy procedure is to assess eligibility for this study.
  - o If the required number of slides cannot be provided, the sponsor or designee should be contacted for further guidance.
  - o (*UNIQUE TO CHINA*: Five FFPE unstained slides are required, as allowed per local policy. The slides should be freshly cut from the FFPE block within the time frame described in the laboratory manual.)

#### Re-Screening:

Subjects who have failed screening are allowed to be re-screened one time after consultation with the Medical Monitor. Upon re-screening, a new subject number will be assigned. Subjects have to re-consent to the study and all screening procedures must be repeated, with the exception of the CLDN18.2 and HER2 testing as well as the radiologic imaging procedure to confirm eligibility if the scan is within 28 days prior to randomization.

Laboratory values re-tested within the original 45-day Screening period are not considered re-screening and no new subject number will be assigned.

#### Treatment Period:

Subjects will be treated with either zolbetuximab (Arm A) or placebo (Arm B) on day 1 of each cycle (for all study treatments, a cycle is defined as approximately 21 days), until the subject meets study treatment discontinuation criteria or zolbetuximab is commercially marketed and locally accessible.

Once the product is commercially marketed and locally accessible, participants should complete the study, transition to commercial supply and follow the local label for treatment.

Astellas is planning to close the clinical study when zolbetuximab (Vyloy) is commercially marketed in all countries with active participants and all participants have successfully transitioned to an alternative means of drug supply.

During treatment on study protocol, subjects will receive up to 8 treatments of CAPOX treatment. Oxaliplatin is administered on day 1 of each cycle, whereas capecitabine is taken twice daily on days 1 through 14. After a maximum of 8 treatments of oxaliplatin, subjects may continue to receive capecitabine taken twice daily on days 1 through 14 of each cycle at the investigator's discretion until the subject meets study treatment discontinuation criteria. (NOTE: An ECG is required to be performed and assessed locally prior to every oxaliplatin infusion [before any antiemetic treatment] and following completion of every oxaliplatin infusion. ECG should be performed up to 48 hours *prior* to and up to 6 hours *following* every oxaliplatin infusion. Oxaliplatin administration and electrolyte levels should be managed according to investigator judgment for subjects with grade 1 or 2 hypokalemia, hypomagnesemia, and/or hypocalcemia.)

Radiologic imaging will be evaluated every 9 weeks ( $\pm$  7 days) counting from cycle 1/day 1 (C1D1) for the first 54 weeks and every 12 weeks ( $\pm$  7 days) thereafter until subject develops radiological disease progression per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 locally or by IRC or starts other systemic anticancer treatment, whichever occurs earlier.

Participants who discontinue zolbetuximab and continue to receive CAPOX or components of CAPOX should complete procedures on the study and transition to commercially marketed and locally accessible product(s) (CAPOX or its applicable components).

## Study Treatment Discontinuation and Safety Follow-up Visits:

Following discontinuation from zolbetuximab/placebo, subjects will have a zolbetuximab/placebo Study Treatment Discontinuation Visit within 7 days after the decision to discontinue, and 30-day and 90-day Safety Follow-up Visits after their last dose of zolbetuximab/placebo. If a participant transitions to commercially marketed zolbetuximab and has discontinued from the study, the 30- and 90-day safety follow up visits are not required.

Once participants have transitioned to commercially marketed zolbetuximab, safety assessment and reporting should continue as per post-marketing product requirements.

Additionally, if CAPOX (both components) is discontinued on a different day than zolbetuximab/placebo, subjects will also have a Study Treatment Discontinuation Visit within 7 days after the decision to discontinue, and 30-day and 90-day Safety Follow-up Visits after the last dose of CAPOX (both components). The CAPOX 30-day and 90-day Safety Follow-up Visits may be conducted by telephone if the subject is unable to visit the study site and will require contact for AE/SAE collection only. If a participant transitions to commercially marketed CAPOX and has discontinued from the study, the 30- and 90-day safety follow up visits are not required.

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the 90-day Safety Follow-up Visit will be conducted by phone; see the Schedule of Assessments [Table 11] in [Section 13].

## Post-treatment Follow-up Period (for PFS):

Note: Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the Post Treatment Follow-up Period (for PFS) is discontinued; see the Schedule of Assessments [Table 11] in [Section 13].

Subjects that completed the 90-Day Safety Follow up Visit(s) treatment period under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) were eligible for the Post-Treatment Follow-up Period (for PFS) with radiological disease progression determined by IRC as outlined in [Table 1]. If a subject discontinues all study treatments (zolbetuximab/placebo and both components of CAPOX) prior to IRC-confirmed radiological disease progression, the subject will enter the Post-treatment Follow-up Period and continue to undergo scheduled imaging assessments every 9 weeks (±7 days) (or every 12 weeks [±7 days] if subject has been on study over 54 weeks) until radiologic disease progression (i.e., PFS event) per IRC, or until the subject starts any other anticancer treatment, whichever occurs earlier.

If study treatments (zolbetuximab/placebo and both components of CAPOX) are discontinued due to disease progression (PFS event), the subject will enter the Long-term and Survival Follow-up Period.

#### Long-term Follow-up Period (for PFS2) and Survival Follow-up (for OS) Period:

Note: Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the Long Term Follow-up Period (for PFS2) and Survival Follow-up (for OS) Period is discontinued; see the Schedule of Assessments [Table 11] in [Section 13].

Subjects that completed the Post-Treatment Follow-up Period (for PFS) under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) were eligible for the Long Term Follow-up Period (for PFS2) and Survival Follow-up (for OS) Period and were followed as outlined in Protocol Version 6.1 as outlined in [Table 1].

Following disease progression on first-line treatment or start of any other anticancer treatment, subjects will be followed in the Long-term and Survival Follow-up Period per institutional guidelines, but not less than every 12 weeks. Subsequent anticancer treatment details, progression status and survival status will be collected until PD following subsequent anticancer therapy (PFS2) is documented, or the subject starts another systemic anticancer treatment, whichever occurs earlier. Radiologic imaging for PFS2 will be done per local standard of care and read locally. Subjects will continue to be followed for survival status (OS) in the Survival Follow-up Period until death (from any cause).

All post-progression details including subsequent anticancer treatment and date and site of progression will be recorded on the electronic case report form (eCRF). Subject contact by phone or other remote method is sufficient during Long-term and Survival Follow-up. Additional follow-up contacts may be required per sponsor request for analysis purposes.

## Independent Data Monitoring Committee and Independent Data Analysis Center:

An IDMC will be established and will monitor the ongoing benefit-risk status of study treatment in an unblinded fashion per a pre-defined IDMC charter. The first IDMC meeting will be approximately 6 weeks after the 40th subject enrolled has completed or discontinued cycle 2 (6 weeks) and meetings will be conducted thereafter, as defined in the IDMC charter.

An Independent Data Analysis Center will conduct an interim analysis of OS at the same time as the final PFS analysis, which will occur when approximately 300 PFS events have occurred. This analysis will be utilized by the IDMC to recommend whether the study should be stopped earlier than planned if zolbetuximab in combination with CAPOX has a favorable outcome compared with placebo in combination with CAPOX. If the OS interim analysis demonstrates a highly more favorable outcome for zolbetuximab in combination with CAPOX, the study may be stopped for success. However, any subject continuing to derive clinical benefit from zolbetuximab/placebo in combination with CAPOX, as assessed by the investigator, will be allowed to continue treatment.

(UNIQUE to JP: In case that zolbetuximab is approved for marketing authorization in Japan, the study will continue as a "phase 4 post-marketing study" in accordance with Good Post-marketing Study Practice on and after the day of marketing authorization. In this case, "Study" in the protocol is read as "Post-marketing study.")

#### 2.2.2 Dose Rationale

The dose of zolbetuximab in this study is an  $800 \text{ mg/m}^2$  loading dose (C1D1) followed by  $600 \text{ mg/m}^2$  every 3 weeks in combination with CAPOX. This dose and schedule of zolbetuximab ( $800/600 \text{ mg/m}^2$  every 3 weeks) were chosen based on the observed data from the GM-IMAB-001-03 (FAST) study. In the FAST study, addition of zolbetuximab  $800/600 \text{ mg/m}^2$  every 3 weeks to EOX (Arm 2) demonstrated a statistically significant and clinically meaningful improvement on PFS and OS in subjects with CLDN18.2-positive advanced gastric/GEJ cancer compared to EOX (Arm 1). The mean serum trough concentration of zolbetuximab was maintained above the targeted value of 50 µg/mL (based on half maximal effective concentration [EC50] of in vitro ADCC and CDC activities) following  $800/600 \text{ mg/m}^2$ 

every 3 weeks administration. A higher zolbetuximab dose (1000 mg/m² every 3 weeks) in combination with EOX was added 18 months later (with the allocation ratio of 1:1:7) as Arm 3 in the FAST study to evaluate safety and efficacy at the higher dose. However, this arm had less treatment benefit compared to Arm 2. Although there were numerical differences observed in some demographics and baseline characteristics, the sample size was not sufficient to evaluate and confirm the impact of such differences; therefore, the reason for underperformance in Arm 3 remains inconclusive.

There is no single standard, globally accepted first-line reference chemotherapeutic regimen for advanced gastric cancer. A fluoropyrimidine (capecitabine or 5-FU) in combination with platinum agent (cisplatin or oxaliplatin) is an accepted standard of care cytotoxic chemotherapy regimen in both Western and Asian countries [NCCN, 2017; Ohtsu et al, 2011; Ajani et al, 2010; Vita et al, 2005; Kim et al, 1993]. Both classes of agents are considered to be interchangeable according to NCCN and European Society for Medical Oncology treatment guidelines. Subjects in this study will receive CAPOX (a combination of capecitabine and oxaliplatin), which is a globally accepted standard-of-care treatment for subjects with locally advanced unresectable or metastatic gastric or GEJ cancer. The safety of this combination regimen is well-documented.

## 2.3 Endpoints

# 2.3.1 Primary Endpoints

The primary endpoint is PFS, which is defined as the time from the date of randomization until the date of radiological PD (per RECIST 1.1 by IRC) or death from any cause, whichever is earliest.

#### 2.3.2 Secondary Endpoints

The secondary endpoints are:

- OS, defined as the time from the date of randomization until the date of death from any cause
- Time to confirmed deterioration (TTCD) using the PF, OG25-Pain and GHS/QoL scores
  as measured by EORTC QLQ-C30 and QLQ-OG25 plus STO22 Belching subscale.
  TTCD is defined as time to first confirmed deterioration, i.e., time from randomization to
  first clinically meaningful deterioration that is confirmed at the next scheduled visit.
- ORR, defined as the proportion of subjects who have a best overall response (BOR) of CR or PR as assessed by IRC per RECIST 1.1
- DOR, defined as the time from the date of the first response (CR/PR) until the date of PD
  as assessed by IRC per RECIST 1.1 or date of death from any cause, whichever is
  earliest
- Safety and tolerability, as measured by AEs, laboratory test results, vital signs, ECGs and Eastern Cooperative Oncology Group (ECOG) performance status
- HRQoL using the additional parameters as measured by EORTC QLQ-C30, QLQ-OG25 plus STO22 Belching subscale, GP and EQ5D-5L questionnaires
- Pharmacokinetics of zolbetuximab, Ctrough

• Immunogenicity of zolbetuximab as measured by the frequency of anti-drug antibody (ADA) positive subjects.

#### 2.3.3 Exploratory Endpoints

The exploratory endpoints are:

- TTP, defined as the time from the date of randomization until the date of PD as assessed by IRC per RECIST 1.1.
- PFS2, defined as the time from the date of randomization until the date of PD (per investigator) following subsequent anticancer therapy, death from any cause or start of any other anticancer therapy, whichever is earliest.
- DCR, defined as the proportion of subjects who have a BOR of CR, PR or SD as assessed by IRC per RECIST 1.1.
- Potential genomic and/or other exploratory biomarkers that may be related to treatment outcome of zolbetuximab. (NOTE: Genomic and exploratory biomarker testing will not be performed on samples from subjects in China.)
- Health Resource Utilization (HRU)

## 3 STUDY POPULATION

# 3.1 Selection of Study Population

Subjects with locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma whose tumors are CLDN18.2 positive, HER2-negative and who have not been previously treated for metastatic disease with chemotherapy (1<sup>st</sup> line).

For the purpose of this study, CLDN18.2-positive is defined as CLDN18.2 expression in  $\geq$  75% of tumor cells demonstrating moderate to strong membranous staining as determined by central IHC testing.

## 3.2 Inclusion Criteria

Waivers to the inclusion criteria will **NOT** be allowed.

#### General Criteria:

- 1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] Authorization for US sites) must be obtained from the subject or legally authorized representative (if applicable) prior to any study-related procedures.
- 2. Subject is considered an adult (e.g.,  $\geq$  18 years of age in the US) according to local regulation at the time of signing the informed consent.
- 3. A female subject is eligible to participate if she is not pregnant (negative serum pregnancy test at screening; female subjects with elevated serum beta human chorionic gonadotropin (βhCG) and a demonstrated non-pregnant status through additional testing are eligible) and at least 1 of the following conditions applies:

• Not a woman of childbearing potential (WOCBP) as defined in [Appendix 12.3 Contraception Requirements]

#### OR

- WOCBP who agrees to follow the contraceptive guidance as defined in [Appendix 12.3 Contraception Requirements] throughout the treatment period and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
- 4. Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study treatment administration.
- 5. Female subject must not donate ova starting at screening and throughout the study period, and for 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs.
- 6. A male subject with female partner(s) of childbearing potential must agree to use contraception as detailed in [Appendix 12.3 Contraception Requirements] during the treatment period and for 6 months after the final study treatment administration.
- 7. A male subject must not donate sperm during the treatment period and for 6 months after the final study treatment administration.
- 8. Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study treatment administration.
- 9. Subject agrees not to participate in another interventional study while receiving study drug in present study.

#### Disease Specific Criteria:

- 10. Subject has histologically confirmed diagnosis of Gastric or GEJ adenocarcinoma.
- 11. Subject has radiologically confirmed locally advanced unresectable or metastatic disease within 28 days prior to randomization.
- 12. Subject has radiologically evaluable disease (measurable and/or non-measurable) according to RECIST 1.1, per local assessment, ≤ 28 days prior to randomization. For subjects with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before randomization, the lesion must either be outside the field of prior radiotherapy or have documented progression following radiation therapy.
- 13. Subject's tumor expresses CLDN18.2 in  $\geq$  75% of tumor cells demonstrating moderate to strong membranous staining as determined by central IHC testing.
- 14. Subject has a HER2-negative tumor as determined by local or central testing on a gastric or GEJ tumor specimen. (*UNIQUE TO CHINA*: Subject has a known HER2 negative gastric or GEJ tumor.)

#### Physical or Laboratory Findings:

- 15. Subject has ECOG performance status 0 or 1.
- 16. Subject has predicted life expectancy  $\geq$  12 weeks in the opinion of the investigator.
- 17. Subject must meet all of the following criteria based on the centrally or locally analyzed laboratory tests collected within 14 days prior to randomization. In the case of multiple sample collections within this period, the most recent sample collection with available results should be used to determine eligibility.
  - a. Hemoglobin (Hgb)  $\geq$  9 g/dL. Subjects requiring transfusions are eligible if they have a post-transfusion Hgb  $\geq$  9 g/dL.
  - b. Absolute Neutrophil Count (ANC)  $\geq 1.5 \times 10^9 / L$
  - c. Platelets  $\geq 100 \times 10^9 / L$
  - d. Albumin  $\geq 2.5 \text{ g/dL}$
  - e. Total bilirubin  $\leq 1.5$  x upper limit of normal (ULN) without liver metastases (or < 3.0 x ULN if liver metastases are present)
  - f. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)  $\leq$  2.5 x ULN without liver metastases (or  $\leq$  5 x ULN if liver metastases are present)
  - g. Estimated creatinine clearance ≥ 30 mL/min
  - h. Prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time (PTT)  $\leq$  1.5 x ULN (except for subjects receiving anticoagulation therapy)

#### 3.3 Exclusion Criteria

Waivers to the exclusion criteria will **NOT** be allowed.

Subject who meets any of the following exclusion criteria prior to enrollment is not eligible for enrollment:

## **Prohibited Treatment or Therapies:**

- 1. Subject has received prior systemic chemotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma. However, subject may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies as long as it was completed at least 6 months prior to randomization.
- 2. Subject has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days prior to randomization and has not recovered from any related toxicity.
- 3. Subject has received treatment with herbal medications or other treatments that have known antitumor activity within 28 days prior to randomization.
- 4. Subject has received systemic immunosuppressive therapy, including systemic corticosteroids within 14 days prior to randomization. Subject using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single dose of

- systemic corticosteroids, or receiving systemic corticosteroids as premedication for radiologic imaging contrast use is eligible.
- 5. Subject has received other investigational agents or devices within 28 days prior to randomization.

#### Medical History or Concurrent Disease:

- 6. Subject has prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibodies, including humanized or chimeric antibodies.
- 7. Subject has known immediate or delayed hypersensitivity, intolerance or contraindication to any component of study treatment.
- 8. Subject has prior severe allergic reaction or intolerance to any component of CAPOX.
- 9. Subject has known dihydropyrimidine dehydrogenase (DPD) deficiency. (NOTE: Screening for DPD deficiency should be conducted per local requirements.)
- 10. Subject has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting.
- 11. Per investigator judgment, subject has significant gastric bleeding and/or untreated gastric ulcers that exclude the subject from participation.
- 12. Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection or known active hepatitis B (positive HBs Ag) or C infection. NOTE: Screening for these infections should be conducted per local requirements.
  - a. For subjects who are negative for HBs Ag, but HBc Ab positive, an HB DNA test will be performed, and if positive, the subject will be excluded.
  - b. Subjects with positive hepatitis C virus (HCV) serology but negative HCV RNA test are eligible.
  - c. Subjects treated for HCV with undetectable viral load results are eligible.
- 13. Subject has an active autoimmune disease that has required systemic treatment within the past 3 months prior to randomization.
- 14. Subject has active infection requiring systemic therapy that has not completely resolved within 7 days prior to randomization.
- 15. Subject has significant cardiovascular disease, including any of the following:
  - a. Congestive heart failure (defined as New York Heart Association [NYHA] Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, coronary artery bypass graft, cerebrovascular accident (CVA), or hypertensive crisis within 6 months prior to randomization;
  - b. History of clinically significant ventricular arrhythmias (i.e., sustained ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes);
  - c. QTc interval > 450 msec for male subjects; QTc interval > 470 msec for female subjects;
  - d. History or family history of congenital long QT syndrome

06 Dec 2024 Astellas 

- e. Cardiac arrhythmias requiring anti-arrhythmic medications (Subjects with rate controlled atrial fibrillation for > 1 month prior to randomization are eligible.)
- 16. Subject has history of central nervous system (CNS) metastases and/or carcinomatous meningitis from gastric/GEJ cancer.
- 17. Subject has known peripheral sensory neuropathy > grade 1 unless the absence of deep tendon reflexes is the sole neurological abnormality.
- 18. Subject has had a major surgical procedure  $\leq$  28 days prior to randomization.
  - a. Subject without complete recovery from a major surgical procedure ≤ 14 days prior to randomization.
- 19. Subject has psychiatric illness or social situations that would preclude study compliance, per investigator judgment.
- 20. Subject has another malignancy for which treatment is required per investigator's clinical judgment.
- 21. Subject has any concurrent disease, infection, or co-morbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data in the opinion of the investigator.

# 4 IDENTIFICATION OF STUDY TREATMENT(S)

# 4.1 Zolbetuximab (Investigational Product)

The investigational product, zolbetuximab, is a sterile lyophilized powder with the chimeric (mouse/human IgG1) monoclonal antibody zolbetuximab as the active pharmaceutical ingredient.

The investigational product is supplied by Astellas in a single-use glass vial containing 105 mg of zolbetuximab, of which 100 mg is extractable from each vial. All excipients are animal component free and of compendial grade (Pharm. Eur. current version). No preservatives are contained, since the vial is designed for single use.

The investigational product should be stored at refrigerated conditions (2°C to 8°C; 36°F to 46°F). Temperature should be controlled and monitored. Details of investigational product receipt, labeling, storage and preparation are provided in the Pharmacy Manual and Infusion Guidelines.

The zolbetuximab used in this study will be prepared, packaged, and labeled under the responsibility of qualified staff at Astellas Pharma Global Development, Inc. (APGD), Astellas US Technologies, Inc. or sponsor's designee in accordance with APGD or sponsor's designee Standard Operating Procedures (SOPs), Good Manufacturing Practices (GMP) guidelines, International Council for Harmonisation (ICH) Good Clinical Practice (GCP) guidelines, and applicable local laws/regulations.

Each vial and carton will bear a label conforming to regulatory guidelines, GMP and local laws and regulations that identifies the contents as investigational drug.

As required, a qualified person of Astellas Pharma Europe B.V. (APEBV) or sponsor's designee will perform the final release of the medication according to the requirements of the EU Directive 2003/94/EC annex 13.

# 4.2 0.9% Sodium Chloride Injection

0.9% Sodium Chloride Injection will be used for infusion solution preparation in this study for both zolbetuximab arm and placebo arm. 0.9% Sodium Chloride Injection will not be manufactured or provided to sites by the sponsor. Sites should use their own commercially obtained supply of 0.9% Sodium Chloride Injection. Details of preparation of infusion solution are provided in the Pharmacy Manual and Infusion Guidelines. *UNIQUE TO JAPAN*: In this study, 0.9% Sodium Chloride Injection is not considered an 'investigational product' as defined in J-GCP. *UNIQUE TO China*, 0.9% Sodium Chloride Injection bags provided by the Sponsor should be used for zolbetuximab and placebo to maintain the blind. In pA V6.0, the related wording is Placebo will not be manufactured by the sponsor. Details of preparation of placebo are provided in the Pharmacy Manual and Infusion Guidelines.

For manufacturing, formulation, storage, handling and preparation details please refer to the package insert, SPC or local product information supplied by the manufacturer.

# 4.3 Comparative Drug (Placebo)

Placebo will not be manufactured or provided by the sponsor. Sites should use their own commercial supply of 0.9% Sodium Chloride Injection as placebo infusion solution. Details of preparation of placebo infusion solution are provided in the Pharmacy Manual and Infusion Guidelines.

# 4.4 CAPOX (Backbone Treatment)

Capecitabine and Oxaliplatin (CAPOX) are administered in combination with zolbetuximab/placebo. CAPOX products should be given according to institutional standards, published guidelines, the respective product package insert(s) or dosed according to this protocol.

CAPOX treatment will be supplied by the responsible site pharmacy of each investigational site or by the sponsor at the sponsor's discretion. Generic drug may be used where approved by the respective regulatory authority. CAPOX treatment will be prepared and/or dispensed by the responsible site pharmacy of each investigational site.

For manufacturing, formulation, storage, handling and preparation details please refer to the package insert, SPC or local product information supplied by the manufacturer.

If CAPOX is supplied by the sponsor, CAPOX used in this study will be packaged and labeled under the responsibility of qualified staff at APGD/Astellas US Technologies, Inc. (AUST) sponsor's designee in accordance with APGD-AUST or sponsor's designee SOPs, GMP guidelines, ICH GCP guidelines, and applicable local laws/regulations.

Each product will bear a label conforming to regulatory guidelines, GMP and local laws and regulations that identifies the contents as investigational drug.

As required, a qualified person of APEBV or sponsor's designee will perform the final release of the medication according to the requirements of the EU Directive 2003/94/EC annex 13.

# 4.5 Other Drug(s)

#### 4.5.1 Antiemetic Premedication

Prophylactic antiemetics will not be provided by the sponsor but rather will be sourced by the Sites via commercial supply.

For manufacturing, formulation, storage, handling and preparation details please refer to the package insert, SPC or local product information supplies by the manufacturer.

# 4.6 Study Drug Handling

Current ICH GCP Guidelines require the investigator to ensure that study treatment and other drug deliveries from the sponsor are received by the investigator or designee and that:

- Such deliveries are recorded,
- Study drug is handled and stored according to labeled storage conditions,
- Study drug with appropriate expiry/retest and is only dispensed to study subjects in accordance with the protocol, and
- Any unused study drug is returned to the sponsor, unless prior approval is received from the sponsor allowing local standard procedures for the alternative disposition of unused study drug.

Study drug inventory and accountability records will be kept by the investigator, head of study site (*SPECIFIC TO SITES IN JAPAN*) or designee. Study drug accountability throughout the study must be documented and reconciled. The following guidelines are therefore pertinent:

- The investigator agrees not to supply study drugs to any persons except the eligible subjects in this study in accordance with the protocol.
- The investigator or designee will keep the study drugs in a pharmacy or other locked and secure storage facility under controlled storage conditions, accessible only to those authorized by the investigator to dispense these study drugs.
- A study drug inventory will be maintained by the investigator or designee. The
  inventory will include details of material received and a clear record of when they were
  dispensed and to which subject.
- At the conclusion or termination of this study, the investigator or designee agrees to
  conduct a final drug supply inventory and to record the results of this inventory on the
  Drug Accountability Record. It must be possible to reconcile delivery records with those
  of used and/or returned study drug. Any discrepancies must be accounted for and
  documented. Appropriate forms of deliveries and returns must be signed by the site staff
  delegated this responsibility.
- The site staff must return unused study drug to the sponsor or designee at the end of the study or upon expiration unless otherwise approved by the sponsor.

06 Dec 2024 Astellas 

## 4.7 Blinding

See [Appendix 12.10] for unblinding procedures following final OS database lock.

## 4.7.1 Blinding Method

The clinical study will be conducted as subject- and investigator-blinded. Subjects will be randomized to receive zolbetuximab or placebo in a blinded fashion such that neither the investigator, sponsor's study management team, clinical staff, nor subject will know which agent is being administered. All pharmacy-related tasks must be conducted by an unblinded pharmacist/designee. The unblinded pharmacist/designee must not share any unblinded information with the blinded site personnel

Upon the need for unblinding (e.g., real-time assessment of the safety data), the chair of the IDMC can ask for the release of the treatment assignment for 1 or more subjects and will identify the sponsor staff who will receive the information.

### 4.7.2 Confirmation of the Indistinguishability of the Study Drugs

The appearance of the diluted zolbetuximab solution for infusion is identical to commercial saline solution (placebo). In order to maintain the blind, the subjects randomized to the placebo treatment arm (Arm B) will receive placebo in a volume and route corresponding to the appropriate zolbetuximab dose (Arm A). The unblinded pharmacist/designee will provide the investigator or designee with blinded study drugs to dose the subjects. Refer to the Pharmacy Manual and Infusion Guidelines for detailed information.

# 4.7.3 Retention of the Assignment Schedule and Procedures for Treatment Code Breaking

The randomization list and study drug blind will be maintained by the Interactive Response Technology (IRT) system.

## 4.7.4 Breaking the Treatment Code for Emergency

The treatment code for each randomized subject will be provided by the IRT in the event of a medical emergency requiring knowledge of the treatment assigned to the subject. The IRT will be programmed with blind-breaking instructions that may only be requested by the investigator or subinvestigators designated to have access to perform blind-break. No subjects or other study personnel, other than the unblinded pharmacist or designee, will be made aware of the treatment given to any subject unless a medical emergency necessitates such disclosure. In case of a medical emergency, the investigator has the sole responsibility for determining if unblinding of subject's treatment assignment is warranted. Subject safety must always be the first consideration in making such determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the sponsor prior to unblinding a subject's treatment assignment unless this could delay emergency treatment for the subject. Any unblinding by the investigators must be reported immediately to the sponsor and must include an explanation of why the study drug was unblinded.

The investigator must have confirmed functionality to access code-break through the IRT system and must have a designated back up (e.g., redundant processes) to support emergency unblinding requirements.

Prior to randomization, subjects should be provided with information that includes the site emergency contact number and back-up contact number in case of a medical emergency. Any unblinding by the investigational staff must be reported immediately to the sponsor and include an explanation of why the study drug was unblinded. If unblinding is associated with a SAE the investigator is to follow the instructions in [Section 5.5.5 Reporting of SAE].

Care should be taken to limit knowledge of the randomization arm, in case this could affect the blinding of other subjects or future study assessment for the subject.

The time, date, subject number and reason for obtaining any of these codes, and therefore breaking the blind, must be documented in the study file.

If possible, the sponsor should be contacted prior to unblinding of the study drug.

#### 4.7.5 Breaking the Treatment Code by the Sponsor

The sponsor may break the treatment code for subjects who experience a Suspected Unexpected Serious Adverse Reaction (SUSAR), in order to determine if the individual case or a group of cases requires expedited regulatory reporting. Individual Emergency Codes will be provided to the limited staff who are responsible to break the codes for all SUSAR cases for reporting purposes.

# 4.8 Assignment and Allocation

Subject randomization will be performed by blinded site user via IRT and treatment assigned in a 1:1 ratio to zolbetuximab or placebo. Prior to the initiation of the study treatment, the unblinded pharmacist/designee will be notified by the IRT system about the randomly assigned treatment. The unblinded pharmacist/designee will dispense the treatment according to the IRT system's assignment. Specific procedures for randomization through the IRT are contained in the IRT manual.

Randomization will be stratified by:

- Region (Asia vs Non-Asia)
- Number of Organs with Metastatic Sites (0 to 2 vs  $\geq$  3)
- Prior Gastrectomy (Yes or No)

#### 5 TREATMENTS AND EVALUATION

# 5.1 Dosing and Administration of Study Drug(s) and Other Medication(s)

#### 5.1.1 Dose/Dose Regimen and Administration Period

#### 5.1.1.1 Zolbetuximab/Placebo

Subjects will be administered zolbetuximab/placebo as a minimum 2-hour intravenous infusion on day 1 of each cycle. **Guidance for slowing the initial infusion to minimize** 

**toxicity can be found in the Pharmacy Manual and Infusion Guidelines.** Subjects will be administered with a loading dose of 800 mg/m<sup>2</sup> of zolbetuximab at C1D1 followed by subsequent doses of 600 mg/m<sup>2</sup> every 3 weeks. Zolbetuximab/placebo should be administered prior to CAPOX. Flow rate data will be collected in the eCRF.

Please also refer to the dosing schematics for details [Section VI].

Intravenous infusion may be interrupted or slowed down to manage toxicity. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information.

Once the product is commercially marketed and locally accessible, participants should complete the study, transition to commercial supply and follow the local label for treatment.

Astellas is planning to close the clinical study when zolbetuximab (Vyloy) is commercially marketed in all countries with active participants and all participants have successfully transitioned to an alternative means of drug supply.

#### 5.1.1.2 Antiemetics

Antiemetic premedication (prophylactic antiemetics) should be administered prior to each study treatment.

(NOTE: Subjects receiving zolbetuximab do not need to be premedicated for prevention of IRRs; however, subjects should be closely monitored for IRRs to facilitate early identification and management.)

- Antiemetic premedication
  - o IV antiemetic premedication should be initiated prior to treatment, or
  - Oral antiemetic premedication should be initiated at a minimum of 30 minutes prior to treatment.
- It is recommended that the prophylactic antiemetic regimen include (but is not limited to) the following agents:
  - NK-1 receptor blockers
  - 5-HT3 receptor blockers\*

Antiemetic premedication should be administered according to institutional standard of care, published guidelines and the respective product package insert(s).

#### **Corticosteroids:**

- The impact of corticosteroids on the potential efficacy of zolbetuximab is not known. Therefore, consideration should be given to avoid or minimize the use of corticosteroids as a prophylactic antiemetic, if possible.
- For a subject's <u>first dose</u> of zolbetuximab/placebo, it is recommended that the prophylactic use of corticosteroids <u>be avoided</u>.

<sup>\*</sup>To minimize the risk of Torsades de Pointes, administer 5-HT3 receptor blockers with caution to subjects who have or may develop QTc prolongation.

#### 5.1.1.3 CAPOX

Subjects will receive CAPOX treatment until locally confirmed or IRC confirmed disease progression or a total of 8 treatments over 8 or more cycles (each cycle is defined as approximately 3 weeks = approximately 21 days). Oxaliplatin is administered on day 1 of each cycle, whereas capecitabine is taken twice daily on days 1 through 14.

After 8 treatments of CAPOX, subjects may continue to receive capecitabine twice daily on days 1 through 14 of each cycle at the investigator's discretion until the subject meets study treatment discontinuation criteria.

CAPOX should be administered after zolbetuximab/placebo infusion.

- Oxaliplatin: 130 mg/m² intravenous infusion on day 1 of each cycle over 2 hours (or longer per institutional standard of care) for a maximum of 8 treatments. (NOTE: ECG is required to be performed and assessed locally prior to every oxaliplatin infusion [before any antiemetic treatment] and following completion of every oxaliplatin infusion. ECG should be performed up to 48 hours *prior* to and up to 6 hours *following* every oxaliplatin infusion. Oxaliplatin administration and electrolyte levels should be managed according to investigator judgment for subjects with grade 1 or 2 hypokalemia, hypomagnesemia, and/or hypocalcemia.)
- Capecitabine: Administered orally at 1000 mg/m<sup>2</sup> twice daily (bid) (total daily dose is 2000 mg/m<sup>2</sup>) on days 1 through 14 of each cycle. Capecitabine can be continued beyond 8 treatments based on investigator's judgment.
  - When possible, the first dose of Capecitabine on day 1 should be administered on site under the supervision of the site staff.
  - o In case the first dose of Capecitabine on day 1 of a cycle is administered too late in the day for the second dose to be administered on the same day, the last dose of that cycle should be taken in the morning of day 15.
  - o Capecitabine should be taken within 30 minutes after a meal.

Participants who discontinue zolbetuximab and continue to receive CAPOX or components of CAPOX should complete procedures on the study and transition to commercially marketed and locally accessible product(s) (CAPOX or its applicable components).

### 5.1.2 Study Treatment Dose Modifications, Delays And Interruptions

#### 5.1.2.1 Increase or Reduction of zolbetuximab/Placebo

Dose increase or dose reduction for zolbetuximab/placebo is not allowed. Body surface area should be recalculated at minimum if there is a weight change of at least 10% since the last dose calculation.

#### 5.1.2.2 Zolbetuximab/Placebo Interruption or Permanent Discontinuation

There is a +7 calendar day allowable window for dosing zolbetuximab/placebo. If zolbetuximab/placebo treatment is delayed more than 7 calendar days then it should be administered as soon as the reason for delay has resolved, which will then become day 1 of the next cycle. The timing of subsequent doses should be scheduled using the date of the last

06 Dec 2024 Astellas 
dose administration. If zolbetuximab/placebo treatment is delayed, CAPOX/Capecitabine administration should also be delayed at the same time and can be restarted when zolbetuximab/placebo administration has been restarted, unless there are other reasons warranting further delay of CAPOX/Capecitabine at the investigator's discretion (refer to Section 5.1.2.4). Refer to the Pharmacy Manual and Infusion Guidelines for more detailed information on incomplete dosing.

A delay of zolbetuximab/placebo treatment of > 28 days from when the next zolbetuximab/placebo treatment was scheduled to begin (> 49 days from when the last dose of zolbetuximab/placebo began) to be administered due to unresolved toxicity associated with zolbetuximab/placebo will result in the subject discontinuing zolbetuximab/placebo.

Radiologic imaging is to be scheduled every 9 weeks (±7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (±7 days) thereafter; the schedule should be maintained regardless of treatment delay.

Note: Intravenous infusion of zolbetuximab/placebo should be administered as a minimum 2-hour infusion. Intravenous infusion may be interrupted or slowed down to manage toxicity. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information.

Guidelines for zolbetuximab/placebo treatment modification due to non-hematologic and hematologic toxicities, regardless of investigator assessment of relationship to zolbetuximab/placebo, are described below in [Table 2] and [Table 3], respectively.

One case of PRES has been reported in subjects receiving zolbetuximab. **Discontinue zolbetuximab/placebo if PRES is suspected.** Confirm PRES diagnosis by brain imaging, preferably by magnetic resonance imaging (MRI).

Table 2 Guidelines for Zolbetuximab/Placebo Treatment Modification Due to Non-hematologic Toxicity

| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Infusion-related reaction (IRR) other than nausea, vomiting or abdominal pain. See Table 4 for further IRR management guidance | Continue<br>Infusion | Interrupt infusion. Infusion may be resumed at a reduced rate when toxicity has improved to grade ≤ 1. | Stop the infusion immediately. Institute appropriate medical m immediately based on the type Permanently Discontinue zolbe | of reaction. |
| Nausea | Continue Infusion | | Interrupt infusion. Hold zolbetuximab/placebo treatment until toxicity has improved to grade ≤ 1, then restart the infusion at a lower rate. If the investigator determines that the toxicity is not related to zolbetuximab and the toxicity has improved to grade ≤ 2, then infusion may be restarted at the investigator's discretion at a lower rate. | Not applicable* |
| Vomiting | Continue Infusion Continue Infusion Continue Infusion Continue infusion; however, if infusion was held due to grade 3 vomiting, hold infusion until vomiting has improved to ≤ grade 1. | | Interrupt infusion. Hold zolbetuximab/placebo treatment until toxicity has improved to grade ≤ 1 and then restart infusion at a lower rate. | Permanently Discontinue zolbetuximab/ placebo |
| Other Non-<br>hematologic<br>toxicity | Continue Infusion | | Interrupt infusion. Hold zolbetuximab/placebo treatment until toxicity has improved to grade $\leq 1$ . If the investigator determines that the toxicity is not related to zolbetuximab and the toxicity has improved to grade $\leq 2$ , then infusion may be restarted at the investigator's discretion.# | Permanently Discontinue zolbetuximab/ placebo |
| PRES | Discontinue | zolbetuximab/place | bo if PRES is suspected. | |

<sup>\*</sup> Grade 4 nausea is not defined in CTCAE v4.03. If investigator assesses nausea as grade 4, manage per local standard of care.

<sup>#</sup> For subjects with a pulmonary embolism, treatment can continue without resolving to grade 2 or less.

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


Table 3 Guidelines for Zolbetuximab/Placebo Treatment Modification Due to Hematologic Toxicity

| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Neutropenia† | ANC < LLN<br>to 1500/mm <sup>3</sup> ;<br>< LLN to 1.5<br>x 10 <sup>9</sup> /L | ANC < 1500 to<br>1000/mm <sup>3</sup> ;<br>< 1.5 to 1.0 x 10 <sup>9</sup> /L | ANC < 1000 to<br>500/mm <sup>3</sup> ;<br>< 1.0 to 0.5 x 10 <sup>9</sup> /L | ANC < 500/mm <sup>3</sup> ;<br>< 0.5 x 10 <sup>9</sup> /L |
| Action | Continue treatment; however, if treatment was held due to ≥ grade 3 neutropenia, hold treatment until ANC improves to ≤ grade 1. | | Hold treatment and recheck blood counts weekly until ANC resolves to $\geq 1.5 \times 10^9/L$ ( $\leq$ grade 1) before restarting treatment. Discontinue zolbetuximab/placebo if ANC remains $< 1.5 \times 10^9/L$ ( $\geq$ grade 2) after a $> 28$ -day treatment delay from when the next study treatment was scheduled to be administered. | |
| Febrile<br>Neutropenia† | | | ANC < $1000/\text{mm}^3$ with a single temperature of > $38.3^{\circ}\text{C}$ ( $101^{\circ}\text{F}$ ) or a sustained temperature of $\geq 38^{\circ}\text{C}$ ( $100.4^{\circ}\text{F}$ ) for more than 1 hour. | Life-threatening<br>consequences;<br>urgent intervention<br>indicated |
| Action | Not | Applicable | Follow standard/local management guidelines. Hold treatment and recheck blood counts weekly until ANC recovers to ≥ 1.5 x 10 <sup>9</sup> /L (grade ≤ 1) and fever has resolved. Discontinue zolbetuximab/placebo if ANC remains < 1.5 x 10 <sup>9</sup> /L (≥ grade 2) after a > 28-day treatment delay from when the next study treatment was scheduled to be administered. | |
| Thrombocytopenia | PLT < LLN to<br>75,000/mm <sup>3</sup> ;<br>< LLN to<br>75.0 x 10 <sup>9</sup> /L | PLT < 75,000 to<br>50,000/mm <sup>3</sup> ;<br>< 75.0 to 50.0 x<br>10 <sup>9</sup> /L | PLT < 50,000 to<br>25,000/mm <sup>3</sup> ; < 50.0<br>to 25.0 x 10 <sup>9</sup> /L | PLT<br>< 25,000/mm <sup>3</sup> ;<br>< 25.0 x 10 <sup>9</sup> /L |
| Action | Continue<br>treatment | Continue treatment; however, if treatment was held due to grade 3 or higher thrombocytopenia, hold treatment until thrombocytopenia improves to $\leq$ grade 1. | Withhold treatment and counts weekly until pla > 75× 10 <sup>9</sup> /L (grade ≤ 1) treatment. Discontinue zolbetuxim platelets remain < 75 x after a > 28-day treatment the next study treatment be administered. | telets recover to before restarting hab/placebo if 10 <sup>9</sup> /L (grade ≥ 2) ent delay from when |


| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Anemia† | Hgb < LLN to<br>10.0 g/dL;<br>< LLN to<br>6.2 mmol/L;<br>< LLN to<br>100 g/L | Hgb < 10.0 to<br>8.0 g/dL;<br>< 6.2 to 4.9 mmol/L;<br>< 100 to 80 g/L | Hgb < 8.0 g/dL;<br>< 4.9 mmol/L;<br>< 80 g/L;<br>transfusion indicated | Life-threatening<br>consequences;<br>urgent intervention<br>indicated |
| Action | 100 g/L | | Withhold treatment. Follow standard treatment guidelines. Transfuse if indicated. Recheck blood counts weekly until Hgb recovers to > 8.0 g/dL (≤ grade 2) before restarting treatment. Discontinue zolbetuximab/ placebo if Hgb remains < 8.0 g/dL (≥ grade 3) after a > 28-day treatment delay from when the next study treatment was scheduled to be administered. | Withhold treatment. Follow standard treatment guidelines including urgent intervention and blood transfusions as required. The subject may be discontinued after discussion with the Medical Monitor. |

ANC: absolute neutrophil count; LLN: lower limit of normal; PLT: platelet count; Hgb: hemoglobin † At the investigator's discretion growth factors may be used according to standard practice guidelines.

#### 5.1.2.3 Guidelines for Infusion-related Reactions for Zolbetuximab/Placebo

Subjects should be closely monitored for IRRs to facilitate early identification and management.

The management of such toxicities should be based on investigator utilizing institutional standard of care, published guidelines and the general guidelines provided in [Table 4] below.

A subject with an infusion reaction should be evaluated specifically for the symptoms and signs that are highly suggestive of anaphylaxis (urticaria, repetitive cough, wheeze and throat tightness/change in voice). A careful examination of the skin is advised in order to detect urticaria, which often appears first in the neck, trunk, abdomen and axillae.

Not all anaphylactic reactions manifest as anaphylactic shock. Because anaphylaxis can recur and worsen with re-exposure, permanently discontinue zolbetuximab/placebo for any subject having a reaction with features (even if mild) that are highly suggestive of anaphylaxis.

Note: Intravenous infusion of zolbetuximab/placebo should be administered as a minimum 2-hour infusion. Intravenous infusion may be interrupted or slowed down to manage

toxicity. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information.

Table 4 Infusion-related Reactions

| Infusion-Related Reactions | |
|---|---|
| Refer to Table 2 for management | Refer to Table 2 for management of infusion related reactions of nausea, vomiting or abdominal pain |
| CTCAE v4.03 Grade | Management |
| Grade 1 standard infusion reactions other than nausea, vomiting or abdominal pain# | Continue infusion and closely monitor the subject. |
| Grade 2 standard infusion reaction other than nausea, vomiting or abdominal pain# | Interrupt. Medical management as per type of reaction. Resume infusion once toxicity grade ≤ 1 and reduce the infusion rate for the remaining infusion. For the next infusion: Increase total infusion time (reduce infusion rate). Pre-medicate as appropriate.* Closely monitor the subject for symptoms and signs of an infusion reaction. |
| Any infusion reaction with features of anaphylaxis OR Grade 3 or 4 standard infusion reactions other than nausea, vomiting or abdominal pain# | Stop the infusion immediately. Institute appropriate medical management immediately based on the type of reaction. Permanently Discontinue zolbetuximab/placebo Once the subject has been stabilized, collect blood for cytokine/chemokine panel and serum total tryptase level (levels typically peak within 3 hours after the onset of symptoms) and send to the central laboratory. |

CTCAE v4.03: Common Terminology Criteria For Adverse Events

#### 5.1.2.4 CAPOX Dose Modification

The CAPOX dose modifications described below are based on [XELOX CCO Formulary, August 2017].

There is a + 7 calendar day allowable window for CAPOX dosing. If CAPOX treatment is delayed more than 7 calendar days then it should be administered at the next scheduled zolbetuximab/placebo treatment visit, i.e. day 1 of the next cycle. The timing of subsequent doses should be scheduled using the date of the last dose administration.

If Capecitabine treatment is delayed or interrupted, Capecitabine can be administered as soon as the reason for delay or interruption is resolved. The delay/interruption in treatment should be regarded as lost treatment days and missed doses should not be replaced; the planned treatment schedule should be maintained.

<sup>\*</sup> At the investigators discretion, antihistamines may be used as premedication for the next infusion. Systemic corticosteroids should be avoided or minimized while subject is on study treatment unless required for management of an emergent medical condition (e.g., severe nausea/vomiting or hypersensitivity reaction). # For grade 3 or 4 IRR of nausea, vomiting or abdominal pain, collect blood for cytokine/chemokine panel and serum total tryptase level and send to the central laboratory.

Dosing and dose modification should be based on investigator utilizing institutional standard of care, approved package insert, SPC or local product information supplied by the manufacturer for each agent (oxaliplatin, capecitabine) and general guidelines provided below.

The first dose of CAPOX should not be modified. After the assessment of tolerability, dose adjustments should be performed based on investigator judgment utilizing institutional standard of care, approved package insert, SPC, or local product information and/or the recommended criteria in [Table 5] based on maximum hematologic or non-hematologic toxicity data from the previous cycle as shown in [Table 6] and [Table 7], respectively. Dose reduction criteria for oxaliplatin-related neurotoxicity are presented in [Table 8]. Each drug may be dose reduced independently based on the specific types of toxicities observed. It is recommended that no more than 2 dose reductions per drug per subject occur (see [Table 5]). Dose re-escalation is not recommended after treatment-related AEs. Dose re-escalation of capecitabine is permitted after the subject has completed 8 cycles or 8 doses of CAPOX and/or has permanently discontinued oxaliplatin if the investigator chooses to continue capecitabine. If further dose reduction is required beyond the criteria in [Table 5], that component of CAPOX should be discontinued.

In subjects experiencing toxicity requiring a delay or discontinuation of CAPOX, subject should continue to receive zolbetuximab/placebo as clinically appropriate. If CAPOX is interrupted, subject should be evaluated weekly (at a minimum) until the toxicity has improved sufficiently at which time treatment can be restarted as described in the tables below (as applicable). A delay of CAPOX treatment for > 28 days from when the next CAPOX treatment was scheduled to begin (> 49 days from when the last CAPOX dose began) due to unresolved toxicity associated with CAPOX will result in the subject discontinuing CAPOX (both components).

Table 5 Recommended Dose Adjustment Levels for Oxaliplatin and Capecitabine

| Drug | | Oxaliplatin | Capecitabine |
|---|---|---|---|
| Initial Dose | | $130 \text{ mg/m}^2$ | $1000 \text{ mg/m}^2 \text{ bid}$ |
| Dana Badaadkan | Level 1 | $100 \text{ mg/m}^2$ | 750 mg/m² bid |
| Dose Reduction | Level 2 | 75 mg/m <sup>2</sup> | 500 mg/m² bid |

For the first 8 treatments, if a subject has capecitabine discontinued or interrupted, oxaliplatin should be discontinued or interrupted until capecitabine is resumed. For additional information, refer to the approved package insert, SPC or local product information supplied by the manufacturer for each agent (oxaliplatin, capecitabine).

In case Capecitabine administration is delayed or interrupted, the missed doses should not be taken later during the cycle. Capecitabine administration is to be stopped at day 14 (or the morning of day 15 as applicable) of each cycle.

#### 5.1.2.5 CAPOX: Dose Modifications for Hematologic Toxicity

The CAPOX dose modifications for hematologic toxicity are presented in [Table 6]. Dose modifications should be maintained until recovery from hematologic toxicity. A delay of CAPOX treatment for > 28 days from when the next CAPOX treatment was scheduled to begin (> 49 days from when the last CAPOX dose began) due to hematologic toxicity associated with CAPOX will result in the subject discontinuing CAPOX (both components).

Dosing and dose modification should be based on investigator utilizing institutional standard of care, approved package insert, SPC or local product information supplied by the manufacturer for each agent (oxaliplatin, capecitabine) and general guidelines provided below.

Table 6 CAPOX Dose Modification Due to Hematologic Toxicity

| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Neutropenia† | ANC < LLN<br>to 1500/mm <sup>3</sup> ;<br>< LLN to 1.5<br>x 10 <sup>9</sup> /L | ANC < 1500 to<br>1000/mm <sup>3</sup> ; < 1.5<br>to 1.0 x 10 <sup>9</sup> /L | ANC < 1000 to<br>500/mm <sup>3</sup> ;<br>< 1.0 to 0.5 x 10 <sup>9</sup> /L | ANC < 500/mm <sup>3</sup> ;<br>< 0.5 x 10 <sup>9</sup> /L |
| Action | Continue<br>treatment. | CAPOX: 1st, 2nd and 3rd events: Interrupt until event resolves to grade ≤ 1. Fourth event: Discontinue treatment permanently | Hold treatment and rech<br>until ANC resolves to ≥<br>restarting treatment.<br>Discontinue CAPOX if A<br>< 1.5 x 10 <sup>9</sup> /L after a > 20<br>from when the next stud<br>scheduled to be administ | ANC remains<br>8-day treatment delay<br>y treatment was |
| Dose Modification<br>(for next<br>treatment) | Maintain dose<br>level. | Oxaliplatin: Maintain dose of oxaliplatin Capecitabine: First event: Maintain dose level Second event: Reduce capecitabine 1 level.† Third event: Reduce capecitabine 2 levels | Oxaliplatin Dose adjustment next cycle: Reduce 1 dose level Capecitabine Dose adjustment next cycle: First event: Reduce capecitabine 1 level Second event: Reduce capecitabine 2 levels.† Third event: Discontinue CAPOX | Discontinue both. If investigator deems it to be in the subject's best interest to continue, resume next dose of oxaliplatin reduced 1 level and capecitabine reduced 2 dose levels |
| Febrile<br>Neutropenia† | | | ANC < 1000/mm <sup>3</sup><br>with a single<br>temperature of<br>> 38.3°C (101°F) or a<br>sustained temperature | Life-threatening<br>consequences;<br>urgent intervention<br>indicated |

| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| | | | of $\geq$ 38°C (100.4°F)<br>for more than 1 hour. | |
| Action | Maintain dose<br>level | CAPOX: 1st, 2nd and 3rd events: Interrupt until event resolves to grade ≤ 1. Fourth event: Discontinue treatment permanently | Follow standard treatment guidelines | Proceed to next treatment when fever has resolved and ANC recovers to ≥ 1.5 x 10 <sup>9</sup> /L within 28 days from when the next study treatment was scheduled to be administered. |
| Dose Modification<br>(at next treatment) | Maintain dose<br>level | Oxaliplatin: Maintain dose of oxaliplatin Capecitabine: First event: Maintain dose level Second event: Reduce capecitabine 1 level.† Third event: Reduce capecitabine 2 levels | Oxaliplatin Dose adjustment next cycle: Reduce 1 dose level Capecitabine First event: Reduce capecitabine 1 level Second event: Reduce capecitabine 2 levels.† Third event: Discontinue CAPOX | Discontinue both. If physician deems it to be in the patient's best interest to continue, interrupt until resolved to grade 0-1 and resume next dose of oxaliplatin reduced 1 level and capecitabine by reducing 2 dose levels |
| Thrombocytopenia | PLT < LLN<br>to<br>75,000/mm <sup>3</sup> ;<br>< LLN to<br>75.0 x 10 <sup>9</sup> /L | PLT < 75,000 to<br>50,000/mm <sup>3</sup> ;<br>< 75.0 to 50.0 x<br>10 <sup>9</sup> /L | PLT < 50,000 to<br>25,000/mm <sup>3</sup> ; < 50.0 to<br>25.0 x 10 <sup>9</sup> /L | PLT<br>< 25,000/mm <sup>3</sup> ;<br>< 25.0 x 10 <sup>9</sup> /L |
| Action | Continue treatment. | CAPOX: 1 <sup>st</sup> , 2 <sup>nd</sup> and 3 <sup>rd</sup> events: Interrupt until event resolves to grade ≤ 1. Fourth event: Discontinue treatment permanently | Withhold treatment and weekly* until platelets r before restarting treatme if PLT remains < 75 x 1 delay from when the new scheduled to be adminis | ecover to > 75× 10 <sup>9</sup> /L<br>ent. Discontinue CAPOX<br>0 <sup>9</sup> /L after a > 28-day<br>ct study treatment was |


| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Dose Modification<br>(for next<br>treatment) | Maintain dose level. | Oxaliplatin: Maintain dose of oxaliplatin Capecitabine: First event: Maintain dose level Second event: Reduce capecitabine 1 level. Third event: Reduce capecitabine 2 levels | Oxaliplatin Dose adjustment next cycle: Reduce 1 dose level Capecitabine First event: Reduce capecitabine 1 level Second event: Reduce capecitabine 2 levels. Third event: Discontinue CAPOX | Discontinue both. If physician deems it to be in the patient's best interest to continue, interrupt until resolved to grade 0-1 and resume next dose of oxaliplatin reduced 1 level and capecitabine by reducing 2 dose levels |

ANC: absolute neutrophil count; CAPOX: Capecitabine and Oxaliplatin; LLN: lower limit of normal; PLT: platelet count † At the investigator's discretion growth factors may be used according to standard practice guidelines.

#### 5.1.2.6 CAPOX: Dose Modification for Non-hematologic Toxicity

CAPOX dose modifications for non-hematologic toxicity should be based on the most severe toxicity experienced during the last treatment [Table 7]. Retreatment should be delayed until recovery of all non-hematologic toxicity to ≤ grade 2 with the exception of increased bilirubin or ALT, which must recover to grade 1 or baseline, whichever was higher. The maximum permitted treatment delay is 28 days from when the next study treatment was scheduled to begin (49 days from when the last dose of study treatment began) for recovery of non-hematologic toxicity. If the subject has not recovered sufficiently to meet retreatment criteria within that timeframe, CAPOX should be discontinued.

ECG is required to be performed and assessed locally prior to every oxaliplatin infusion (before any antiemetic treatment) and following completion of every oxaliplatin infusion. ECG should be performed up to 48 hours *prior* to and up to 6 hours *following* every oxaliplatin infusion. Ensure that potassium, magnesium, and calcium levels are grade 2 or less prior to oxaliplatin infusion. Oxaliplatin may be administered in the setting of grade 1 or grade 2 hypokalemia, hypomagnesemia, and/or hypocalcemia, based on investigator judgment.

During or following study treatment, additional ECG monitoring should be initiated per local standard of care for subjects who experience syncope, presyncope, palpitations and/or bradycardia.

- If the QTc interval is > 450 msec, medically manage per local standard of care, including correction of hypokalemia, hypomagnesemia, and/or hypocalcemia.
- If the QTc interval is > 500 msec, medically manage per local standard of care, withhold capecitabine and oxaliplatin treatment, ensure appropriate (continuous) ECG monitoring,

<sup>\*</sup> Weekly recheck with ±3 day window for thrombocytopenia

and obtain cardiology consultation. If the QTc interval resolves to  $\leq$  450 msec, the subject may resume treatment at 1 reduced dose level.

Dosing and dose modification should be based on investigator utilizing institutional standard of care, approved package insert, SPC or local product information supplied by the manufacturer for each agent (oxaliplatin, capecitabine) and general guidelines provided below.

Table 7 CAPOX Dose Modification Due to Non-hematologic Toxicity

| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Diarrhea | | | | |
| Action | Continue treatment | Start medical<br>management for<br>diarrhea. Continue<br>treatment. | Start medical managemen<br>Withhold all CAPOX trea<br>treatment after diarrhea re | tment. Restart |
| Dose<br>Modification (for<br>next treatment) | None | First event: None Second event: Reduce capecitabine 1 dose level. | First event: Reduce oxaliplatin 1 level and capecitabine 1 level. Second event: Reduce oxaliplatin 1 dose level and capecitabine 2 levels. | oxaliplatin 1 dose level and |
| Other Non-hemato | ologic Toxicities <sup>†‡</sup> | | | |
| Action | Continue treatment | CAPOX: 1st, 2nd and 3rd events: Interrupt until event resolves to grade ≤ 1 Fourth event: Discontinue treatment permanently | Withhold all CAPOX trea<br>improves to ≤ grade 2. | ntment until toxicity |
| Dose<br>Modification (for<br>next treatment) | None | Oxaliplatin: Maintain dose of oxaliplatin Capecitabine: First event: Maintain dose level Second event: Reduce capecitabine 1 level.† Third event: Reduce capecitabine 2 levels | Oxaliplatin Dose adjustment next cycle: Reduce 1 dose level Capecitabine First event: Reduce capecitabine 1 level Second event: Reduce capecitabine 2 levels.† Third event: Discontinue CAPOX | Discontinue both If physician deems it to be in the patient's best interest to continue, interrupt until resolved to grade 0-1 and resume next dose of oxaliplatin reduced 1 level and capecitabine by reducing 2 dose levels |

CAPOX: Capecitabine and Oxaliplatin

<sup>†</sup> For skin toxicity, reduce capecitabine only, not oxaliplatin.

<sup>‡</sup> Exceptions: alopecia, fatigue, anorexia, nausea/vomiting (if can be controlled by antiemetics) and constipation (if can be controlled with laxatives, stool softeners, etc.).

#### 5.1.2.7 Guidelines for Infusion-related Reactions for Oxaliplatin

Subjects should be closely monitored for IRRs to facilitate early identification and management. The management of such toxicities should be based on investigator utilizing institutional standard of care.

#### **5.1.2.8** Oxaliplatin-induced Neurotoxicity

Oxaliplatin is known to be associated with peripheral neuropathy, including paresthesia and dysesthesia of the hands, feet and perioral region. Subjects treated with oxaliplatin in this study should be advised to avoid cold drinks and exposure to cold water or air, especially within 3 to 5 days of receiving oxaliplatin. Dose modifications for oxaliplatin related to neurotoxicity are presented in [Table 8].

Cases of PRES have been reported in subjects receiving Oxaliplatin combination chemotherapy. Discontinue Oxaliplatin if PRES is suspected. Confirm PRES diagnosis by brain imaging, preferably by MRI.

Table 8 Oxaliplatin Dose Modification for Associated Neurotoxicity

| Toxicity/Duration | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Paresthesia or dysesthesia | Paresthesia or<br>dysesthesia‡<br>that does not<br>interfere with<br>function | Paresthesia or<br>dysesthesia‡,<br>interfering with<br>function, but<br>not activities of<br>daily living | Paresthesia or<br>dysesthesia‡ with<br>pain or with<br>functional<br>impairment that<br>also interferes<br>with activities of<br>daily living | Persistent<br>paresthesia or<br>dysesthesia that<br>is disabling or<br>life-threatening |
| 1 to 7 Days > 7 Days | No dose<br>reduction | No dose<br>reduction | First Event: Reduce oxaliplatin by 1 dose level at next treatment. Second Event: Reduce oxaliplatin by a second dose level at next treatment. For Grade 3 neurotoxicity > 7 days/persistent between treatments, discuss oxaliplatin discontinuation with Medical Monitor. | Discontinue<br>oxaliplatin |
| Persistent between treatments† | | Reduce<br>oxaliplatin by<br>1 dose level at<br>next treatment | For Grade 3 neurotoxicity > 7 days/persistent between treatments, discuss oxaliplatin discontinuation with Medical Monitor | |
| Acute laryngopharyngeal | Discontinue curi | | ı | |
| dysesthesia‡ | | | ment with benzodiaze | pines and |
| (during or after the 2-hour | At next treatment, consider pretreatment with benzodiazepines and increasing duration of infusion as clinically indicated per investigator | | | |
| infusion) | discretion. | | | |

NA: not applicable

#### 5.1.2.9 Oxaliplatin-induced Laryngopharyngeal Dysesthesia

Oxaliplatin has also been associated with laryngopharyngeal dysesthesia, which is an unusual loss of sensation of breathing (acute respiratory distress) without any objective evidence of respiratory distress (hypoxia, laryngospasm or bronchospasm). Laryngopharyngeal dysesthesia may be induced or exacerbated upon exposure to cold.

<sup>†</sup> Not resolved by the beginning of the next treatment.

<sup>‡</sup> May be cold induced.

Subjects developing laryngopharyngeal dysesthesia should have their oxygen saturation evaluated via a pulse oximeter. If results are normal, reassurance should be provided, a benzodiazepine or other anxiolytic agent should be considered, and the subject should remain for observation in the clinic until the episode has resolved. After resolution, the oxaliplatin infusion may then be continued at one-third the rate.

Because laryngopharyngeal dysesthesia may be associated with the rate of oxaliplatin infusion, subsequent infusions of oxaliplatin should be prolonged from a normal 2-hour infusion to a 6-hour infusion.

Subjects receiving oxaliplatin should avoid consuming cold drinks or ice chips on day 1 of each cycle, as this may exacerbate oral or throat dysesthesia, as well as laryngopharyngeal dysesthesia. Administration of prophylactic medication such as Mg<sup>2+</sup>/Ca<sup>2+</sup> infusions or others is at the discretion of the investigator.

The symptoms and treatments of laryngopharyngeal dysesthesia and platinum HSRs are compared in [Table 9].

Table 9 Comparison of the Symptoms and Treatment of Laryngopharyngeal Dysesthesia and Platinum Hypersensitivity Reactions

| Clinical Symptoms | Laryngopharyngeal Dysesthesia | Platinum Hypersensitivity |
|---|---|---|
| Dyspnea | Present | Present |
| Bronchospasm | Absent | Present |
| Laryngospasm | Absent | Present |
| Anxiety | Present | Present |
| O <sub>2</sub> saturation | Normal | Decreased |
| Difficulty swallowing | Present (loss of sensation) | Absent |
| Pruritus | Absent | Present |
| Urticaria/rash | Absent | Present |
| Cold-induced symptoms | Yes | No |
| Blood pressure | Normal or increased | Normal or decreased |
| Treatment | Reassurance, anxiolytics, observation in a controlled clinical setting until symptoms abate or at the physician's discretion | Oxygen, steroids, epinephrine,<br>bronchodilators; fluids and<br>vasopressors, if appropriate |

#### **5.1.2.10** Allergic Reaction to Oxaliplatin

Subjects developing grade 1 or 2 allergic reaction to oxaliplatin should receive premedication according to institutional practice prior to further administration of oxaliplatin. Appropriate premedication should also be given if grade 1 to 2 allergic reaction persists into the next cycle. Oxaliplatin should be discontinued in subjects developing grade 3 to 4 allergic reactions.

Oxaliplatin should be interrupted pending further investigation in subjects experiencing respiratory symptoms indicative of pulmonary fibrosis such as nonproductive cough, dyspnea, crackles, rales, hypoxia, tachypnea or radiological pulmonary infiltrates. Oxaliplatin should be permanently discontinued in subjects with confirmed interstitial pulmonary fibrosis.

#### 5.1.2.11 Extravasation of Oxaliplatin

Necrosis has been seen in conjunction with extravasation of oxaliplatin. Subjects with suspected extravasation should have their infusion stopped and the drug administered at another site. Extravasation should be treated according to institutional guidelines.

#### **5.1.3** Treatment Compliance

The dose and schedule of zolbetuximab/placebo and CAPOX administered to each subject will be recorded on the appropriate eCRF at every cycle. Reasons for dose delay or omission will also be recorded. This information will be used to assess compliance with the treatment. Subjects will be provided with Capecitabine tablets for self-administration and are asked to return any unused tablets and empty packaging at the next scheduled visit for accountability.

#### 5.1.4 Criteria for Continuation of Treatment

Zolbetuximab may be made available after conclusion of the study to subjects who are still receiving and benefitting from study treatment until a study-defined treatment discontinuation criterion is met.

Once the product is commercially marketed and locally accessible, participants should complete the study, transition to commercial supply and follow the local label for treatment.

Astellas is planning to close the clinical study when zolbetuximab (Vyloy) is commercially marketed in all countries with active participants and all participants have successfully transitioned to an alternative means of drug supply.

## 5.1.4.1 Discontinuation of CAPOX (both components) and Continuation of Zolbetuximab/Placebo

If a subject discontinues CAPOX (or either component of CAPOX) due to any reason other than locally confirmed or IRC confirmed disease progression, they may continue on zolbetuximab/placebo at the discretion of the investigator and until zolbetuximab is commercially marketed and locally accessible, provided that all of the following have been met:

- the subject completed at least 2 treatments of CAPOX treatment;
- the subject will not receive another systemic chemotherapy, immunotherapy, radiotherapy or other treatment intended for antitumor activity; and
- in the investigator's opinion the subject continues to derive clinical benefit with acceptable toxicity.

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), radiological disease progression will be determined locally and subjects should continue to follow the Study Treatment Period Schedule of Assessments [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) radiological disease progression was determined by IRC and subjects followed the Study Treatment Period Schedule of Assessments [Table 1].

## **5.1.4.2** Discontinuation of Zolbetuximab/Placebo and Continuation of CAPOX (One or Both Components)

If zolbetuximab/placebo is permanently discontinued first for reasons other than PD as confirmed locally or by IRC and no other anticancer treatment is started, subjects may continue to receive CAPOX/Capecitabine until treatment discontinuation criteria are met. Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), radiological disease progression will be determined locally and subjects should continue to follow the Study Treatment Period Schedule of Assessments [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), radiological disease progression was determined by IRC and subjects followed the Study Treatment Period Schedule of Assessments [Table 1].

Participants who discontinue zolbetuximab and continue to receive CAPOX or components of CAPOX should complete procedures on the study and transition to commercially marketed and locally accessible product(s) (CAPOX or its applicable components).

## 5.1.4.3 If Both Zolbetuximab/Placebo and CAPOX (Both Components) are Discontinued

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), if both zolbetuximab/placebo and CAPOX (both components) are discontinued for reasons other than locally or IRC confirmed radiological PD, the subject should enter 30-day safety follow up and continue to undergo imaging assessments per Schedule of Assessments [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1),

if both zolbetuximab/placebo and CAPOX (both components) are permanently discontinued for reasons other than IRC-confirmed radiological PD, the subject should enter the Post-Treatment Follow-up Period and continue to undergo imaging assessments per Schedule of Assessments [Table 1].

# 5.1.5 Previous and Concomitant Treatment (Medication and Non-Medication Therapy)

All medications and concomitant treatments administered from the time of full main informed consent through the 90-day safety follow-up visit must be recorded in the eCRF. Documentation will include the medication name, indication, route and dates of administration.

#### **Prohibited Concomitant Treatment**

The following are strictly prohibited:

- Sorivudine or analogs (during capecitabine treatment)
- Concurrent non-steroid systemic immunosuppressive agents (for systemic corticosteroids, see cautionary concomitant treatment below).
- Live vaccines should be avoided during the treatment period in which subject is receiving oxaliplatin or capecitabine and up to 6 months after final oxaliplatin or

capecitabine dose. In cases where a live vaccine is needed for COVID-19 prevention and allowed per local regulations, please contact the Medical Monitor for discussion.

- Other systemic chemotherapy, immunotherapy, radiotherapy, herbal medications or other treatments intended for antitumor activity.
  - Palliative radiotherapy for peripheral bone metastases is allowed.
  - For gastric bleeding, palliative radiotherapy is prohibited, but esophagogastroduodenoscopy with epinephrine injection is allowed.
- Investigational products or therapy other than zolbetuximab.

#### **Cautionary Concomitant Treatment**

Considerations should be given to avoid or minimize the use of the following concomitant medications, if possible, during <u>zolbetuximab/placebo</u> treatment:

- Systemic corticosteroids, because their impact on the potential efficacy of zolbetuximab is not known.
  - Systemic corticosteroids should be avoided or minimized while subject is on study treatment unless required for management of an emergent medical condition (e.g., severe nausea/vomiting or hypersensitivity reaction).
  - o For a subject's <u>first dose</u> of zolbetuximab/placebo, it is recommended that the prophylactic use of corticosteroids <u>be avoided</u>.
  - o Inhaled, intranasal, ophthalmic, otic and topically applied steroids are allowed.
  - Subjects are allowed to use a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg/day of hydrocortisone or up to 10 mg/day of prednisone), receive a single dose of systemic corticosteroids or receive systemic corticosteroids as pre-medication for radiologic imaging contrast use.
- Administer 5-HT3 blockers with caution in subjects who have or may develop QTc prolongation.
- Nonsteroidal anti-inflammatory drugs (NSAIDs) because of the potential to cause gastric ulcers and covert bleeding.
  - In such cases where NSAID use is necessary, the use of NSAIDs with lower gastric ulcerogenic potential is preferred and concomitant gastric protection with proton pump inhibitors is recommended.

The following should be avoided or used with caution and closely monitored during capecitabine administration:

- Cytochrome P450 2C9 substrates (Subjects taking coumarin-derivative anticoagulants concomitantly with capecitabine should have PT/INR monitored regularly and anticoagulant dose adjusted accordingly).
- Anti-epileptic medications (e.g., phenobarbital, phenytoin and primidone)

The following should be avoided or used with caution and closely monitored during oxaliplatin administration:

 Medications known to prolong the QT or QTc interval (refer to https://www.crediblemeds.org for a list of these medications Prohibited and cautionary treatments are described in Appendix 12.4.

## **5.2** Demographics and Baseline Characteristics

## 5.2.1 Demographics

Demographic information will be collected for all subjects and will include initials (where permitted), age, date of birth (where permitted), sex, race (where permitted) and ethnicity (where permitted).

#### **5.2.2 Medical History**

Medical history includes all significant medical conditions per the judgment of the investigator that have resolved prior to informed consent or are ongoing at the time of full main consent. Details that will be collected include the onset date and recovery date and CTCAE v4.03 grade, if applicable for ongoing conditions.

#### 5.2.3 Diagnosis of the Target Disease, Severity, and Duration of Disease

A complete medical history of the target disease will be recorded during Screening. This will include the subject's medical condition, date of initial diagnosis, tumor location, and other disease specific information as designated in the eCRF.

## 5.3 Efficacy Assessments

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), radiologic imaging will be evaluated locally [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), radiographic imaging was evaluated centrally by IRC.

Radiologic imaging will be evaluated at Screening (within 28 days prior to randomization) and every 9 weeks (±7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (±7 days) thereafter until subject develops radiological disease progression per RECIST 1.1 by local confirmation or IRC confirmation or starts other systemic anticancer treatment, whichever comes earlier.

All radiologically-evaluable disease (measurable and/or non-measurable), per local assessment, must be documented at Screening and re-assessed at each subsequent radiologic evaluation. Imaging will include CT scans with contrast of the thorax, abdomen, and pelvis. If CT scan with contrast is medically not feasible, MRI may be used for imaging. Bone scans (or focal X-ray) or brain imaging should be performed if metastatic disease in bone or brain is suspected, respectively. The same mode of imaging should be utilized throughout the study unless medical necessity requires a change. For randomized subjects, screening imaging should be sent to the central imaging vendor no later than at the time of submission of the first on-treatment imaging. All imaging acquired post randomization will be sent to the local or central imaging vendor within 7 days of scanning for the blinded IRC assessment of radiological tumor response based on RECIST 1.1 [Eisenhauer et al, 2009]. The investigator should make every effort to immediately submit radiologic assessments for IRC review when

PD is suspected. Refer to Imaging Acquisition Guidelines for further detail on scan modality and contrast options.

### 5.4 Safety Assessment

#### 5.4.1 Vital Signs

Vital signs, including systolic and diastolic blood pressures (mmHg) and radial pulse rate (beats/minute) and temperature, will be obtained and recorded at the times specified in the Schedule of Assessments [Table 1]. All vital sign measurements will be obtained in a consistent manner (sitting or supine) throughout their study participation. Height and weight will be measured using normal institutional standards.

If clinically significant vital sign changes from baseline (pretreatment) are noted, the changes will be documented as AEs on the AE page of the eCRF. Clinical significance will be defined as a variation in vital signs, which has medical relevance as deemed by the investigator that could result in an alteration in medical care. For clinically significant vital sign changes, the investigator will continue to monitor the subject until the parameter returns to grade  $\leq 1$ , or to the baseline (pretreatment) value, or until the investigator determines that follow up is no longer medically necessary.

#### 5.4.2 Observation Period Following Zolbetuximab/Placebo Infusion

Following the first dose of zolbetuximab/placebo on C1D1, the subject must be observed for 2 hours post zolbetuximab/placebo infusion. The post-infusion observation period can be conducted during the CAPOX administration. If  $\geq$  grade 2 AEs are observed during infusion or during the post-infusion observation period, subsequent zolbetuximab/placebo infusion times should be extended and subjects should continue to be observed for 2 hours post zolbetuximab/placebo infusion. If the subject does not develop any  $\geq$  grade 2 AEs, the subject should be observed for 1 hour post-infusion for their subsequent zolbetuximab/placebo infusions. The subject should be instructed to notify site personnel if they develop any AEs during this post-infusion observation time period.

In the event of an IRR with features of anaphylaxis (regardless of grade) or grade 3 or 4 IRR, blood samples for cytokine/chemokine panel and serum total tryptase level (levels typically peak within 3 hours after the onset of symptoms) should be collected once the subject has stabilized, for shipment to the central laboratory.

#### 5.4.3 Laboratory Assessments

Below is a table of the laboratory tests that will be performed during the conduct of the study.

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), laboratory tests will be performed according to the Schedule of Assessments [Table 11] and must be sent to the local laboratory for analysis.

Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), laboratory tests will be performed according to the Schedule of Assessments [Table 1] and must be sent to the central laboratory for analysis.

- Eligibility can be determined based on central and/or local laboratory testing:
  - O The most recent laboratory data must be used to confirm the subject's eligibility. In the case of multiple sample collections within 14 days prior to randomization, the most recent sample collection with available results should be used to determine eligibility.
  - Central labs must be collected and submitted to the central laboratory during the Screening period.
  - If retesting of lab values is necessary to confirm eligibility, local labs can be used without requiring additional sample collection for central laboratory submission.
  - The screening labs used to determine eligibility should be collected within 14 days prior to randomization.
- Laboratory test results (central or local) will be reviewed by the investigator prior to any study treatment. Clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician.
- Local laboratory results may be used for treatment decisions; however, central laboratory samples must also be drawn per protocol and sent to the central laboratory. (*UNIQUE TO CHINA*: Local laboratory results may be used for treatment decisions; however, central laboratory samples should also be drawn per protocol and sent to the central laboratory unless otherwise approved by the sponsor.)
- Central and local labs may be collected up to 48 hours prior to study treatment.
- Holidays and weekends should be taken into account when scheduling these sample collections.
- Additional assessments may be done centrally or locally to monitor AEs or as clinically indicated.

| Panel/Assessment | Parameters to be Analyzed |
|------------------|--------------------------------------------------|
| Hematology | Hematocrit (Hct) |
| | Hemoglobin (Hgb) |
| | Red Blood Cell Count (RBC) |
| | White Blood Cell Count (WBC) |
| | WBC differential |
| | Absolute Neutrophil Count (ANC) |
| | Platelets |
| | Mean Corpuscular Volume (MCV) |
| | Mean Corpuscular Hemoglobin (MCH) |
| | Mean Corpuscular Hemoglobin Concentration (MCHC) |
| Biochemistry | Albumin |
| | Blood Urea Nitrogen (BUN) |
| | Calcium |
| | Bicarbonate |
| | Chloride |

| Creatinine Glucose Magnesium Phosphate Potassium Sodium Total Bilirubin Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Cytokine/Chemokine Panel† Serum total tryptase† Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid simulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | Panel/Assessment | Parameters to be Analyzed |
|---|---|---|
| Magnesium Phosphate Potassium Sodium Total Bilirubin Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Human chorionic gonadotropin (HCG) | | Creatinine |
| Phosphate Potassium Sodium Total Bilirubin Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Serum total tryptase† Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Glucose |
| Potassium Sodium Total Bilirubin Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (IPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Human chorionic gonadotropin (HCG) | | Magnesium |
| Sodium Total Bilirubin Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Phosphate |
| Total Bilirubin Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Cytokine/Chemokine Panel† Serum total tryptase† Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Potassium |
| Total Protein Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (IPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Sodium |
| Alanine Aminotransferase (ALT) Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Human chorionic gonadotropin (HCG) | | Total Bilirubin |
| Alkaline Phosphatase (ALP) Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Total Protein |
| Aspartate Aminotransferase (AST) Creatinine Clearance Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Alanine Aminotransferase (ALT) |
| Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Alkaline Phosphatase (ALP) |
| Grade 3 or 4 Infusion-related Reactions (IRR) Cytokine/Chemokine Panel† Serum total tryptase† Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Aspartate Aminotransferase (AST) |
| Any reaction with features of anaphylaxis Scrum total tryptase† Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thrombop Test Human chorionic gonadotropin (HCG) | | Creatinine Clearance |
| Any reaction with features of anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Cytokine/Chemokine Panel† |
| anaphylaxis Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | (IRR) | Serum total tryptase† |
| Dihydropyrimidine dehydrogenase (DPD) deficiency screening† Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test DPD deficiency alleles DPD deficiency alleles POPD deficiency alleles DPD deficiency alleles POPD deficiency alleles DPD deficiency alleles POPD deficiency alleles Potherial type Human chorionic gonadotropin (HCG) | Any reaction with features of | Cytokine/Chemokine Panel† |
| Urinalysis Color Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Serum total tryptase† |
| Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | DPD deficiency alleles |
| Clarity/turbidity pH Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | Urinalysis | Color |
| Specific gravity Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Clarity/turbidity |
| Glucose Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | |
| Ketones Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Specific gravity |
| Nitrites Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Glucose |
| Leukocyte esterase Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Ketones |
| Bilirubin Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Nitrites |
| Urobilinogen Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Leukocyte esterase |
| Blood Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Bilirubin |
| Protein RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Urobilinogen |
| RBCs WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Blood |
| WBCs Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Protein |
| Coagulation Prothrombin time (PT) (sec) Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | RBCs |
| Partial Thromboplastin Time (PTT) International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | WBCs |
| International normalized ratio (INR) Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | Coagulation | Prothrombin time (PT) (sec) |
| Thyroid Function Test Thyroid stimulating hormone (TSH) Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | Partial Thromboplastin Time (PTT) |
| Free T4 (thyroxine) Urine Pregnancy Test Human chorionic gonadotropin (HCG) | | International normalized ratio (INR) |
| Urine Pregnancy Test Human chorionic gonadotropin (HCG) | Thyroid Function Test | Thyroid stimulating hormone (TSH) |
| | | Free T4 (thyroxine) |
| Serum Pregnancy Test Human chorionic gonadotropin (HCG) | Urine Pregnancy Test | Human chorionic gonadotropin (HCG) |
| | Serum Pregnancy Test | Human chorionic gonadotropin (HCG) |

<sup>†</sup> As applicable

#### 5.4.4 Physical Examination

Physical examinations will be conducted at visits as outlined in the Schedule of Assessments [Table 1]. Each physical exam should include height (at Screening only), weight and ECOG performance status. A full physical exam is required at Screening. The physical exam only needs to be repeated on C1D1 if clinically significant changes from Screening are observed (in the opinion of the investigator). For all cycles, the physical examination, weight and ECOG performance status assessments can be completed up to 48 hours prior to zolbetuximab/placebo administration. Targeted (symptom driven) physical exams should be conducted every 3 weeks on day 1 of each cycle. If clinically significant worsening of findings from baseline is noted at any study visit, the changes will be documented as AEs on the AE eCRF. Clinical significance is defined as any variation in physical findings, which has medical relevance that could result in an alteration in medical care. The investigator will continue to monitor the subject until the parameter returns to grade  $\leq 1$ , or to the baseline condition, or until the investigator determines that follow up is no longer medically necessary.

## 5.4.5 Electrocardiogram

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), a single 12-lead ECG will be performed at the time points outlined in the Schedule of Assessments [Table 11].

Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), a single 12-lead ECG will be performed at the time points outlined in the Schedule of Assessments [Table 1]. Prior to performing ECG, subjects should rest in supine position for 10 minutes. When collected on the same day, ECG should be collected prior to pharmacokinetic samples. Additional ECG may be performed based on medical history and investigator medical judgment. ECGs will be assessed locally. Clinically significant findings should be recorded as an AE.

#### 5.4.6 Performance Status

The ECOG Scale [Oken et al, 1982] will be used to assess performance status. Refer to [Appendix 12.8].

## 5.5 Adverse Events and Other Safety Aspects

AE collection will begin from time of full main informed consent and continue through the 90 days following the last dose of zolbetuximab/placebo and CAPOX (both components).

Serious adverse events (SAEs), regardless of causality will be collected from the time of full main informed consent through 90 days following the last dose of zolbetuximab/placebo and CAPOX (both components). If a participant transitions to commercially marketed zolbetuximab or CAPOX and has discontinued from the study, the 30- and 90-day safety follow up visits are not required.

Once participants have transitioned to commercially marketed zolbetuximab, safety assessment and reporting should continue as per post-marketing product requirements.

06 Dec 2024 Astellas 

AEs will be documented at each clinic visit, but can be collected at any time. Any AE that meets the definition of an SAE will also be reported on a separate form to the sponsor.

#### **5.5.1** Definition of Adverse Events

An AE is any untoward medical occurrence in a subject administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.

In order to identify any events that may be associated with study procedures and could lead to a change in the conduct of the study, Astellas collects AEs even if the subject has not received study drug treatment. AE collection begins after the signing of the full main informed consent and will be collected until 90 days after the last dose of study drug or the subject is determined to be a screen failure.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the subject is the preferred method to inquire about AE occurrences.

#### 5.5.1.1 Abnormal Laboratory Findings

Any abnormal laboratory test result (e.g., hematology, clinical chemistry or urinalysis) or other safety assessment (e.g., ECGs, radiology scans, vital signs measurements, physical examination), including those that worsen from baseline, that is considered to be clinically significant in the medical and scientific judgment of the investigator and not related to underlying disease, is to be reported as an (S)AE.

Any clinically significant abnormal laboratory finding or other abnormal safety assessment which is associated with the underlying disease does not require reporting as an (S)AE, unless judged by the investigator to be more severe than expected for the subject's condition.

Repeating an abnormal laboratory test or other safety assessment, in the absence of any of the above criteria, does not constitute an AE. Any abnormal test result that is determined to be an error does not require reporting as an AE.

#### 5.5.1.2 Potential Cases of Drug-Induced Liver Injury

Refer to [Appendix 12.5 Liver Safety Monitoring and Assessment] for detailed instructions on drug induced liver injury. Abnormal values in AST and/or ALT concurrent or with abnormal elevations in total bilirubin that meet the criteria outlined in [Appendix 12.5 Liver Safety Monitoring and Assessment] in the absence of other causes of liver injury, are considered potential cases of drug-induced liver injury (potential Hy's Law cases) and are always to be considered important medical events and reported per [Section 5.5.5 Reporting of Serious Adverse Events].

#### 5.5.1.3 Disease Progression and Study Endpoints

Under this protocol, the following event(s) will not be considered as an (S)AE:

- Disease Progression: events including defined study endpoints that are clearly consistent with the expected pattern of progression of the underlying disease are <u>not to</u> be recorded as AEs unless resulting in death. These data will be captured as efficacy assessment data as outlined in [Section 5.3 Efficacy Assessments]. If there is any uncertainty as to whether an event is due to anticipated disease progression and/or if there is evidence suggesting a causal relationship between the study treatment and the event, it should be reported as an (S)AE. All deaths up to 90 days after the last dose of study drug must be reported as an SAE, even if attributed to disease progression.
- Disease progression can be considered as the worsening of a subject's condition attributable to Gastric or GEJ cancer. It may be an increase in the severity of the disease under study and/or increases in the symptoms of the disease. The development of new, or progression of existing metastases to the primary cancer under study should be considered as disease progression not an AE. Events which are unequivocally due to disease progression should not be reported as an AE during the study.

#### **5.5.2** Definition of Serious Adverse Events

An AE is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Results in death
- Results in life-threatening event (an AE is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death)
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly, or birth defect
- Requires inpatient hospitalization (except for planned procedures as allowed per study) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE). Hospitalization for treatment/observation/examination caused by AE is to be considered as serious.
- Other medically important events (defined in paragraph below)

Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above. These events, including those that may result in disability/incapacity, usually are considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

#### 5.5.2.1 Important Medical Events

If an AE occurs that the sponsor determines to be an Important Medical Event, additional information on the event (e.g., investigator confirmation of seriousness, causality) will be requested.

Progression of Gastric or GEJ cancer, including signs and symptoms of progression, should not be reported as an SAE unless it results in death within 90 days of the last dose of study treatment. For progression-related death reported as an SAE, there should be available immediate cause of death reported as the event term. "Death due to disease progression" should be recorded as the AE term only when the cause of death cannot be otherwise determined

#### 5.5.3 Criteria for Causal Relationship to Study Treatment

A medically qualified investigator is obligated to assess the relationship between each study treatment and each occurrence of each (S)AE. This medically qualified investigator will use medical judgment as well as the RSI [Section 1.3] to determine the relationship. The causality assessment is 1 of the criteria used when determining regulatory reporting requirements. The medically qualified investigator is requested to provide an explanation for the causality assessment for each (S)AE and must document in the medical notes that he/she has reviewed the (S)AE and has provided an assessment of causality.

Following a review of the relevant data, the causal relationship between the study treatment and each (S)AE will be assessed by answering 'yes' or 'no' to the question "Do you consider that there is a reasonable possibility that the event may have been caused by the study treatment".

When making an assessment of causality, the following factors are to be considered when deciding if there is evidence and/or arguments to suggest there is a 'reasonable possibility' that an (S)AE may have been caused by the study treatment (rather than a relationship cannot be ruled out) or if there is evidence to reasonably deny a causal relationship:

- Plausible temporal relationship between exposure to the study treatment and (S)AE onset and/or resolution. Has the subject actually received the study treatment? Did the (S)AE occur in a reasonable temporal relationship to the administration of the study treatment?
- Plausibility; i.e., could the event have been caused by the study treatment? Consider biologic and/or pharmacologic mechanism, half-life, literature evidence, drug class, preclinical and clinical study data, etc.
- Dechallenge/Dose reduction/Rechallenge:
  - Did the (S)AE resolve or improve after stopping or reducing the dose of the suspect drug? Also consider the impact of treatment for the event when evaluating a dechallenge experience.
  - Did the (S)AE reoccur if the suspected drug was reintroduced after having been stopped?

- Laboratory or other test results; a specific lab investigation supports the assessment of the relationship between the (S)AE and the study treatment (e.g., based on values pre, during and post-treatment)
- Available alternative explanations independent of study treatment exposure; such as
  other concomitant drugs, past medical history, concurrent or underlying disease, risk
  factors including medical and family history, season, location, etc. and strength of the
  alternative explanation

There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the medically qualified investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor. With limited or insufficient information about the event to make an informed medical judgment and in absence of any indication or evidence to establish a causal relationship, a causality assessment of 'no' is to be considered. In such instance, the investigator is expected to obtain additional information regarding the event as soon as possible and to re-evaluate the causality upon receipt of additional information. The medically qualified investigator may revise his/her assessment of causality in light of new information regarding the SAE and shall send an SAE follow-up report and update the eCRF with the new information and updated causality assessment.

## 5.5.4 Criteria for Defining the Severity of an Adverse Event

AEs, including abnormal clinical laboratory values, will be graded using the NCI-CTCAE v4.03 guidelines. The items that are not stipulated in the NCI-CTCAE v4.03 will be assessed according to the criteria below and entered into the eCRF.

| Grade | Assessment Standard |
|---|---|
| 1-Mild | Asymptomatic or mild symptoms, clinical or diagnostic observations noted; intervention not indicated. |
| 2-Moderate | Local or noninvasive intervention indicated. |
| 3-Severe | Medically significant but not immediately life threatening, hospitalization or prolonged hospitalization. |
| 4-Life Threatening | Life threatening consequences, urgent intervention indicated |
| 5-Death | Death related to AE |

#### **5.5.5** Reporting of Serious Adverse Events

The collection of AEs and the expedited reporting of SAEs will start following receipt of the signed full main informed consent and will continue until 90 days after the last dose of study treatment or the subject is determined to be a screen failure. Once patients have transitioned to commercially marketed zolbetuximab, safety assessment and reporting should continue as per post-marketing product requirements.

In the case of a SAE, the investigator must contact the sponsor by fax or email immediately (within 24 hours of awareness).

The investigator must complete and submit an SAE worksheet containing all information that is required by local and/or regional regulations to the sponsor by email or fax immediately (within 24 hours of awareness).

The SAE worksheet must be signed by a medically qualified investigator (as identified on Delegation of Authority Log). Signature confirms accuracy and completeness of the SAE data as well as the investigator causality assessment including the explanation for the causality assessment.

If the SAE is associated with emergency unblinding as outlined in [Section 4.7.4 Breaking the Blind in Emergency] this is to be recorded on the SAE worksheet. Within the SAE worksheet, the investigator is to include when unblinding took place in association with the SAE.

JAPAN SITES ONLY: In the case of a SAE, the investigator or sub-investigator must report to the head of the study site and must contact the sponsor by email or fax immediately (within 24 hours of awareness). The investigator should complete and submit JUTOKUNA YUUGAIJISHOU HOUKOKUSHO containing all information that is required by the Regulatory Authorities to the sponsor by email or fax immediately (within 24 hours of awareness) and to the head of the hospital.

After marketing authorization in Japan, the sponsor collects all AEs and the following special situations in accordance with Good Post-marketing Study Practice.

- Drug Exposure During Pregnancy
- Drug Exposure via Breast Milk
- Lack of Efficacy
- Medication Error
- Abuse, Misuse, Overdose
- Off-Label Use
- Occupational Exposure
- Drug-Drug Interaction
- Unexpected Benefit

For contact details, see [Section II] Contact Details of Key Sponsor's Personnel. Fax or email the SAE and Special Situations Worksheet to:

Astellas Pharma Global Development, Inc.
Pharmacovigilance
North American Fax: +1-888-396-3750
(North America Alternate Fax: +1-847-317-1241)

International Fax: +44-800-471-5263 Email: safety-us@us.astellas.com

# **UNIQUE TO JAPAN REGION**: JUTOKUNA YUUGAIJISHOU HOUKOKUSHO the SAE and Special Situations Worksheet to:

PAREXEL International Fax number: 03-6888-5798

If there are any questions, or if clarification is needed regarding the SAE, please contact the sponsor's Medical Monitor/Study Physician or his/her designee [Section II] Contact Details of Key Sponsor's Personnel.

Follow-up information for the event should be sent promptly (within 7 days of the initial notification (*UNIQUE TO JAPAN REGION*: within 2 days for the initial notification).

Full details of the SAE or Special Situation should be recorded on the medical records, SAE or Special Situation Worksheet and on the (e)CRF.

The following minimum information is required:

- International Study Number (ISN)/Study number,
- Subject number, sex and age,
- The date of report,
- A description of the SAE (event, seriousness criteria),
- Causal relationship to the study treatment (including reason), and
- The drug provided (if any). Note: blinded regimen is also an option.

The sponsor or sponsor's designee will medically evaluate the SAE and determine if the report meets the requirements for expedited reporting based on seriousness, causality, and expectedness of the events (e.g., SUSAR reporting) according to current local/regional regulatory requirements in participating countries. The sponsor or sponsor's designee will submit expedited safety reports (e.g., Investigational New Drug [IND] Safety Reports, SUSAR, Council for International Organizations of Medical Sciences I Form) to Competent Authorities and concerned Ethics Committee per current local regulations, and will inform the investigators of such regulatory reports as required. Investigators must submit safety reports as required by their IRB/local IEC within timelines set by regional regulations (e.g., EMA, FDA) where required. Documentation of the submission to and receipt by the IRB/local IEC of expedited safety reports should be retained by the study site.

The sponsor will notify all investigators responsible for ongoing clinical studies with the study treatment of all SUSARs which require submission per local requirements IRB/local IEC/ head of the study site (as applicable).

The heads of the study sites (if applicable) and investigators should provide written documentation of IRB/IEC notification for each report to the sponsor.

#### 5.5.6 Follow-up of Adverse Events

All AEs occurring during or after the subject has discontinued the study are to be followed up until resolved or judged to be no longer clinically significant, or until they become chronic to the extent that they can be fully characterized by the investigator.

If after the protocol defined AE collection period [see Section 5.5.1 Definition of Adverse Event], an AE progresses to an SAE, or the investigator learns of any (S)AE including death, where he/she considers there is reasonable possibility it is related to the study treatment or study participation, the investigator must promptly notify the sponsor. Once patients have transitioned to commercially marketed zolbetuximab, safety assessment and reporting should continue as per post-marketing product requirements.

#### 5.5.7 Monitoring of Common Serious Adverse Events

Common SAEs are SAEs commonly anticipated to occur in the study population independent of drug exposure. SAEs classified as "common" are provided in [Appendix 12.6 Common Serious Adverse Events] for reference. The list does NOT change the investigator's reporting obligations, nor his obligations to perform a causality assessment, or prevent the need to report an AE meeting the definition of an SAE as detailed above. The purpose of this list is to alert the investigator that some events reported as SAEs may not require expedited reporting to the regulatory authorities based on the classification of "common SAEs" as specified in [Appendix 12.6 Common Serious Adverse Events]. The sponsor will monitor these events throughout the course of the study for any change in frequency. Any changes to this list will be communicated to the participating investigational sites. Investigators must report individual occurrences of these events as stated in [Section 5.5.5 Reporting of Serious Adverse Events].

#### **5.5.8** Adverse Events of Special Interest

In case of zolbetuximab induced nausea, vomiting or hypersensitivity/IRR, infusion rate of zolbetuximab/placebo may be reduced or infusion paused or discontinued based on investigator's clinical judgment about severity of toxicity and local standard of care. See [Section 5.1.2 Study Treatment Dose Modifications, Delays and Interruptions] and the Pharmacy Manual and Infusion Guidelines.

If the AEs of interest are classified as serious, they are to be collected via the SAE worksheet and reported within 24 hours as described in [Section 5.5.5 Reporting of Serious Adverse Events].

#### **5.5.9** Special Situations

Certain Special Situations observed in association with the study treatment(s), such as incorrect administration (e.g., wrong dose of study treatment, comparator or background therapy) are collected in the eCRF, as Protocol Deviations per [Section 8.2 Major Protocol Deviations] or may require special reporting, as described below. These Special Situations are not considered AEs, but do require to be communicated to Astellas as per the timelines defined below.

If a Special Situation is associated with, or results in, an AE, the AE is to be assessed separately from the Special Situation and captured as an AE in the eCRF. If the AE meets the definition of a SAE, the SAE is to be reported as described in [Section 5.5.5 Reporting of Serious Adverse Events] and the details of the associated Special Situation are to be included in the clinical description on the Special Situation worksheet.

06 Dec 2024 Astellas 

#### The Special Situations are:

- Pregnancy
- Medication error, Overdose and "Off label use"
- Misuse/abuse
- Occupational exposure
- (Suspicion of) Transmission of infectious agent
- Suspected Drug-Drug interaction

#### 5.5.9.1 Pregnancy

If a female subject becomes pregnant during the study dosing period or within 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs, or if a partner of a male subject becomes pregnant during the study dosing period or within 6 months from the discontinuation of dosing, the investigator is to report the information to the sponsor according to the timelines in [Section 5.5.5 Reporting of Serious Adverse Events] using the Pregnancy Reporting Form and in the eCRF.

The expected date of delivery or expected date of the end of the pregnancy, last menstruation, estimated conception date, pregnancy result and neonatal data etc., should be included in this information.

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or termination (including elective termination) of a pregnancy is to be reported for a female study subject as an AE in the eCRF or SAE per [Section 5.5.5 Reporting of Serious Adverse Events]. For (S)AEs experienced by a female partner of a male subject, (S)AEs are to be reported via the Pregnancy Reporting Form.

Additional information regarding the outcome of a pregnancy when also categorized as an SAE is mentioned below:

- "Spontaneous abortion" includes miscarriage, abortion and missed abortion.
- Death of a newborn or infant within 1 month after birth is to be reported as an SAE regardless of its relationship with the study drug.
- If an infant dies more than 1 month after the birth, is to be reported if a relationship between the death and intrauterine exposure to the study drug is judged as "possible" by the investigator.
- Congenital anomaly (including anomaly in miscarried fetus)

Unless a congenital anomaly is identified prior to spontaneous abortion or miscarriage, the embryo or fetus should be assessed for congenital defects by visual examination. (S)AEs experienced by the newborn/infant should be reported via the Pregnancy Reporting Form. Generally, follow up will be no longer than 6 to 8 weeks following the estimated delivery date.

#### 5.5.9.2 Medication Error, Overdose and "Off-Label Use"

If a Medication Error, Overdose or "Off-label Use" (i.e., use outside of what is stated in the protocol) is suspected, refer to [Section 8.2 Major Protocol Deviations]. Any associated

06 Dec 2024 Astellas 

(S)AEs are to be reported in the eCRF. If the AE meets the definition of a SAE, the SAE is also to be reported as described in [Section 5.5.5 Reporting of Serious Adverse Events] together with the details of the medication error, overdose and/or "Off-Label Use".

There is no antidote for overdose of the study drug. In the event of suspected zolbetuximab overdose, the subject should receive supportive care and monitoring (including, but not limited to, inpatient hospitalization). The Medical Monitor should be contacted as applicable.

In the event of suspected CAPOX overdose, refer to the approved package insert, SPC or local product information supplied by the manufacturer for each agent.

## 5.5.9.3 Misuse/Abuse

If misuse or abuse of the study drug(s) is suspected, the investigator must forward the Special Situation worksheet to the sponsor/delegated contract research organization (CRO) by fax or email immediately (within 24 hours of awareness). Any associated (S)AEs are to be reported in the eCRF. If the AE meets the definition of a SAE, the SAE is also to be reported as described in [Section 5.5.5 Reporting of Serious Adverse Events] together with details of the misuse or abuse of the study drug(s).

#### 5.5.9.4 Occupational Exposure

If occupational exposure (e.g., inadvertent exposure to the study drug(s) of site staff whilst preparing it for administration to the subject) to the study drug(s) occurs, the investigator must forward the Special Situation worksheet to the sponsor/delegated CRO by fax or email immediately (within 24 hours of awareness). Any associated (S)AEs occurring to the individual associated with or resulting from the Special Situation are to be reported on the Special Situations worksheet.

#### 5.5.9.5 Suspected Drug-Drug Interaction

If a suspected drug-drug interaction associated with the study drug(s) is suspected, the investigator must forward the Special Situation worksheet to the sponsor/delegated CRO by fax or email immediately (within 24 hours of awareness). Any associated (S)AEs are to be reported in the eCRF. If the AE meets the definition of a SAE, the SAE is also to be reported as described in [Section 5.5.5 Reporting of Serious Adverse Events] together with details of the suspected drug-drug interaction.

## 5.5.10 Supply of New Information Affecting the Conduct of the Study

When new information becomes available necessary for conducting the clinical study properly, the sponsor will inform all investigators involved in the clinical study as well as the regulatory authorities. Investigators should inform the IRB/IEC of such information when needed.

The investigator will also inform the subjects, who will be required to sign an updated ICF in order to continue in the clinical study.

#### UNIQUE TO JAPAN REGION:

- 1. When information is obtained regarding serious and unexpected adverse drug reactions (or other) that are specified in Article 273 of the Act on Securing Quality, Efficacy and Safety of Pharmaceuticals, Medical Devices, Regenerative and Cellular Therapy Products, Gene Therapy Products, and Cosmetics, in compliance with Article 80-2 Paragraph 6 of the Pharmaceutical Affairs Law, the sponsor should inform all the investigators involved in the clinical study, the head of the study site, and the regulatory authorities of such information. The head of the study site who receives such information will decide whether the clinical study should be continued after hearing the opinions of the IRB. The investigator will supply the new information to the subjects, in compliance with [Appendix 12.1.4.2 Supply of New and Important Information Influencing the Subject's Consent and Revision of the Written Information].
- 2. In addition to the above item (1), when the head of the study site receives the revisions of the IB, protocol or written information, information on the matters covering the quality of the study drug, efficacy and safety, information necessary for conducting the clinical study properly, or documents to be examined by the IRB these documents should be sent to the IRB.

#### 5.5.11 Urgent Safety Measures

An Urgent Safety Measure (USM) is an intervention, which is not defined by the protocol and can be put in place with immediate effect without needing to gain prior approval by the sponsor, relevant Competent Authorities, IRB/IEC, where applicable, in order to protect study participants from any immediate hazard to their health and/or safety. Either the investigator or the sponsor can initiate a USM. The cause of a USM can be safety, product or procedure related.

## 5.5.12 Reporting Urgent Safety Measures

In the event of a potential USM, the investigator must contact the Astellas Study Physician and/or – unique for JP region – Astellas team member (within 24 hrs of awareness). Full details of the potential USM are to be recorded in the subject's medical records. The sponsor may request additional information related to the event to support their evaluation.

If the event is confirmed to be an USM the sponsor will take appropriate action to ensure the safety and welfare of the patients. These actions may include but are not limited to a change in study procedures or study treatment, halting further enrollment in the study, or stopping the study in its entirety. The sponsor or sponsor's designee will notify CA and cEC within the timelines required per current local regulations, and will inform the investigators as required. When required, investigators must notify their IRB/IEC within timelines set by regional regulations.

## 5.6 Test Drug Concentration

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), pharmacokinetic sampling will no longer be collected at the 30-Day Safety Follow-up visit or 90-Day Follow-up visit; see the Schedule of Assessments in [Table 11] in [Section 13].

Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), pharmacokinetic sampling will be conducted as outlined in [Table 1]. Serum concentrations of zolbetuximab will be measured. Samples will be collected as outlined in the Schedule of Assessments [Table 1]. Blood sampling, processing, storage and shipment instructions will be provided in the Laboratory Manual. Samples will be shipped to and analyzed by a sponsor-designated analytical laboratory using validated analytical methods. Please refer to the Laboratory Manual for more detailed information.

Samples remaining after pharmacokinetic assessments may be used for additional biomarker analysis described in [Section 5.7.1 Biomarkers].

## 5.7 Other Measurements, Assessments or Methods

#### 5.7.1 Biomarkers

Tumor tissue and blood/serum/plasma samples described in [Sections 5.7.2 Blood/Serum/ Plasma Samples and 5.7.3 Tumor Tissue Samples] may be used for research purposes as allowed per local policy to identify genomic and/or other biomarkers that may be associated with clinical outcome or dynamic changes associated with zolbetuximab treatment (in terms of dose, safety, tolerability and efficacy). Since the identification of exploratory biomarkers that correlate with the efficacy or safety of zolbetuximab treatment may continue to evolve as new findings becomes available, additional analyses related to zolbetuximab activity on tumor signaling pathways or clinical outcomes may be conducted as allowed per local policy. Tumor tissue and blood/serum samples remaining after the specified biomarker assessments (e.g., aliquots of tumor cell RNA or DNA) may be used for re-testing, additional analyses as defined above or developing, and validating assays related to prediction of response or dynamic changes associated with zolbetuximab treatment. The tumor tissue and blood/serum/plasma samples (e.g., aliquots of tumor cell RNA or DNA, peripheral blood mononuclear cells) will be stored at the study sponsors' facility or a contract laboratory facility for up to 15 years after database closure, at which time the samples will be destroyed. The procedures for the collection, handling and shipping of laboratory samples being submitted to the local or central laboratory will be specified in a laboratory manual.

## 5.7.2 Blood, Serum and Plasma Samples

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), blood, serum and plasma samples will be collected as allowed per local policy according to the Schedule of Assessments [Table 11]. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), blood, serum and plasma samples will be collected as allowed per local policy according to the Schedule of Assessments [Table 1] for exploratory biomarker measurements. Blood, serum and plasma samples may be analyzed for

biomarkers including but not limited to chemokines, cytokines, CDC activation, circulating DNA soluble factors and genetic markers.

#### **5.7.3** Tumor Tissue Samples

FFPE tumor tissue samples will be obtained for all subjects and sent for central IHC testing to evaluate for CLDN18.2, and HER2 status if a previously documented HER2 test result is not available. (*UNIQUE FOR CHINA*: FFPE tumor tissue samples will be obtained for all subjects and sent for central IHC testing to evaluate for CLDN18.2 status.) Tissue from the primary site is preferred, however, if a metastatic site is used (excluding bone metastasis), the sample should be gastric or GEJ in origin. Archival tumor tissue is preferred, but if the specimen is insufficient or unavailable, a biopsy may be performed to obtain a primary tumor tissue or tumor tissue from metastatic site (excluding bone metastasis). Sponsor preapproval is required when a biopsy procedure is needed for the sole purpose of determining study eligibility. Optional post-progression tumor tissue sample for exploratory biomarker analysis may be collected as allowed per local policy following local or IRC confirmation of disease progression and prior to initiation of subsequent anticancer therapy for subjects who sign a separate ICF. Tumor specimens may be analyzed for exploratory biomarkers including but not limited to CLDN18.2 expression, immune cells, genetic markers and gene/protein expression, as allowed per local policy.

The investigator, in consultation with other specialists, as needed (e.g., radiology staff) will assess the risk associated with obtaining a tumor tissue sample and determine if the subject is an appropriate candidate for the procedure. Biopsies should be obtained in accordance with institutional policies/guidelines to minimize risk. Procedures requiring general anesthesia should not be performed to obtain a tumor tissue sample; however, if a surgical procedure under general anesthesia is performed for a clinical indication, excess tumor tissue may be used for research purposes with the consent of the subject.

(UNIQUE TO CHINA: The tumor tissue will be stored at the study sponsor's facility or at a contract laboratory facility for up to 10 years after study completion, at which time the samples will be destroyed, as allowed per local policy. The procedures for the collection, handling and shipping of tissue samples being submitted to the central laboratory will be specified in a laboratory manual.)

#### **Tumor Tissue Requirements**

| Visit | Tumor Tissue Requirement |
|---|---|
| Screening | A minimum of 1 FFPE tumor tissue block (preferred) OR a minimum* of 15 FFPE unstained slides are required as allowed per local policy. If local HER2 results are available, a minimum* of 12 slides are required along with the pathology report/documented test results. If local HER2 results are unavailable, follow guidance above. (UNIQUE TO CHINA: Five FFPE unstained slides are required, as allowed per local policy. The slides should be freshly cut from the FFPE block within |
| | the time frame described in the laboratory manual.) |
| Post-Progression (optional) | A minimum of 1 FFPE tumor tissue block (preferred) OR a minimum* of 15 FFPE unstained slides are required as allowed per local policy. |
| | ( <i>UNIQUE TO CHINA</i> : Optional post-progression tumor sample is not applicable for China.) |

FFPE: formalin-fixed paraffin embedded; HER2: human epidermal growth factor receptor 2

#### 5.7.4 Immunogenicity Assessment (Anti-drug Antibody)

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), serum samples to assess the formation of ADAs against zolbetuximab will be collected as outlined in the Schedule of Assessments [Table 11].

Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), serum samples to assess the formation of anti-drug antibodies (ADAs) against zolbetuximab will be collected as outlined in the Schedule of Assessments [Table 1]. Blood sampling, processing, storage and shipment instructions will be provided in the Laboratory Manual. Samples will be shipped to and analyzed by a sponsor designated analytical laboratory using validated analytical methods. Please refer to the Laboratory Manual for more detailed information.

(*UNIQUE TO CHINA*: Exploratory biomarker testing will not be performed on samples from subjects in China.)

Samples remaining after immunogenicity assessments may be used for additional biomarker analysis as allowed per local policy and as described in [Section 5.7.1 Biomarkers].

#### 5.7.5 Optional Samples for Banked Pharmacogenomics Sample Analysis

For subjects who signed a separate ICF, an optional whole blood sample for pharmacogenomics (PGx) will be collected at C1D1 prior to first study drug administration, as allowed per local policy. PGx research may be conducted in the future to analyze or determine genes of relevance to clinical response, pharmacokinetics and toxicity/safety issues. A sample of whole blood for possible retrospective PGx analysis will be collected and processed as allowed per local policy. Blood sampling, processing, storage and shipment instructions will be provided in the Laboratory Manual. Samples will be shipped to a sponsor-designated analytical storage laboratory. Please refer to the Laboratory Manual for more detailed information.

<sup>\*</sup>If the required minimum number of slides is not able to be submitted, sponsor notification and approval is required.

(*UNIQUE TO CHINA*: Exploratory biomarker testing will not be performed on samples from subjects in China.)

See [Appendix 12.7 Pharmacogenomic Analysis With Banked Sample] for further details on the banking procedures.

#### **5.7.6** Electronic Clinical Outcome Assessments

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), all eCOAs are discontinued as outlined in the Schedule of Assessments [Table 11].

Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), subjects will be asked to complete HRQoL and HRU questionnaires as specified in the Schedule of Assessments [Table 1]. The electronic Clinical Outcomes Assessment (eCOA) questionnaires should be completed by the subject at Screening (except for HRU), day 1 of each cycle (or up to 48 hours) before any antiemetic or drug treatment and before the disease status is discussed with the subject using the electronic device provided. When completion by the subject is not possible, the questionnaires may be administered to the subject by site personnel using the electronic tablet device. For subjects with low literacy or situations where required translation is not available, please contact the sponsor for further guidance. Assessments will also be collected at study treatment discontinuation and 30 and 90 days post zolbetuximab/placebo treatment. HRQoL and HRU questionnaires are not required at CAPOX dosing visits (if different from zolbetuximab/placebo dosing visit), CAPOX treatment discontinuation, 30 day safety follow-up and 90 day safety follow-up visits. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day and HRQoL and HRU questionnaires will be required at those combined visits. HRQoL will be measured by EORTC QLQ-C30, QLQ-OG25 plus STO22 Belching subscale, GP and the EQ5D-5L.

(*UNIQUE TO CHINA*: Genomic testing will not be performed on samples from subjects in China.)

#### 5.7.6.1 Quality of Life Questionnaire C30

The EORTC-QLQ-C30 is a 30-item cancer-specific instrument consisting of 5 functional scales (physical, role, emotional, social and cognitive), 9 symptom scales/items (fatigue, nausea/vomiting, general pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) and a global health status scale. For functional scales, higher scores indicate better functioning, while for symptom scales/items, higher scores indicate worse symptoms.

#### 5.7.6.2 Oesophago-Gastric Module 25 plus STO22 Belching Subscale

The EORTC QLQ-OG25 questionnaire is a 25-item instrument that evaluates gastric and GEJ cancer-specific symptoms. This module consists of 6 scales: dysphagia (3 items), eating restrictions (4 items), reflux (2 items), odynophagia (2 items), pain and discomfort (2 items) and anxiety (2 items), as well as 10 single items: eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with

coughing, trouble talking, weight loss and hair loss. For symptom scales/items, higher scores indicate worse symptoms. To ensure relevant symptoms are adequately covered, 2 items from the EORTC-QLQ-STO22 instrument related to belching and bile or acid coming in mouth will be asked following the EORTC QLQ-OG25 questionnaire.

#### 5.7.6.3 Global Pain

The GP instrument is a single assessment of overall pain.

#### 5.7.6.4 EuroQOL Five Dimensions Questionnaire

The EQ-5D-5L is a standardized instrument for use as a measure of health outcome consisting of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale for health status.

#### 5.7.6.5 Health Resource Utilization

The HRU questionnaire is used to assess the number of office visits, hospital stays, and other healthcare resource utilization that occur outside of the clinical study.

#### 5.8 Total Amount of Blood

The total amount of blood collected for study assessments for each subject will vary depending on how long they stay on treatment.

At any time during the study, if any laboratory abnormalities are found for a subject or for disease assessment, additional blood may be drawn for monitoring.

Additional blood beyond standard monitoring that will be drawn for this study will include draws for eligibility assessment, hematology, chemistry, and coagulation at specific study-defined time points, pharmacokinetics, and biomarker sampling.

The maximum amount of blood collected is approximately 40 mL in cycle 1, and less in later cycles.

(UNIQUE TO CHINA: The maximum amount of blood collected is approximately 10 mL at screening, and less in subsequent cycles.)

#### 6 DISCONTINUATION

## 6.1 Discontinuation of Individual Subject(s) From Study Treatment

A subject who enrolled in the study and for whom study treatment (zolbetuximab/placebo and <u>both</u> components of CAPOX) is permanently discontinued for any reason will be assessed as having met study treatment discontinuation criteria.

As overall survival is the key secondary end-point of the study, all subjects will be followed for survival after meeting study treatment discontinuation criteria unless the subject withdraws consent or is considered lost to follow-up after repeated attempts to contact or if the sponsor discontinues the study. The reason for discontinuation from study treatment must be documented in the subject's medical records.
A subject is free to withdraw from the study treatment and/or study for any reason and at any time without giving reason for doing so and without penalty or prejudice. The investigator is also free to terminate a subject's involvement in the study at any time if the subject's clinical condition warrants it. The subject will be discontinued from study treatment (zolbetuximab/placebo and both components of CAPOX) if any of the following occur:

- Investigator determines it is in the subject's best interest to discontinue study treatment
- Subject develops radiological disease progression per RECIST 1.1 criteria based on assessment locally or by IRC.
  - o If the investigator believes that the subject is continuing to derive clinical benefit (asymptomatic and/or without worsening of performance status or overall health) from study treatment, and an increase in tumor burden is not likely to affect vital organ function, the subject may remain on study treatment until an additional radiologic assessment is completed (≤ 9 weeks from previous radiologic assessment).
    - If the additional radiologic assessment locally or by IRC indicates PD per RECIST 1.1, then the subject must be discontinued from study treatment.
    - If the additional radiologic assessment locally or by IRC does not confirm the initial assessment of PD, the subject may continue to receive study treatment.
- Subject develops clinical progression per investigator assessment and radiologic assessment is not medically feasible to confirm radiologic progression due to the subject's condition.
- Subject starts another systemic chemotherapy, immunotherapy, radiotherapy or other treatment intended for antitumor activity.
- Subject starts another investigational agent or device.
- Subject develops unacceptable toxicity.
- Subject has a delay of zolbetuximab/placebo <u>and</u> both components of CAPOX treatment for > 28 days from when the next zolbetuximab/placebo <u>and</u> both components of CAPOX treatment was scheduled to begin (> 49 days from when the last dose of zolbetuximab/placebo and both components of CAPOX treatment began).
- Any clinical AE, laboratory abnormality, or inter-current illness, in the opinion of the investigator, indicates continued treatment is not in the best interest of the subject
- Female subject becomes pregnant.
- Significant deviation from the protocol or eligibility criteria as determined by the sponsor.
- Subject declines further treatment.
- Subject is lost to follow-up despite reasonable efforts by the investigator to locate the subject.
- Subject is noncompliant with the protocol based on investigator or Medical Monitor assessment.

Note, if a subject discontinues both components of CAPOX and zolbetuximab/placebo due to any reason other than locally confirmed or IRC confirmed disease progression (and is not

receiving any other anticancer therapy), the subject must be followed according to the protocol-specified radiologic assessment schedule until radiological disease progression per RECIST 1.1 criteria is confirmed locally or by IRC assessment.

## **Study Discontinuation Criteria**

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), the Post Treatment Follow-up Period (for PFS) is discontinued with radiological disease progression determined locally; see the Schedule of Assessments [Table 11] in [Section 13].

Participation in the study will end when subjects transition to the commercially marketed and locally accessible product (zolbetuximab and/or CAPOX).

Subjects that completed the 90-Day Safety Follow up Visit(s) treatment period under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1) were eligible for the Post-Treatment Follow up Period (for PFS) and were to remain in the study through the Survival Follow-up Period (OS is a key secondary study endpoint). A subject will be discontinued from the Post-treatment, Long-term and Survival Follow-up Periods if any of the following occur:

- Subject specifically withdraws consent for any further contact with him/her or persons previously authorized by the participant to provide this information
- Subject is lost to follow-up despite reasonable efforts by the investigator to locate the subject
- Death (from any cause)
- Study termination by the sponsor

## 6.1.1 Lost to Follow Up

Every reasonable effort is to be made to contact any subject lost to follow-up during the course of the study to complete study-related assessments, record outstanding data, and retrieve study drug.

## 6.2 Discontinuation of the Site

If an investigator intends to discontinue participation in the study, the investigator must immediately inform the sponsor and, **SPECIFIC TO SITES IN JAPAN**, the head of the study site must also be informed immediately.

# 6.3 Discontinuation of the Study

If the study is prematurely terminated or suspended the sponsor or designee shall promptly inform the investigators, the IECs/IRBs, the regulatory authorities, and any contract research organization(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements.

The study may also be terminated if it is not possible for the sponsor to make a necessary adjustment to the maximum insurance sum as required by local law/regulation.

In case of premature study termination, zolbetuximab may be made available to subjects who are still receiving and benefitting from study treatment until a study-defined treatment discontinuation criterion is met.

Astellas is planning to close the study when zolbetuximab (Vyloy) is commercially marketed in all countries with active participants.

## 7 STATISTICAL METHODOLOGY

A statistical analysis plan (SAP) will be written to provide details of the analysis, along with specifications for tables, listings and figures to be produced The final SAP will be approved prior to database hardlock and unblinding the subject treatment assignment. Changes that affected the statistical analyses from the planned analyses in the SAP will be documented in the Clinical Study Report (CSR).

In general, continuous data will be summarized with descriptive statistics (number of subjects, mean, standard deviation, minimum, median and maximum) for continuous variables, and frequency and percentage for categorical variables.

Baseline will be defined as the last observation prior to first dose, unless otherwise specified.

# 7.1 Sample Size

Approximately 500 subjects will be randomized in a 1:1 ratio to receive zolbetuximab in combination with CAPOX chemotherapy (Arm A) or placebo in combination with CAPOX chemotherapy (Arm B). The planned 300 PFS events during the study will provide 93.4% power to detect a difference in PFS between Arm A (zolbetuximab+CAPOX) with the assumption of 9 months median PFS time and Arm B (placebo+CAPOX) with the assumption of 6 months median PFS time (hazard ratio = 0.67) at the overall 1-sided 0.025 significance level. Similarly, the planned 386 OS events during the study will provide 80% power to detect a difference in OS between Arm A (zolbetuximab+CAPOX) with the assumption of 14.7 months median survival time and Arm B (placebo+CAPOX) with the assumption of 11 months median OS time (hazard ratio = 0.75) at the overall 1-sided 0.025 significance level.

# 7.2 Analysis Sets

The allocation of subjects to analysis sets will be determined prior to database hard-lock. For each treatment group, the number and percentage of subjects will be characterized for all randomized subjects and by each analysis set.

## 7.2.1 Full Analysis Set

The full analysis set (FAS) will consist of all subjects who are randomized to 1 of the treatment arms. Subjects would be analyzed according to the treatment they were randomized to. The FAS would be used for description of baseline characteristics and all efficacy analyses.

## 7.2.2 Safety Analysis Set

The safety analysis set (SAF) will consist of all subjects who received at least 1 dose of any study drug (zolbetuximab/placebo/CAPOX). The SAF will be used for all safety analyses. Subjects would be analyzed according to the actual treatment they received.

## 7.2.3 Pharmacokinetic Analysis Set (PKAS)

The pharmacokinetic analysis set (PKAS) consists of the subset of the SAF for which at least 1 concentration data is available. Additional subjects may be excluded from the PKAS at the discretion of the pharmacokineticist. The PKAS would be used for description of pharmacokinetic data.

## 7.3 Demographics and Baseline Characteristics

Demographics and other baseline characteristics will be summarized by treatment group and overall for FAS and SAF.

## 7.3.1 Subject Disposition

The number and percentage of subjects who discontinued treatment and reasons for treatment discontinuation will be presented for FAS by treatment group and overall. Similar tables for subjects who do not have a PFS event and subjects who do not have observed death will also be presented. All disposition details and dates of first and last evaluations for each subject will be listed.

### 7.3.2 Previous and Concomitant Medications

All previous and concomitant medications will be presented in a listing. The frequency of concomitant medications (prescription, over-the-counter, and nutritional supplements) will be summarized. Any component of CAPOX is not considered concomitant medications.

## 7.3.3 Medical History

Medical history for each subject will be presented in a listing and summarized.

# 7.4 Analysis of Efficacy

Efficacy analysis will be conducted on the FAS. The interpretation of results from statistical tests will be primarily based on the FAS. All randomized subjects will be analyzed according to the treatment to which they are randomized.

## 7.4.1 Analysis of Primary Endpoint

## 7.4.1.1 Primary Analysis

The primary endpoint is PFS assessed by the blinded IRC. For each subject, PFS is defined as the time from the date of randomization until the date of radiological disease progression (i.e., PFS) assessed by IRC, or until death due to any cause, whichever is earlier. If a subject has neither progressed nor died, the subject will be censored at the date of last radiological assessment. Subjects who receive new anticancer therapy before radiological progression will be censored at the date of the last radiological assessment before the new anticancer therapy

started. If progression or death occurs after missing 2 or more scheduled radiological assessments, the subject will be censored at the date of last radiological assessment or at the date of randomization if no post-baseline radiological assessment is available.

The primary analysis will be performed when approximately 300 PFS events have been observed.

The distribution of PFS will be estimated for each treatment arm using Kaplan-Meier methodology and compared between Arm A and Arm B using log-rank test stratified by:

- Region (Asia vs Non-Asia)
- Number of Organs with Metastatic Sites (0 to 2 vs  $\geq$  3)
- Prior Gastrectomy (Yes or No)

The hypothesis testing on the primary analysis will be performed at an overall 1-sided 0.025 significance level to test the null hypothesis that PFS is not prolonged in Arm A compared to Arm B versus the alternative hypothesis that PFS is prolonged in Arm A compared to Arm B.

In addition, stratified Cox proportional hazard model will be used to estimate the hazard ratio and the corresponding 95% CI.

The primary analysis will be performed using the FAS.

## 7.4.1.2 Sensitivity Analysis

Sensitivity analyses with different censoring rules will be described in the SAP.

## 7.4.1.3 Subgroup Analysis

The analysis described in [Section 7.4.1.1 Primary Analysis] will be conducted in the subgroups using the FAS. Subgroups defined by baseline factors will be described in the SAP.

Forest plot will be presented to illustrate the strength of treatment effects across subgroups.

## 7.4.2 Analysis of Secondary Endpoints

## 7.4.2.1 Overall Survival

A key secondary endpoint OS is defined as the time from the date of randomization until the documented date of death from any cause. All events of death will be included, regardless of whether the event occurred while the subject is still taking study drug or after the subject discontinue study drug. Subjects who are still alive at the time of analysis will be censored at the last day known to be alive.

The distribution of OS will be estimated for each treatment arm using Kaplan-Meier methodology and compared between Arm A and Arm B using the log-rank test stratified by the same stratification factors used for PFS analysis. To maintain the overall Type I error rate at the 0.025 significance level, the hypothesis testing on OS will be performed only if the null hypothesis on the primary analysis is rejected at the overall 1-sided 0.025 significance level. In addition, stratified Cox proportional hazard model will be used to estimate the hazard ratio and the corresponding 95% CI.

## 7.4.2.2 PF, OG25-Pain, and GHS/QoL Scores

A key secondary endpoint, TTCD, is defined for the following 3 HRQoL domains: physical functioning (PF) and Global Health Status/Quality of Life (GHS/QoL) as collected in the EORTC QLQ-C30, and abdominal pain and discomfort (OG25-Pain) as collected in the EORTC QLQ-OG25 plus STO22). TTCD is defined as the time from the date of randomization until the date of first clinically meaningful deterioration that is confirmed at a next scheduled assessment or followed by drop-out resulting in missing data.

Clinically meaningful deterioration will be defined if a subject's change from baseline exceeds a pre-specified threshold denoting a clinically meaningful change. While clinically meaningful thresholds have been derived for EORTC QLQ-30 for some domains (e.g., 10 for GHS/QoL in Osoba 1998), an appropriate threshold for this population and for all domains of interest will be derived using the study's data. A separate analysis plan will be developed where methods for the estimation of the clinically meaningful threshold will be defined in detail and signed off before database lock. The execution of these analysis and derivation of the threshold value to be used in the TTCD analysis will also be performed before database lock, and the resulting value will be inserted in the clinical SAP in a last amendment again before the study is unblinded.

Subjects who did not experience a confirmed deterioration will be censored at the last eCOA assessment. Subjects who have no baseline or post-baseline assessment, or are not able to show deterioration due to their baseline value will be censored at randomization. For example, if a subject has a baseline GHS/QoL value of 5 and the clinically meaningful threshold proves to be 8, then this subject will be censored at baseline. Death or disease progression will not be considered as an event.

Similarly to PFS and OS endpoints, the distribution of TTCD will be estimated for each treatment arm using Kaplan-Meier methodology and compared between Arm A and Arm B using the log-rank test stratified by the same stratification factors used for PFS and OS analysis. To maintain the overall Type I error rate at the 0.025 significance level, the hypothesis testing on TTCD will be performed only if the null hypothesis on the OS is rejected at the overall 1-sided 0.025 significance level. Specifically, if the null hypothesis on the OS is rejected at the overall 1-sided 0.025 significance level, then the TTCD will be tested using the gatekeeping procedure with the following order:

- 1. Non-inferiority testing for TTCD in PF at 0.025 significance level
- 2. Non-inferiority testing for TTCD in OG25-Pain at 0.025 significance level
- 3. Non-inferiority testing for TTCD in GHS/QoL at 0.025 significance level
- 4. Superiority testing for TTCD in PF at 0.025 significance level
- 5. Superiority testing for TTCD in OG25-Pain at 0.025 significance level
- 6. Superiority testing for TTCD in GHS/QoL at 0.025 significance level

A stratified Cox proportional hazard model will be used to estimate the hazard ratio and the corresponding 95% CI for the three time-to-event eCOA endpoints.

## 7.4.2.3 Objective Response Rate

Best overall response (BOR) is determined once all tumor response data for the subject is available. Subjects will be classified by BOR on study as outlined in RECIST 1.1 criteria. For BOR of SD, SD must be documented as present at least once after study entry and at least 8 weeks after first dose.

The ORR is defined as the proportion of subjects with a BOR of CR or PR based on IRC per RECIST V1.1.

The comparison of ORR between Arm A and Arm B will be performed using stratified Cochran-Mantel-Haenszel (CMH) test with the same stratification factor used for the PFS analysis. In addition, ORR for each arm will be estimated and corresponding 95% CI will be constructed.

In addition, percent of subjects with CR will be summarized.

## 7.4.2.4 **Duration of Response**

DOR is defined as the time from the date of the first response of CR or PR (whichever is first recorded) as assessed by IRC to the date of radiological progression or death, whichever is earlier. If a subject has not progressed, the subject will be censored at the date of last radiological assessment or at the date of first CR/PR if no post-baseline radiological assessment is available. Other censoring used for the PFS analysis will apply to DOR too.

The distribution of DOR will be estimated for each treatment arm using Kaplan-Meier methodology and compared between Arm A and Arm B using the log-rank test stratified by the same stratification factors used for the PFS analysis. In addition, stratified Cox proportional hazard model will be used to estimate the hazard ratio and the corresponding 95% CI.

## 7.4.2.5 Health-Related Quality of Life

HRQoL endpoints will be summarized by descriptive statistics with respect to change from baseline for the FAS for each treatment arm. Completion rate for each questionnaire will be summarized by time point. Additional analyses will be described in the SAP.

## 7.4.3 Analysis of Exploratory Endpoints

### 7.4.3.1 Time to Progression

TTP is defined as the time from the date of randomization until the date of PD (per RECIST 1.1 by IRC). TTP does not include deaths as event. For deaths before the first documented PD by IRC, subjects will be censored at the time of last radiological assessment. Kaplan-Meier and log-rank methods will be applied to TTP endpoint.

## 7.4.3.2 Progression Free Survival After Subsequent Therapy (PFS2)

PFS2 is defined as the time from the date of randomization until the date of PD (per investigator) following subsequent anticancer therapy, death from any cause or start of any other anticancer therapy, whichever is earliest. In cases where PFS2 cannot be reliably

determined, discontinuation of subsequent anticancer treatment may be used as the event date. Otherwise, subjects will be censored. Subjects who are alive and for whom a PFS2 event date has not been observed should be censored at the last time known to be alive and without second objective disease progression.

The distribution of PFS2 will be estimated for each treatment arm using Kaplan-Meier methodology and compared between Arm A and Arm B using stratified log-rank test with the same stratification factors used for the PFS analysis. In addition, stratified Cox proportional hazard model will be used to estimate the hazard ratio and the corresponding 95% CI.

## 7.4.3.3 Disease Control Rate

The DCR is defined as the proportion of subjects with a BOR of CR, PR or SD based on RECIST 1.1 by IRC.

The comparison of DCR between Arm A and Arm B will be performed using CMH test with the same stratification factor used for PFS analysis. In addition, DCR for each arm will be estimated and corresponding 95% CI will be constructed.

#### 7.4.3.4 Biomarkers

Biomarkers may be summarized graphically or descriptively, and summary statistics may be tabulated. Associations between biomarkers and clinical (e.g., efficacy, safety or pharmacodynamics, pharmacokinetics) measures may be performed on subjects who have sufficient baseline and on-study measurements to provide interpretable results for specific parameters. Additional post-hoc statistical analyses may be outlined in the SAP.

## 7.4.3.5 Health Resource Utilization

HRU variables will be summarized for each treatment arm.

# 7.5 Analysis of Safety

All treated subjects will be analyzed according to the treatment they received.

### 7.5.1 Adverse Events

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and graded using NCI-CTCAE v4.03.

Treatment-emergent adverse event (TEAE) is defined as an AE observed after starting administration of the study treatment and within 30 days after the last dose of study treatment. Late SAE and/or AE is defined as (S)AE that is collected after 30 days post last dose of study drug.

A study drug-related TEAE is defined as any TEAE with a causal relationship of YES by the investigator.

AEs of special interest described in [Section 5.5.8 Adverse Events of Special Interest] will be summarized.

The number and percentage of AEs, SAEs, AEs leading to interruption/discontinuation, AEs leading to death and AEs related to study drug will be summarized by SOC, preferred term (PT) for SAF. The number and percentage of AEs by toxicity grade will also be summarized. Late (S)AEs will be summarized. All AEs will be listed.

## 7.5.2 Laboratory Assessments

For quantitative laboratory measurements descriptive statistics will be used to summarize results and change from baseline for subjects in the SAF by treatment group and time point.

Shifts from baseline to the worst grade based on NCI-CTCAE v4.03 in laboratory tests will also be tabulated.

## 7.5.3 Vital Signs

Descriptive statistics will be used to summarize vital sign results and changes from baseline for subjects in the SAF by treatment group and time point.

## 7.5.4 Routine 12-lead Electrocardiograms

The 12-lead ECG results will be summarized by treatment group and time point.

## 7.5.5 Eastern Cooperative Oncology Group Performance Status

Summary statistics (number and percent of subjects) for each category of the ECOG performance status at each assessment will be provided. The change from baseline to final visit or early termination will also be summarized. Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

# 7.6 Analysis of Pharmacokinetics

Descriptive statistics will include the number of subjects (n), mean, standard deviation, minimum, median, maximum, coefficient of variation (CV), geometric mean and geometric CV.

### 7.6.1 Serum Concentrations

Serum concentrations of zolbetuximab will be listed and summarized using descriptive statistics by scheduled time point. Box and whisker plots of trough concentrations against cycle and dosing day will be provided.

## 7.6.2 Immunogenicity

Immunogenicity of zolbetuximab will be summarized using the frequency of ADA positive subjects. The potential relationship between zolbetuximab immunogenicity and zolbetuximab pharmacokinetics, efficacy, safety profile in subjects may be assessed.

Additional model-based analyses may be performed and reported separately for zolbetuximab pharmacokinetics.

## 7.7 Major Protocol Deviations and Other Analyses

Major protocol deviations as defined in [Section 8.2 Major Protocol Deviations] will be summarized for all randomized subjects by treatment group and total as well as by site. A data listing will be provided by site and subject.

The major protocol deviation criteria will be uniquely identified in the summary table and listing.

# 7.8 Interim Analysis (and Early Discontinuation of the Clinical Study)

To evaluate whether zolbetuximab + CAPOX (Arm A) is beneficial compared to placebo + CAPOX (Arm B) while the study is ongoing, a formal OS interim analysis is planned when the final PFS analysis occurs with the pre-specified number of PFS events. A group sequential design using the O'Brien-Fleming type alpha-spending function [Lan & DeMets, 1983] for efficacy will be utilized to control the overall 1-sided 0.025 significance level (East®) for the OS analyses.

The IDMC may recommend terminating the study for favorable results at the formal efficacy interim analysis using OS. In the case of favorable results, the 1-sided significance level for superiority is 0.0074, assuming about 70% of the target number of OS events is obtained, for the interim OS analysis and 0.0228 for the final OS analysis (Note: The OS significance level will be adjusted depending on the number of OS events at the time of interim analysis). If the 1-sided P value of the interim analysis is less than the significance level (and PFS is also significant at 1-sided 0.025 alpha), the IDMC may recommend terminating the study for success. If the study is not stopped after the interim analysis, a final OS analysis will occur after 100% of the planned death events have been observed.

The interim OS analysis will be conducted by an Independent Data Analysis Center for IDMC. In addition, safety data reviews during the study will be conducted by the IDMC on a periodic basis. For example, the IDMC will have its first safety data review 6 weeks after the 40<sup>th</sup> subject has been randomized and on study drug for 2 cycles (6 weeks) and meetings will be conducted regularly thereafter, as determined by the IDMC.

The full procedures for IDMC safety review will be described in a separate IDMC Charter.

The analysis for the eCOA endpoints will be performed as the final analysis once OS is significant either at the interim OR or at final OS analysis hence there is no interim analysis planned for eCOA endpoints.

# 7.9 Handling of Missing Data, Outliers, Visit Windows, and Other Information

Imputation for missing data, if applicable, will be addressed in the SAP.

## 8 OPERATIONAL CONSIDERATIONS

# 8.1 Procedure for Clinical Study Quality Control

### 8.1.1 Data Collection

The investigator or site designee will enter data collected using an electronic data capture system. In the interest of collecting data in the most efficient manner, the investigator or site designee should record data (including laboratory values, if applicable) in the eCRF within 5 days after the subject visit.

The investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF. These documents should be appropriately maintained by the site.

Local laboratory results may be used for treatment decisions; however, central laboratory samples must also be drawn per protocol and sent to the central laboratory unless otherwise approved by sponsor. (*UNIQUE TO CHINA*: Local laboratory results may be used for treatment decisions; however, central laboratory samples should also be drawn per protocol and sent to the central laboratory unless otherwise approved by the sponsor.) Central Laboratory data will be transferred electronically to the sponsor or designee at predefined intervals during the study. The central laboratory will provide the sponsor or designee with a complete and clean copy of the data.

Imaging results are read by a local or central imaging laboratory. Central imaging data will be transferred electronically to the sponsor or designee at predefined intervals during the study. The central imaging laboratory will provide the sponsor or designee with a complete and clean copy of the data.

For Screen failures the demographic data, reason for failing, informed consent, inclusion and exclusion criteria and AEs will be collected in the eCRF.

## 8.1.1.1 Collection of Data Via Electronic Source

All procedures conducted under the protocol must be documented. For screen failures, the minimum demographic data (sex, birth date, race and informed consent date), outcome of eligibility assessment (inclusion and exclusion criteria), reason for screen failure and AEs details must be documented.

The investigator or designee will be responsible for eCRF completion and for ensuring the source data are attributable, legible, contemporaneous, original, accurate and complete whether the data are handwritten on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved or transmitted electronically via computerized systems (and/or other kind of electronic devices) as part of regulated study activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records, protocol-related assessments, AE tracking, electronic clinical outcome assessment and/or drug accountability.

(UNIQUE TO CHINA: The investigator or designee will be responsible for eCRF completion and that all data and queries are accurate, complete and are verifiable with the source. The investigator or designee will also be responsible for ensuring the source data are attributable, legible, contemporaneous, original, accurate and complete whether the data are handwritten on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved or transmitted electronically via computerized systems (and/or other kind of electronic devices) as part of regulated study activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records, protocol-related assessments, AE tracking, electronic clinical outcome assessment and/or drug accountability.)

Electronic data sources and any supporting documents should be available for review/retrieval by the sponsor/designee at any given time.

Study monitors will perform ongoing source data review to confirm that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

## 8.1.1.2 Electronic Clinical Outcomes Assessment

Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), eCOA assessments will be discontinued according to the Schedule of Assessments [Table 11].

Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), eCOA assessments will be performed according to the Schedule of Assessments [Table 1]. Subject HRQoL and HRU questionnaires will be completed by the subject or, if not possible, administered to the subject by site personnel on an electronic tablet device for subject visits. The subject questionnaire responses captured on the electronic device will be transferred to the eCOA vendor's central portal (web portal). The investigator or site designee should review the questionnaire data on the web portal for correct completion while the subject is at the site. The questionnaire data will be transferred electronically to sponsor or designee at predefined intervals during the study. Sponsor/CRO staff also have access to the vendor web portal for continuous review of the data and access to reports. The vendor will provide sponsor or designee with a complete and clean copy of the data.

For further details please refer to the eCOA guidelines/manual (e.g., ERT Site Guide to eCOA Product).

# **8.2** Major Protocol Deviations

A major protocol deviation is generally an unplanned excursion from the protocol that is not implemented or intended as a systematic change. All deviations from the protocol are to be recorded. A protocol waiver is a documented prospective approval of a request from an investigator to deviate from the protocol. Protocol waivers are strictly prohibited.

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol and must protect the rights, safety, and welfare of subjects. The investigator should not implement any deviation from, or changes of, the protocol, unless it is necessary to eliminate an immediate hazard to study subjects.

When a major deviation from the protocol is identified for an individual subject, the investigator or designee must ensure the sponsor is notified. The sponsor will follow up with the investigator, as applicable, to assess the deviation and the possible impact to the safety of the subject to determine subject continuation in the study.

Major protocol deviation criteria will be summarized at the end of the study.

The investigator will also assure that deviations meeting IRB/IEC and applicable regulatory authorities' criteria are documented and communicated appropriately. All documentation and communications to the IRB/IEC and applicable regulatory authorities will be provided to the sponsor and maintained within the trial master file.

## 9 END OF TRIAL

The end of the study is defined as the last visit or scheduled procedure shown in the Schedule of Assessments [Table 1] and [Table 11] for the last study participant in the study.

Study completion is defined as the conclusion of data collection for the defined study endpoints. The study may be closed within a participating country per local regulations once the study has completed and if all subjects enrolled in the country are no longer receiving study treatment. In addition, the sponsor may prematurely terminate the study for reasonable cause at any time.

## 10 STUDY ORGANIZATION

# **10.1** Independent Data Monitoring Committee

An IDMC will evaluate the unblinded safety data of subjects enrolled on a periodic basis during this study. IDMC members will be clinicians with expertise in gastric cancer studies and are not investigators participating in this study or Astellas employees. A separate charter will outline the activities of this committee.

# 10.2 Other Study Organization

**SPECIFIC TO SITES IN JAPAN**: The Japan site contact list is kept as a separate attachment to the protocol.

## 11 REFERENCES

- Ajani JA, Rodriguez W, Bodoky G, Moiseyenko V, Lichinitser M, Gorbunova V, et al. Multicenter phase III comparison of cisplatin/S-1 with cisplatin/infusional fluorouracil in advanced gastric or gastroesophageal adenocarcinoma study: the FLAGS trial. J Clin Oncol. 2010 Mar;28(9):1547-53.
- Amiri M, Janssen F, Kunst AE. The decline in stomach cancer mortality: exploration of future trends in seven European countries. Eur J Epidermiol. 2011;26:23-8.
- Bang Y, Chung H, Xu J, Lordick F, Sawaki A, Al-Sakaff N, et al. Pathological features of advanced gastric cancer (GC): Relationship to human epidermal growth factor receptor 2 (HER2) positivity in the global screening programme of the ToGA trial. J Clin Oncol. 2009;27(155):4556.
- Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet 2010;376:687-97.
- Cancer Fact Sheet. World Health Organization; February 2018.
- CYRAMZA Prescribing Information. Indianapolis, IN: Eli Lilly and Company; 2017.
- Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer 2009;45:228-247.
- Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, et al. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014;383:31-39.
- Gunzel D, Yu SL. Claudins of the modulation of tight junction permeability. Physiol. Rev. 2013;93(2): 525-69.
- HERCEPTIN (trastuzumab) [package insert]. South San Francisco, CA: Genentech, Inc.; 2016.
- Karanjawala ZE, Illei PB, Ashfaq R, Infante JR, Murphy K, Pandey A, et al. New markers of pancreatic cancer identified through differential gene expression analyses: claudin 18 and annexin A8. Am J Surg Pathol. 2008;32:188-96.
- Kim GM, Jeung HC, Rha SY, Kim HS, Jung I, Nam BH, et al. A randomized phase II trial of S-1-oxaliplatin versus capecitabine-oxaliplatin in advanced gastric cancer. Eur J Cancer. 2012 Mar;48(4):518-26.
- Kim NK, Park YS, Heo DS, Suh C, Kim SY, Park KC, et al. A phase III randomized study of 5-fluorouracil and cisplatin versus 5-fluorouracil, doxorubicin and mitomycin C versus 5-fluorouracil alone in the treatment of advanced gastric cancer. Cancer. 1993;71:3813-18.
- Lan KKG and De Mets DL. Discrete sequential boundaries for clinical trials. Biometrika. 1983;70:659-663.

- Lederman L. Gastric Cancer: local and global burden. Supplement: the current and future management of gastric cancer. Am J Manag Care. 2017:2-5.
- Lee JH, Kim KS, Kim TJ, Hong SP, Song SY, Chung JB, et al. Immunohistochemical analysis of claudin expression in pancreatic cystic tumors. Oncol Rep. 2011;25:971-978.
- National Comprehensive Cancer Network Clinical Practice Guidelines in Oncology (NCCN Guidelines): Gastric cancer. National Comprehensive Cancer Network (NCCN). 2017; version 1.2017.
- Niimi T, Nagashima K, Ward JM, Minoo P, Zimonjic DB, Popescu NC, et al. claudin-18, a novel downstream target gene for the T/EBP/NKX2.1 homeodomain transcription factor, encodes lung- and stomach-specific isoforms through alternative splicing. Mol Cell Biol. 2001;21(21):7380-7390.
- Ohtsu A, Shah MA, Van Cutsem E, Rha SY, Sawaki A, Park SR, et al. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a randomized, double-blind, placebo-controlled phase III study. J Clin Oncol. 2011;29:3968-3976.
- Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982;5(6):649-55.
- Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol.1998;16(1):139-44.
- Pasini F, Fraccon AP, De Manzoni G. The role of chemotherapy in metastatic gastric cancer. Cancer Res. 2011;31:3543-3554.
- Pennathur A, Gibson MK, Jobe BA, Luketich JD. Oesophageal carcinoma. Lancet. 2013;381:400-12.
- Sahin U, Koslowski M, Dhaene K, Usener D, Brandenburg G, Seitz G, et al. Claudin-18 splice variant 2 is a pan-cancer target suitable for therapeutic antibody development. Clin Cancer Res. 2008;14(23):7624-34.
- Sanada Y, Hirose Y, Osada S, Tanaka Y, Takahashi T, Yamaguchi K, et al. Immunohistochemical study of claudin 18 involvement in intestinal differentiation during the progression of intraductal papillary mucinous neoplasm. Anticancer Res. 2010;30:2995-3003.
- Shah MA, Bang YJ, Lordick F, Alsina M, Chen M, Hack SP, et al. Effect of Fluorouracil, Leucovorin, and Oxaliplatin With or Without Onartuzumab in HER2-Negative, MET-Positive Gastroesophageal Adenocarcinoma The METGastric Randomized Clinical Trial. JAMA Oncol. 2017;3(5):620-7.
- Vita FDe, Orditura M, Matano E, Bianco R, Carlomagno C, Infusino S, et al. A phase II study of biweekly oxaliplatin plus infusional 5-fluorouracil and folinic acid (FOLFOX-4) as first-line treatment of advanced gastric cancer patients. Br J Cancer. 2005;92(9):1644-49.
- Waddell T, Chau I, Cunningham D, Gonzalez D, Okines AF, Wotherspoon A, et al. Epirubicin, oxaliplatin, and capecitabine with or without panitumumab for patients with previously untreated advanced oesophagogastric cancer (REAL3): a randomized, open-label phase 3 trial. Lancet Oncol. 2013;14(6):481-9.

06 Dec 2024 Astellas 

- Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, et al. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014;15:1224-35.
- Wöll S, Schlitter AM, Dhaene K, Roller M, Esposito I, Sahin U, et al. Claudin 18.2 is a target for IMAB362 antibody in pancreatic neoplasms. Int. J. Cancer. 2014;134:731-9.

XELOX CCO Formulary, August 2017.

## 12 APPENDICES

# 12.1 Ethical, Regulatory, and Study Oversight Considerations

## 12.1.1 Ethical Conduct of the Study

The study will be conducted in accordance with the protocol, ICH guidelines, all applicable regulations and guidelines governing clinical study conduct and the ethical principles that have their origin in the Declaration of Helsinki.

# 12.1.2 Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/Competent Authorities (CA)

GCP requires that the clinical protocol, any protocol amendments, the IB, the informed consent and all other forms of subject information related to the study (e.g., advertisements used to recruit subjects) and any other necessary documents be reviewed by an IEC/IRB. The IEC/IRB will review the ethical, scientific and medical appropriateness of the study before it is conducted. IEC/IRB approval of the protocol, informed consent and subject information and/or advertising, as relevant, will be obtained prior to the authorization of drug shipment to a study site.

Any substantial amendments to the protocol will require IRB/IEC approval before to implementation, except for changes necessary to eliminate an immediate hazard to subjects.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
- Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/IEC, European regulation 536/2014 for clinical studies (if applicable), and all other applicable local regulations

## 12.1.3 Protocol Amendment and/or Revision

Any changes to the study that arise after approval of the protocol must be documented as protocol amendments: substantial amendments and/or non-substantial amendments. Depending on the nature of the amendment, either IRB/IEC, Competent Authority approval or notification may be required. The changes will become effective only after the approval of the sponsor, the investigator, the regulatory authority, and the IRB/IEC (if applicable).

Amendments to this protocol must be signed by the sponsor and the investigator. Written verification of IRB/IEC approval will be obtained before any amendment is implemented. Modifications to the protocol that are administrative in nature do not require IRB/IEC approval, but will be submitted to the IRB/IEC for their information, if required by local regulations.

If there are changes to the informed consent, written verification of IRB/IEC approval must be forwarded to the sponsor. An approved copy of the new informed consent must also be forwarded to the sponsor.

## 12.1.4 Informed Consent of Subjects

## 12.1.4.1 Subject Information and Consent

The investigator or his/her representative will explain the nature of the study to the subject or his/her guardian or legal representative (if applicable), and answer all questions regarding this study.

An optional partial screening ICF may be available to allow central testing of tissue for CLDN18.2 and HER2 only. (*UNIQUE TO CHINA*: A partial screening ICF may be available for central testing of tissue for CLDN18.2 only.)

Prior to any study-related screening procedures being performed on the subject, the informed consent statement will be reviewed and signed (*UNIQUE TO JAPAN REGION*: place a personal seal) and dated by the subject or his/her guardian or legal representative, the person who administered the informed consent and any other signatories according to local requirements. A copy of the signed (*UNIQUE TO JAPAN REGION*: or sealed) ICF will be given to the subject and the original will be placed in the subject's medical record. An entry must also be made in the subject's dated source documents to confirm that informed consent was obtained prior to any study-related procedures and that the subject received a signed copy. The signed consent forms will be retained by the investigator and made available (for review only) to the study monitor and auditor regulatory authorities and other applicable individuals upon request.

# 12.1.4.2 Supply of New and Important Information Influencing the Subject's Consent and Revision of the Written Information

- 1. The investigator or his/her representative will immediately inform the subject orally whenever new information becomes available that may be relevant to the subject's consent or may influence the subject's willingness to continue to participate in the study (e.g., report of serious drug adverse drug reaction). The communication must be documented in the subject's medical records and whether the subject is willing to remain in the study or not must be confirmed and documented.
- 2. The investigator must update their ICF and submit it for approval to the IRB/IEC. The investigator or his/her representative must obtain written informed consent from the subject on all updated ICFs throughout their participation in the study. The investigator or his/her designee must re-consent subjects with the updated ICF even if relevant information was provided orally. The investigator or his/her representative who obtained the written informed consent and the subject should sign and date the ICF (*UNIQUE TO JAPAN REGION:* place a personal seal). A copy of the signed (*UNIQUE TO JAPAN REGION:* or sealed) ICF will be given to the subject and the original will be placed in the subject's medical record. An entry must be made in the subject's records documenting the re-consent process.

### 12.1.5 Source Documents

Source data must be available at the site to document the existence of the study subjects and to substantiate the integrity of study data collected. Source data must include the original documents relating to the study, as well as the medical treatment and medical history of the subject.

The investigator is responsible for ensuring the source data are attributable, legible, contemporaneous, original, accurate and complete whether the data are hand-written on paper or entered electronically. If source data are created (first entered), modified, maintained, achieved, retrieved or transmitted electronically via computerized systems (and/or other kind of electric devices) as part of regulated clinical study activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records, protocol related assessments, AE tracking, and/or drug accountability.

Paper records from electronic systems used in place of electronic format must be certified copies. A certified copy must be an exact copy and must have all the same attributes and information as the original. Certified copies must include signature and date of the individual completing the certification. Certified copies must be a complete and chronological set of study records (including notes, attachments, and audit trail information (if applicable). All printed records must be kept in the subject file and available for archive.

(UNIQUE TO CHINA: Paper records from electronic systems used in place of electronic format should be certified copies. A certified copy should be an exact copy and must have all the same attributes and information as the original. Certified copies should include signature and date of the individual completing the certification. Certified copies should be a complete and chronological set of study records (including notes, attachments, and audit trail information (if applicable). All printed records should be kept in the subject file and available for archive.)

## 12.1.6 Record Retention

The investigator will archive all study data (e.g., subject identification code list, source data, eCRFs and investigator's file) and relevant correspondence. These documents are to be kept on file for the appropriate term determined by local regulation (for US sites, two years after approval of the NDA or discontinuation of the IND). The sponsor will notify the site/investigator if the NDA/MAA/J-NDA is approved or if the IND/IMPD/CHIKEN TODOKE is discontinued. The investigator agrees to obtain the sponsor's agreement prior to disposal, moving, or transferring of any study-related records. The sponsor will archive and retain all documents pertaining to the study according to local regulations.

Data generated by the methods described in the protocol will be recorded in the subjects' medical records and/or study progress notes.

## 12.1.7 Subject Confidentiality and Privacy

Individual subject medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited unless otherwise the subject provides written consent or approval. Additional medical information may be given only after approval of the subject to the investigator or to other appropriate medical personnel responsible for the subject's well-being.

The sponsor shall not disclose any confidential information on subjects obtained during the performance of their duties in the clinical study without justifiable reasons.

Even though any individuals involved in the study, including the study monitors and auditors, may get to know matters related to subject's privacy due to direct access to source documents, or from other sources, they may not leak the content to third parties.

The sponsor affirms the subject's right to protection against invasion of privacy. Only a subject identification number will identify subject data retrieved by the sponsor. However, the sponsor requires the investigator to permit the sponsor, sponsor's representative(s), the IRB/IEC and when necessary, representatives of the regulatory health authorities to review and/or to copy any medical records relevant to the study.

The sponsor agrees to comply and process personal data in accordance with all applicable privacy laws and regulations, including, without limitation, the Personal Information Protection Law in Japan and Privacy laws in the US. If the services will involve the collection or processing of personal data (as defined by applicable data protection legislation) within the European Economic Area (EEA), then sponsor shall serve as the controller of such data, as defined by the European Union (EU) Data Protection Directive, and Investigator and/or third party shall act only under the instructions of the sponsor in regard to personal data. If sponsor is not based in the EEA, sponsor must appoint a third party to act as its local data protection representative or arrange for a co-controller established in the EU for data protection purposes in order to comply with the Directive.

## 12.1.8 Arrangement for Use of Information and Publication of the Clinical Study

Information concerning the study drug, patent applications, processes, unpublished scientific data, the IB and other pertinent information is confidential and remains the property of the sponsor. Details should be disclosed only to the persons involved in the approval or conduct of the study. The investigator may use this information for the purpose of the study only. It is understood by the investigator that the sponsor will use the information obtained during the clinical study in connection with the development of the drug and therefore may disclose it as required to other clinical investigators or to regulatory agencies. In order to allow for the use of the information derived from this clinical study, the investigator understands that he/she has an obligation to provide the sponsor with all data obtained during the study.

Publication of the study results is discussed in the clinical study agreement.

# 12.1.9 Insurance of Subjects and Others (UNIQUE TO JAPAN REGION/STUDIES ENROLLING SUBJECTS IN EU)

If a subject suffers any study-related injury, the sponsor will compensate appropriately according to the severity and duration of the damage. However, if it was caused intentionally or was due to gross negligence by the study site, the sponsor will consult with the study site about handling the injury, based on the agreed study contract. Compensation for the study-related injury is provided by the following procedures:

- 1. If a subject incurs an injury as a result of participation in the clinical study, the study site should provide medical treatment and other necessary measures. The sponsor should be notified of the injury.
- 2. When the subject claims compensation from the study site for the above study-related injury, or such compensation may be claimed, the study site should immediately communicate the fact to the sponsor. Both parties should work together towards compensation settlement.
- 3. The sponsor shall pay compensation or indemnification and bear expenses necessary for the settlement as provided in the clinical contract.
- 4. The sponsor shall make an arranging for insurance and take measures necessary to ensure the compensation or indemnification mentioned above.

The sponsor has covered this study by means of an insurance of the study according to national requirements. The name and address of the relevant insurance company, the certificate of insurance, the policy number and the sum insured are provided in the investigator's file.

## 12.1.10 Signatory Investigator for Clinical Study Report

ICH E3 guidelines recommend and EU Directive 2001/83/EC requires that a final study report, which forms part of a marketing authorization application, be signed by the representative for the coordinating investigator(s) or the principal investigator(s). The representative for the coordinating investigator (s) or the principal investigator(s) will have the responsibility to review the final study results to confirm to the best of his/her knowledge it accurately describes the conduct and results of the study. The representative for coordinating investigator(s) or the principal investigator(s) will be selected from the participating investigators by the sponsor prior to database lock.

# 12.2 Procedures for Clinical Study Quality Control

## 12.2.1 Clinical Study Monitoring

The sponsor or delegated CRO is responsible for monitoring the clinical study to ensure that subject's human rights, safety, and well-being are protected, that the study is properly conducted in adherence to the current protocol and GCP, and study data reported by the investigator/sub-investigator are accurate and complete and that they are verifiable with study-related records such as source documents. The sponsor is responsible for assigning study monitor(s) to this study for proper monitoring. They will monitor the study in accordance with planned monitoring procedures.

## 12.2.2 Direct Access to Source Data/Documents

The investigator and the study site must accept monitoring and auditing by the sponsor or delegated CRO as well as inspections from the IRB/IEC and relevant regulatory authorities. In these instances, they must provide all study-related records, including source documents when they are requested by the sponsor monitors and auditors, the IRB/IEC or regulatory authorities. The confidentiality of the subject's identities shall be well protected consistent with local and national regulations when the source documents are subject to direct access.

Remote source data review will be used when needed. It will focus on the quality control of critical data such as primary efficacy data and important safety data. Important secondary efficacy data will be monitored simultaneously, provided this does not result in a need to access additional documents and therefore increase the burden for site staff. The sponsor will determine the extent and nature of remote source data review that is needed for any exceptional situations and will carefully weigh it against the extra burden that introduction of any alternative measures would put on site staff and facilities.

(UNIQUE TO CHINA: Remote source data review and/or verification will be used when needed. The sponsor will determine the extent and nature of remote source data review and/or verification that is needed for any exceptional situations and will carefully weigh it against the extra burden that introduction of any alternative measures would put on site staff and facilities.)

### 12.2.3 Data Management

Data Management will be coordinated by the Data Science of the sponsor in accordance with the SOPs for data management. All study-specific processes and definitions will be documented by Data Management. eCRF completion will be described in the eCRF instructions. Coding of medical terms and medications will be performed using MedDRA and World Health Organization (WHO) Drug Dictionary, respectively.

## 12.2.4 QUALITY ASSURANCE

The sponsor is implementing and maintaining quality assurance and quality control systems with written SOPs to ensure that studies are conducted and data are generated, documented, recorded, and reported in compliance with the protocol, GCP, and applicable regulatory

requirement(s). Where applicable, the quality assurance and quality control systems and written SOPs of the CRO will be applied.

The sponsor or sponsor's designee may arrange to audit the clinical study at any or all investigational sites and facilities. The audit may include on-site review of regulatory documents, case report forms, and source documents. Direct access to these documents will be required by the auditors.

# 12.3 Contraception Requirements

WOCBP participants who choose complete abstinence must continue to have pregnancy tests, as specified in Schedule of Assessments [Table 1] and [Table 11].

# WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION DEFINITIONS (WOCBP)

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile.

## Women in the following categories are not considered WOCBP

- Premenarchal
- Premenopausal female with 1 of the following:
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy
- Postmenopausal

Documentation of any of these categories can come from the site personnel's review of the female subject's medical records, medical examination, or medical history interview.

A postmenopausal state is defined as at least 12 months after last regular menstrual bleeding without an alternative medical cause.

• In case the last regular menstrual bleeding cannot be clearly determined, confirmation with repeated FSH measurements of at least > 40 IU/L (or higher per local institutional guidelines), is required.

Females on HRT and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status by repeated FSH measurements before study enrollment.

# CONTRACEPTION GUIDANCE FOR FEMALE PARTICIPANTS OF CHILD BEARING POTENTIAL

One of the highly effective methods of contraception listed below is required at the time of informed consent and until the end of relevant systemic exposure, defined as 9 months after the final administration of oxaliplatin and 6 months after the final administration of all other study drugs<sup>a</sup>.

**Highly Effective Contraceptive Methods** (Failure rate of <1% per year when used consistently and correctly)<sup>b</sup>

Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation

- oral
- intravaginal

### transdermal

Progestogen-only hormonal contraception associated with inhibition of ovulation

- oral
- injectable
- implantable

Hormonal methods of contraception containing a combination of estrogen and progesterone, vaginal ring, injectables, implants and intrauterine hormone-releasing system (IUS)

- intrauterine device (IUD)
- bilateral tubal occlusion

Vasectomized partner (A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.)

Sexual abstinence (Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant. It is not necessary to use any other method of contraception when complete abstinence is elected.)

# CONTRACEPTION GUIDANCE FOR MALE PARTICIPANTS WITH PARTNER(S) OF CHILD BEARING POTENTIAL.

Male participants with female partners of childbearing potential are eligible to participate if they agree to the following during treatment and until the end of relevant systemic exposure defined as 6 months after final drug administration.

- Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
- Male participants are required to use a condom during treatment and until end of relevant systemic exposure defined as 6 months after final drug administration.
- Female partners of male participants who have not undergone a vasectomy with the absence of sperm confirmed or a bilateral orchiectomy should consider use of effective methods of contraception until the end of relevant systemic exposure, defined as 6 months after final drug administration.

<sup>&</sup>lt;sup>a</sup> Local laws and regulations may require use of alternative and/or additional contraception methods

<sup>&</sup>lt;sup>b</sup> Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies.

## 12.4 Concomitant Medication Restrictions or Requirements

## **Prohibited Concomitant Treatment**

The following are strictly prohibited:

- Sorivudine or analogs (during capecitabine treatment)
- Concurrent non-steroid systemic immunosuppressive agents (for systemic corticosteroids, see cautionary concomitant treatment below).
- Live vaccines should be avoided during the treatment period in which subject is receiving oxaliplatin or capecitabine and up to 6 months after final oxaliplatin or capecitabine dose. In cases where a live vaccine is needed for COVID-19 prevention and allowed per local regulations, please contact the Medical Monitor for discussion.
- Other systemic chemotherapy, immunotherapy, radiotherapy, herbal medications or other treatments intended for antitumor activity.
  - Palliative radiotherapy for peripheral bone metastases is allowed.
  - For gastric bleeding, palliative radiotherapy is prohibited, but esophagogastroduodenoscopy with epinephrine injection is allowed.
- Investigational products or therapy other than zolbetuximab.

## **Cautionary Concomitant Treatment**

Considerations should be given to avoid or minimize the use of the following concomitant medications, if possible, during zolbetuximab/placebo treatment:

- Systemic corticosteroids, because their impact on the potential efficacy of zolbetuximab is not known.
  - Systemic corticosteroids should be avoided or minimized while subject is on study treatment unless required for management of an emergent medical condition (e.g., severe nausea/vomiting or hypersensitivity reaction).
  - For a subject's <u>first dose</u> of zolbetuximab/placebo, it is recommended that the prophylactic use of corticosteroids <u>be avoided</u>.
  - o Inhaled, intranasal, ophthalmic, otic and topically applied steroids are allowed.
  - Subjects are allowed to use a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg/day of hydrocortisone or up to 10 mg/day of prednisone), receive a single dose of systemic corticosteroids or receive systemic corticosteroids as pre-medication for radiologic imaging contrast use.
- Administer 5-HT3 blockers with caution in subjects who have or may develop QTc prolongation.
- Nonsteroidal anti-inflammatory drugs (NSAIDs) because of the potential to cause gastric
  ulcers and covert bleeding.
  - In such cases where NSAID use is necessary, the use of NSAIDs with lower gastric ulcerogenic potential is preferred and concomitant gastric protection with proton pump inhibitors is recommended.

The following should be avoided or used with caution and closely monitored during capecitabine administration:

- Cytochrome P450 (CYP) 2C9 substrates (Subjects taking coumarin-derivative anticoagulants concomitantly with capecitabine should have PT/INR monitored regularly and anticoagulant dose adjusted accordingly).
- Anti-epileptic medications (e.g., phenobarbital, phenytoin and primidone)

The following should be avoided or used with caution and closely monitored during oxaliplatin administration:

 Medications known to prolong the QT or QTc interval (refer to https://www.crediblemeds.org for a list of these medications)

# 12.5 Liver Safety Monitoring and Assessment

Any subject enrolled in a clinical study with active drug therapy and reveals an increase of serum aminotransferases (AT) to > 3 x ULN (to > 5 x ULN in subjects with liver metastases) or bilirubin > 2 x ULN should undergo detailed testing for liver enzymes (including at least ALT, AST, alkaline phosphatase [ALP] and total bilirubin). Testing should be repeated within 72 hours of notification of the test results. For studies for which a central laboratory is used, alerts will be generated by the central laboratory regarding moderate and severe liver abnormality to inform the investigator, study monitor and study team. Subjects should be asked if they have any symptoms suggestive of hepatobiliary dysfunction.

## **Definition of Liver Abnormalities**

Confirmed abnormalities will be characterized as moderate and severe where ULN:

| | ALT or AST | | Total Bilirubin |
|---|---|---|---|
| Moderate | <ul><li>3 x ULN (in subjects without liver metastases),</li><li>5 x ULN (in subjects with liver metastases)</li></ul> | or | > 2 x ULN |
| Severe* | > 3 x ULN (in subjects with five inclastases) | and | > 2 x ULN |

In addition, the subject should be considered to have severe hepatic abnormalities for any of the following:

- ALT or AST  $> 8 \times ULN$ .
- ALT or AST > 5 x ULN for more than 2 weeks (in the absence of liver metastases).
- ALT or AST > 3 x ULN and International Normalized Ratio (INR) > 1.5 (If INR testing is applicable/evaluated).
- ALT or AST > 3 x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).

The investigator may determine that abnormal liver function results, other than as described above, may qualify as moderate or severe abnormalities and require additional monitoring and follow-up.

## **Follow-up Procedures**

Confirmed moderate and severe abnormalities in hepatic functions should be thoroughly characterized by obtaining appropriate expert consultations, detailed pertinent history, physical examination and laboratory tests. The site staff is to complete the liver abnormality case report form (LA-CRF). Subjects with confirmed abnormal liver function testing should be followed as described below.

Confirmed moderately abnormal LFTs should be repeated 2 to 3 times weekly then weekly or less if abnormalities stabilize or the study treatment has been discontinued and the subject is asymptomatic.

Severe hepatic liver function abnormalities as defined above, in the absence of another etiology may be considered an important medical event and may be reported as a SAE. The sponsor

should be contacted and informed of all subjects for whom severe hepatic liver function abnormalities possibly attributable to study treatment are observed.

To further assess abnormal hepatic laboratory findings, the investigator is expected to:

- Obtain a more detailed history of symptoms and prior or concurrent diseases. Symptoms and new-onset diseases is to be recorded as "AEs" in the (e)CRF. Illnesses and conditions such as hypotensive events, and decompensated cardiac disease that may lead to secondary liver abnormalities should be noted. Nonalcoholic steatohepatitis is seen in obese hyperlipoproteinemic, and/or diabetic subjects and may be associated with fluctuating AT levels. The investigator should ensure that the medical history form captures any illness that predates study enrollment that may be relevant in assessing hepatic function.
- Obtain a history of concomitant drug use (including nonprescription medication, complementary and alternative medications), alcohol use, recreational drug use and special diets. Medications, including dose, is to be entered in the (e)CRF. Information on alcohol, other substance use and diet should be entered on the LA-CRF or an appropriate document.
- Obtain a history of exposure to environmental chemical agents.
- Based on the subject's history, other testing may be appropriate including:
  - o Acute viral hepatitis (A, B, C, D, E or other infectious agents),
  - o Ultrasound or other imaging to assess biliary tract disease,
  - o Other laboratory tests including INR, direct bilirubin.
- Consider gastroenterology or hepatology consultations.
- Submit results for any additional testing and possible etiology on the LA-CRF or an appropriate document.

## **Study Treatment Discontinuation**

In the absence of an explanation for increased LFT's, such as viral hepatitis, preexisting or acute liver disease, presence of liver metastases or exposure to other agents associated with liver injury, the subject may be discontinued from study treatment. The investigator may determine that it is not in the subject's best interest to continue study treatment.

Discontinuation of study treatment should be considered if:

- ALT or AST  $> 8 \times ULN$ .
- ALT or AST  $\geq$  5 x ULN for more than 2 weeks (in subjects without liver metastases).
- ALT or AST > 3 x ULN and total bilirubin > 2 x ULN or INR > 1.5 (If INR testing is applicable/evaluated).
- ALT or AST > 5 x ULN and (total bilirubin > 2 x ULN in subjects with liver metastases).
- ALT or AST > 3 x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).

In addition, if close monitoring for a subject with moderate or severe hepatic laboratory tests is not possible, study treatment should be discontinued.

- \*Hy's Law Definition—The 2 "requirements" for Hy's Law are:
- 1. Evidence that a drug can cause hepatocellular-type injury, generally shown by a higher rate than control of people with 3 x and greater transaminase elevations over ULN (2 x elevations are too common in treated and untreated subjects to be discriminating).
- 2. Cases of increased bilirubin (to at least 2 x ULN) in people with concurrent transaminase elevation to at least 3 x ULN (but it is almost invariably higher) and no evidence of intra-or extra-hepatic bilirubin obstruction (elevated ALP) or Gilbert's syndrome. [Temple, 2006]

FDA Guidance for Industry, "Drug-Induced Liver Injury: Premarketing Clinical Evaluation" 2009:

- 1. The drug causes hepatocellular injury, generally shown by a higher incidence of 3-fold or greater elevations above the ULN of ALT or AST than the (non-hepatotoxic) control drug or placebo.
- 2. Among study subjects showing such AT elevations, often with ATs much greater than 3 x ULN, 1 or more also show elevation of serum total bilirubin to > 2 x ULN, without initial findings of cholestasis (elevated serum ALP).
- 3. No other reason can be found to explain the combination of increased AT and total bilirubin, such as viral hepatitis A, B or C; preexisting or acute liver disease; or another drug capable of causing the observed injury.

### References

Temple R. Hy's law: Predicting Serious Hepatotoxicity. Pharmacoepidemiol Drug Saf. 2006 April;15(Suppl 4):241-3.

Guidance for Industry titled "Drug-Induced Liver Injury: Premarketing Clinical Evaluation" issued by FDA on July 2009.

## 12.6 Common Serious Adverse Events

The following is a list of SAEs that the sponsor considers to be associated with the disease state being studied. The list does NOT change your reporting obligations or prevent the need to report an AE meeting the definition of an SAE as detailed in [Section 5.5.2 Definition of Serious Adverse Events]. The purpose of this list is to alert the investigator that some events reported as SAEs may not require expedited reporting to the regulatory authorities based on the classification of "common SAEs". The investigator is required to follow the requirements detailed in [Section 5.5.5 Reporting of Serious Adverse Events].

For IND safety reporting, single occurrences of the following events may be excluded from expedited reporting to the FDA. If aggregate analysis of these events indicates they occur more frequently with study treatment, an expedited IND safety report may be submitted to the FDA.

AEs most likely related to Gastric or GEJ adenocarcinoma:

- Gastric reflux
- Abdominal pain
- Abdominal distention
- Dysphagia
- Loss of appetite

# 12.7 Pharmacogenomic Analysis with Banked Sample

## **INTRODUCTION**

The pharmacogenomic (PGx) research aims to provide information regarding how naturally occurring differences in a subject's gene and/or expression of genes based on genetic variation may impact what treatment options are best suited for the subject. Through investigation of PGx by technologies such as genotyping, gene sequencing, statistical genetics and Genome-Wide Association Studies, the relationship between gene profiles and a drug's kinetics, efficacy or toxicity may be better understood. As many diseases may be influenced by 1 or more genetic variations, PGx research may identify which genes are involved in determining the way a subject may or may not respond to a drug. Samples for PGx are optional and will only be collected as allowed per local policy.

## **OBJECTIVES**

The PGx research that may be conducted in the future with acquired blood samples is exploratory. The objective of this research will be to analyze or determine genes of relevance to clinical response, pharmacokinetics and toxicity/safety issues.

By analyzing genetic variations, it may be possible to predict an individual subject's response to treatment in terms of efficacy and/or toxicity.

## SUBJECT PARTICIPATION

Subjects who have consented to participate in this study may participate in this PGx sub-study, if applicable per local policy. Subjects must provide written consent prior to providing any blood samples that may be used at a later time for PGx analysis.

## SAMPLE COLLECTION AND STORAGE

Subjects who consent to participate in this sub-study will provide one tube of whole blood of approximately 4–6 mL per Astellas' instructions. Each sample will be identified by the unique subject number. Samples will be shipped to a designated banking CRO as directed by Astellas.

### **PGx ANALYSIS**

Details on the potential PGx analysis cannot be established yet. Astellas may initiate the PGx analysis if evidence suggests that genetic variants may be influencing the drug's kinetics, efficacy and/or safety.

## DISPOSAL OF PGx SAMPLES/DATA

All PGx samples collected will be stored for a period of up to 15 years following study database hard-lock. If there is no requirement for analysis, the whole blood sample will be destroyed after the planned storage period. The subject has the right to withdraw consent at any time. When a subject's withdraw notification is received, the PGx sample will be destroyed. The results of any PGx analysis conducted on a sample prior to its withdrawal will be retained at Astellas indefinitely unless otherwise specified by local regulation.

## INFORMATION DISCLOSURE TO THE SUBJECTS

Exploratory PGx analysis may be conducted following the conclusion of the clinical study, if applicable. The results of the PGx analysis will not be provided to any investigators or subjects, nor can the results be requested at a later date. Any information that is obtained from the PGx analysis will be the property of Astellas.


# 12.8 Eastern Cooperative Oncology Group Performance Status Scale

| GRADE | ECOG PERFORMANCE STATUS |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work) |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care; confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled; cannot carry on any self-care; totally confined to bed or chair |
| 5 | Dead |

Reference: Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982;5(6):649-55.

# 12.9 Clinical Study Continuity

## **INTRODUCTION**

The purpose of this appendix is to provide acceptable alternate methods to assess safety and efficacy parameters, as appropriate, in the event the clinical study is interrupted at the country, state, site or participant level during any crisis (e.g., natural disaster, pandemic).

### BENEFIT-RISK RATIONALE

Maintaining the safety of clinical study participants and delivering continuity of care in the clinical study setting is paramount during any crisis. The site is expected to follow the protocol and associated Schedule of Assessments [Table 1] and [Table 11] unless the site PI determines the need to implement the alternate measures. The PI should notify Astellas and/or their CRA when these alternate measures are needed.

The approach outlined within this appendix defines which assessments are required to maintain a favorable benefit/risk to the participant, to maintain overall study integrity and to provide acceptable alternate methods to complete the study required assessments and procedures if study activities are unable to be performed as described in [Table 1] and [Table 12] due to a crisis.

### INFORMED CONSENT

Participants who need to follow any or all of the alternate measures outlined in this Appendix will be required to provide informed consent, which explicitly informs them of the nature of, and rationale for these changes, and gain their agreement to continue participation in the study prior to the implementation of any of these changes. In the event the urgency of implementing the alternate measures does not allow for the participant to provide written consent prior to implementation, the PI or designee will obtain oral agreement from the subject followed by written documentation as soon as is feasible. A separate addendum to the study informed consent will be provided to document the participant's consent of the changes.

#### PARTICIPANT PROCEDURES ASSESSMENT

Sites with participants who are currently enrolled into this clinical study may consider implementing the alternate methods outlined below if one or more of the following conditions are met due to the crisis:

- Regional or local travel has been restricted, inclusive of mandatory shelter in place measures, which makes participant travel to/from the study site nearly impossible
- Site facilities have been closed for clinical study conduct
- Site has been restricted to treating patients with conditions outside of the scope of the study
- Site personnel have temporarily relocated the conduct of the study to a location that place a burden on the participant with respect to time and travel
- Participant(s) have temporarily relocated from the current study site to an alternate study site to avoid placing a burden on the participant with respect to travel

- Participant(s) have temporarily relocated from their home location and the new distances from the site would cause undue burden with respect to time and travel
- Participant has risk factors for which traveling to the site poses an additional risk to the participant's health and safety
**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

# 12.10 Unblinding Procedures Following Final Overall Survival Database Lock

Following completion of the final OS database lock, all principal investigators will be unblinded and informed of the treatment arm for each subject. Subject unblinding will be at the discretion of the principal investigator. Subjects allocated to the placebo arm will be given the option to continue with the CAPOX backbone chemotherapy treatment according to protocol, or discontinue from the study and enter the follow-up period. As the study has achieved the primary objective and key secondary objectives, subjects allocated to zolbetuximab may continue on study treatment until discontinuation criteria is met [Section 6.1].

Adherence to the original protocol as reflected in the Schedule of Assessments [Table 1] and [Table 11] is expected, where plausible, in the case of a crisis. The alternate measures as noted in [Table 10] and [Table 12] below are only permissible in the event of a crisis, and after discussing the need with the Astellas Medical Monitor to implement the alternate measures. This is to allow for continuity of receiving investigational medicinal product (IMP) and maintaining critical safety and efficacy assessments for patients participating in the study at a time of crisis.

If one or more of the alternate measures noted below is implemented for a participant, the site should document in the participant's source document the justification for implementing the alternate measure and the actual alternate measures that were implemented, along with the corresponding time point(s).

Table 10 Up Through Protocol Version 6.1 or Earlier (Original Protocol Version 1 through 6.1): Alternative Schedule of Assessments in Response to a Crisis

| | | | | | Cı | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21, 31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Treatments | | • | • | • | • | • | • | | | | | |
| Antiemetic Pretreatment <sup>5</sup> | Oral antiemetics can be administered at home as per SoC | X | | | X | | | | | | | |
| Zolbetuximab/Placebo <sup>6</sup> | Window of -2 days acceptable; at least<br>every other cycle must be conducted at the<br>study site for zolbetuximab/placebo and<br>oxaliplatin administration and capecitabine<br>dispensing | х | | | х | | | | | | | |
| Post-infusion Observation Period <sup>7</sup> | Decrease of initial observation period to<br>1 hour and subsequent observation period<br>to 30 min is acceptable if there are no AEs<br>of ≥ grade 2 | Х | | | х | | | | | | | |
| Table continued on next page | | | | | | | | | | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | | | | Cı | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21, 31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Oxaliplatin | If previous cycle Day 1 zolbetuximab/placebo administration was conducted at the study site, the following cycle can be administered (oxaliplatin) and dispensed (capecitabine) locally per SoC only (not zolbetuximab/placebo administration) by oncology qualified | X | | | | | | | | | | |
| CAPOX <sup>8</sup> Capecitabine Table continued on next page | personnel, and if dosing records can be obtained from the treating facility. The next cycle then must be administered at the study site for zolbetuximab/placebo administration. At least every other cycle must be conducted at the study site for zolbetuximab/placebo and oxaliplatin administration and capecitabine dispensing. | X | x | | X | X | | | | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | | | | C | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21,31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Safety Assessments | | | | | | | | | | | | |
| Physical Examination <sup>9</sup> | Targeted exam is allowed after C1D1. Physical exam not completed at Study Treatment Discontinuation Visit and 30- Day Safety Follow-up Visit acceptable if no active AE. | X | | | X | | | | | | | |
| Weight <sup>9</sup> | If there are no associated active AEs, it is acceptable if weight is not done at Study Treatment Discontinuation Visit and 30-Day Safety Follow-up Visit. | х | | | Х | | | | | | | |
| Vital Signs <sup>10</sup> | If a cycle is administered at a local facility for SoC regimen administration, SoC can be applied. Missed assessments at Study Treatment Discontinuation Visit and 30-Day Safety Follow-up visit acceptable if there are no associated active AEs. Vital sign frequency during post observation period can be decreased. | Х | | | Х | | | | | | | |
| ECOG Performance Status <sup>9</sup> Table continued on next page | Not required at Study Treatment Discontinuation visit; ECOG Performance Status may be assessed and captured via phone contact. | X | | | Х | | | | | | | |

| | | | | | C | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21, 31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| 12-lead ECG <sup>11</sup> | ECGs allowed up to 4 days prior to treatment visits after C1D1 and can be done locally but must be reviewed prior to dosing; if dosing visits are conducted at local facility, SoC ECG monitoring would be acceptable; if capecitabine only is dispensed and ECG is not able to be performed, this is acceptable; Study Treatment Discontinuation Visit and 30-Day Safety Follow-up Visit required only if clinically indicated. | | X | | | ly indicated<br>al requirem | | (if clin indic | • | | | |
| Image Assessment <sup>12</sup> Table continued on next page | At select visits, efficacy assessment using radiological examinations are required. Independent central reading of locally obtained scans can be facilitated by sharing of Image Acquisition Guidelines from the study site to local site, if applicable. Imaging assessment can be done locally but must be available for submission to central imaging vendor. Investigational site will be requested to re-read the scan performed at local site. If investigational site read is not an option, the investigator should discuss the case with the local institution radiologist. The local site imaging report is required. | Every 9 w | reeks ±7 days | s from C1D1 | for the first | : 54 weeks a | nd then ever | y 12 wee | ks ±7 da | ays there | after <sup>31</sup> | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | | | | C | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | 1 | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21,31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Subject Contact | Long Term Survival and Safety follow-up visits can be conducted via phone. | | | | | | | | | | | X <sup>31</sup> |
| Laboratory Tests | | | | | | | | | | | | |
| Biochemistry <sup>13</sup> | Sample may be collected up to 4 days prior to treatment visit; collection of samples at local facility acceptable if results can be made available to investigative site. | x x | | | | | | X | х | | | |
| TSH and Free T4 <sup>13</sup> | If this testing is unable to be performed, this is acceptable | | | If clinically | y indicated | | | | | | | |
| Hematology <sup>13</sup> | Sample may be collected up to 4 days prior to treatment visit; collection of samples at local facility acceptable if results can be made available to investigative site. | x x | | | | | X | X | | | | |
| Coagulation Parameters (PT, PTT and INR) <sup>14</sup> | None as protocol allows SoC if clinically indicated. If the subject is not on a concomitant medication that affects these parameters, it is acceptable if these are not done. | | | If clinically | y indicated | | | | | | | |
| Urinalysis <sup>13</sup> | Sample may be collected up to 4 days prior to treatment visit; collection at local facility also allowed. | X | | | X <sup>31</sup> | | | X <sup>31</sup> | X <sup>31</sup> | | | |
| Serum Pregnancy Test <sup>15</sup> Table continued on next page | Collection at local facility also allowed. | I | f clinically i | ndicated and | or per local | requiremen | ts | | | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | | | | Cı | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21, 31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Urine Pregnancy Test <sup>16</sup> | Sample may be collected up to 4 days prior to treatment visit; collection at local facility also allowed if results can be made available to investigative site. | X | | | X | | | X | X | | | |
| Sampling | | | | | | | | | | | | |
| Pharmacokinetics of Zolbetuximab (Serum) <sup>23</sup> | Samples at predose/End of Infusion will be collected if subject receives treatment at investigative site. If central lab cannot receive samples, samples can be stored at sites in -70°C freezer until shipping is accepted again. Follow-up samples will be collected if subject visits the investigative site. | X | | | X | | | | X <sup>31</sup> | X <sup>31</sup> | | |
| Antidrug-Antibodies (ADA) for Immunogenicity <sup>24</sup> Table continued on next page | If subject is dosed or visits investigative site, ADA samples should be collected. Samples cannot be collected at local facility. Sample collection prioritized if clinically indicated. If central lab cannot receive samples, samples can be stored at sites in -70°C freezer until shipping is accepted again. | X | | | х | | | | X <sup>31</sup> | X <sup>31</sup> | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | | | | Cı | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21,31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Genetic Immune Polymorphisms (Whole Blood) <sup>25</sup> | In general, biomarker samples are collected<br>on zolbetuximab treatment days and do not<br>require a unique visit to the study site. If<br>samples can be collected but central labs<br>cannot receive samples, samples can be<br>stored at sites until shipping is accepted<br>again. | х | | | | | | | | | | |
| Exploratory Biomarkers (Serum) <sup>26</sup> | In general, biomarker samples are collected<br>on zolbetuximab treatment days and do not<br>require a unique visit to the study site. If<br>samples can be collected but central labs<br>cannot receive samples, samples can be<br>stored at sites until shipping is accepted<br>again. | Х | | | | | | X <sup>31</sup> | | | | |
| Exploratory Biomarkers (Plasma) <sup>26</sup> Table continued on next page | In general, biomarker samples are collected on zolbetuximab treatment days and do not require a unique visit to the study site. If samples can be collected but central labs cannot receive samples, samples can be stored at sites until shipping is accepted again. | X | | | | | | X <sup>31</sup> | | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


| | | | | | Cı | ritical Time | point† | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycles 1-8 | | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>18</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>19</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>20</sup> | Post-treatment<br>Follow-up Period <sup>21, 31</sup> | Long-term and Survival<br>Follow-up Periods <sup>22,31</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | 1 | 2-14 | 15-21 | | | | | |
| Whole Blood Sample for PGx (optional) <sup>27</sup> | In general, biomarker samples are collected on zolbetuximab treatment days and do not require a unique visit to the study site. If samples can be collected but central labs cannot receive samples, samples can be stored at sites until shipping is accepted again. | х | | | | | | | | | | |
| Post-progression Tumor Sample<br>(optional) <sup>28</sup> | In general, biomarker samples are collected on zolbetuximab treatment days and do not require a unique visit to the study site. If samples can be collected but central labs cannot receive samples, samples can be stored at sites until shipping is accepted again. | | | | | | | Х | | | | |
| Concomitant Medication <sup>29</sup> | Remote/Virtual/Telemedicine "Visits" allowed for non-dosing visits. Please refer to protocol schedule of assessments. | X | | | X | | | X | X | X <sup>31</sup> | | |
| AE/SAE <sup>30</sup> | Remote/Virtual/Telemedicine "Visits" allowed for non-dosing visits. Please refer to protocol schedule of assessments. | X | | | X | | | X | X | X <sup>31</sup> | | |

Footnotes appear on next page

ADA: antidrug antibody; AE: adverse event; βhCG: beta human chorionic gonadotropin; C1D1: Cycle 1 Day 1; CAPOX: capecitabine and oxaliplatin; CLDN: claudin; CT: computerized tomography; DPD: dihydropyrimidine dehydrogenase; ECG: electrocardiogram; eCOA: electronic Clinical Outcomes Assessment; ECOG: Eastern Cooperative Oncology Group; eCRF: electronic case report form; FFPE: formalin fixed paraffin embedded; HER2: human epidermal growth factor receptor 2; HRQoL: health-related quality of life; HRU: Health Resource Utilization; ICF: informed consent form: INR: international normalized ratio; IRC: independent review committee; IRR: infusion-related reaction; IRT: interactive response technology; IV: intravenous; MRI: magnetic resonance imaging; OS: overall survival; PD: progressive disease; PFS: progression free survival; PFS2: progression


free survival following subsequent anticancer treatment; PGx: pharmacogenomics; PT: prothrombin time; PTT: partial thromboplastin time; RECIST: Response Evaluation Criteria In Solid Tumors; SAE: serious adverse event; SoC: standard of care; T4: thyroxine; TSH: thyroid stimulating hormone

†In case subjects are unable to be evaluated in person on Day 1 of each cycle, the site will contact the subject by phone for a safety assessment at the time the next visit would be due. ††Additional non-protocol-specific testing may be required per local regulations. Local and/or regional protocols or precautions for COVID-19 management should be followed as applicable.

\*+7 calendar day visit window does not apply to C1D1.

- 1. <u>Screening</u>: The Screening period is 45 days from full main ICF signature. Retesting of lab values is allowed within the 45-day Screening period. Re-screening outside the 45-day window under a new subject number may be allowed once and upon discussion with the Medical Monitor. CT scans and MRIs conducted as part of a subject's routine clinical management (i.e., standard of care) obtained before signing the ICF may be utilized for screening or baseline purposes, provided the procedures met the protocol-specified criteria and were performed within the Screening period.
  - Optional partial screening: A partial screening ICF may be available for central testing of tissue for CLDN18.2 and HER2 only. (UNIQUE TO CHINA: A partial screening ICF may be available for central testing of tissue for CLDN18.2 only).
  - Laboratory testing:
    - Eligibility can be determined based on central and/or local laboratory testing; **however**:
      - o The most recent laboratory tests with available results must be used to confirm the subject's eligibility.
      - o Central labs must be collected and submitted to the central laboratory during the Screening period.
      - o If retesting of lab values is necessary to confirm eligibility, local labs can be used without requiring additional sample collection for central laboratory submission.
    - The screening labs used to determine eligibility should be collected within 14 days prior to randomization.
  - Radiologic imaging used to confirm eligibility must be conducted within 28 days prior to randomization.
- 2. CLDN18.2 and HER2 Testing: FFPE tumor tissue will be collected for central testing to determine CLDN18.2 and HER2 status. (UNIQUE TO CHINA: FFPE tumor tissue will be collected for central testing to determine CLDN18.2 status.) Archival tumor tissue from the primary tumor (gastric or GEJ) is preferred. If primary tumor tissue is not available, tumor tissue from a metastatic site (excluding bone metastasis) may be used. A minimum of 1 FFPE tumor tissue block (preferred) OR a minimum of 15 FFPE unstained slides are required as allowed per local policy. If slides are submitted, the slides should be freshly cut from the FFPE block within the time frame described in the laboratory manual. If local HER2 results are already available from local testing, a minimum of 12 FFPE unstained slides are required to be submitted to the central lab as allowed per local policy. If the specimen is insufficient or unavailable, a biopsy may be performed to obtain primary tumor tissue (preferred) or tumor tissue from metastatic site (excluding bone metastasis). Sponsor pre-approval is required when the sole purpose of the biopsy procedure is to assess eligibility for this study. (UNIQUE TO CHINA: Five FFPE unstained slides are required, as allowed per local policy.) If the required number of slides cannot be provided, the sponsor or designee should be contacted for further guidance. See [Section 5.7.3 Tumor Tissue Samples].
- 3. Confirmation of Inclusion/Exclusion Criteria must be completed prior to randomization.
- 4. <u>Randomization</u>: After confirmation of eligibility, the blinded site user will perform the randomization IRT transaction. The unblinded pharmacist/designee will be notified by the IRT system about the randomly assigned treatment. Randomization may be performed prior to C1D1. If C1D1 cannot be performed within 5 calendar days from Randomization please contact the Medical Monitor for discussion. Details of infusion preparation and storage requirements are defined in the Pharmacy Manual and Infusion Guidelines.


5. <u>Antiemetic Pretreatment</u>: Antiemetic premedication (prophylactic antiemetics) should be administered prior to each study treatment. IV antiemetic premedication should be initiated prior to treatment, or oral antiemetic premedication should be initiated at a <u>minimum of 30 minutes</u> prior to treatment. Antiemetic premedication should be given according to institutional standard of care, published guidelines and the respective product package insert(s). For further details, see [Section 5.1.1.2 Antiemetics].

- 6. <u>Zolbetuximab/placebo</u> will be administered as a minimum 2-hour intravenous infusion every 3 weeks starting on C1D1. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information. Zolbetuximab/placebo should be administered prior to CAPOX. For further details, see [Section 5.1.1.1 Zolbetuximab/Placebo].
- 7. Post-infusion Observation Period: Following the first dose of zolbetuximab/placebo on C1D1, the subject must be observed for 2 hours post-zolbetuximab/placebo infusion. The post-infusion observation period can be conducted during the CAPOX administration. If any ≥ grade 2 AEs are observed during infusion or during the post-infusion observation period, subsequent zolbetuximab/placebo infusion times should be extended and subjects should continue to be observed for 2 hours post zolbetuximab/placebo infusion. If the subject does not develop any grade ≥ 2 AEs, the subject should be observed for 1 hour post-infusion for their subsequent zolbetuximab/placebo infusions. The subject should be instructed to notify site personnel if they develop any AEs during this observation time period. In the event of an IRR with features of anaphylaxis (regardless of grade) or grade 3 or 4 IRR, blood samples for cytokine/chemokine panel and serum total tryptase level (levels typically peak within 3 hours after the onset of symptoms) should be collected once the subject has stabilized, for shipment to the central laboratory. See Observation Period following zolbetuximab/placebo infusion [Section 5.4.2] for further details.
- 8. CAPOX is a combination of oxaliplatin intravenous infusion and capecitabine tablets and will be administered starting at C1D1 for up to 8 treatments. See [Section 5.1.1.3].
- 9. <u>Physical Exam</u>: should include height (at Screening only), <u>weight</u> and <u>ECOG performance status</u>. A full physical exam is required at Screening. The physical exam only needs to be repeated on C1D1 if clinically significant changes from screening are observed (in the opinion of the investigator). For all cycles, the physical examination, weight and ECOG performance status assessments can be completed up to 48 hours prior to zolbetuximab/placebo administration. Targeted (symptom driven) physical exams should be conducted every 3 weeks on day 1 of each cycle. For further details, see [Section 5.4.4 Physical Examination]
- 10. Vital signs (pulse, blood pressure, temperature) should be taken during every visit at the following time points (see [Section 5.4.1 Vital Signs]):
  - o Predose at every visit
  - o C1D1: Every 30 (±10) minutes during zolbetuximab/placebo infusion
  - o If the subject did not develop any ≥ grade 2 AEs during the C1D1 zolbetuximab/placebo infusion or Post-infusion Observation Period, the site may do the following for subsequent zolbetuximab/placebo infusions:
    - The post-infusion observation period can be 1 hour for subsequent visits after C1D1
    - The vital signs can be assessed every 60 minutes for subsequent visits after C1D1
  - Every 60 (±10) minutes post zolbetuximab/placebo infusion during the Post-infusion Observation Period (for 1 or 2 hours. See footnote 7)
  - o Unscheduled if clinically indicated


- 11. <u>ECGs</u>: ECGs will be locally assessed. When collected on the same day, ECG should be collected prior to pharmacokinetic samples. For further details, see [Section 5.4.5 Electrocardiogram]. A single ECG will be performed at the following time points:
  - Screening
  - o Up to 48 hours prior to every oxaliplatin infusion (before any antiemetic treatment administration)
  - o Up to 6 hours following completion of every oxaliplatin infusion
  - o Zolbetuximab/placebo Discontinuation Visit (if clinically indicated)
  - o Zolbetuximab/placebo 30-day Follow-up Visit (if clinically indicated)
  - o If clinically indicated or per local requirements
- 12. Imaging Assessments: Radiologic imaging will be evaluated at Screening (must be conducted within 28 days prior to randomization) and every 9 weeks (± 7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (± 7 days) thereafter until subject develops radiological disease progression per RECIST 1.1 by IRC or starts other systemic anticancer treatment, whichever comes earlier. Imaging schedule should be maintained regardless of treatment delay. Imaging will include CT scans with contrast of the thorax, abdomen, and pelvis. If CT scan with contrast is medically not feasible, MRI may be used for imaging. Bone scans (or focal X-ray) or brain imaging should be performed if metastatic disease in bone or brain is suspected, respectively. The same mode of imaging should be utilized throughout the study unless medical necessity requires a change. For randomized subjects, screening imaging should be sent to the central imaging vendor no later than at the time of submission of the first on-treatment imaging. All imaging acquired post randomization will be sent to the central imaging vendor within 7 days of scanning for the blinded independent central assessment of radiological tumor response based on RECIST 1.1. The investigator should make every effort to immediately submit radiologic assessments for IRC review when PD is suspected. See [Section 5.3 Efficacy Assessments]. Refer to Imaging Acquisition Guidelines for further detail on scan modality and contrast options.
- 13. <u>Laboratory Assessments</u>: See [Section 5.4.3 Laboratory Assessments] for list of laboratory assessments. Laboratory tests must be sent to the central laboratory for analysis. For screening/eligibility laboratory assessments, see footnote number 1.
  - <u>Laboratory test results (central or local) will be reviewed by the investigator prior to any study treatment</u>. Clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician.
  - Local laboratory results may be used for treatment decisions; however, central laboratory samples must also be drawn per protocol and sent to the central laboratory (*UNIQUE TO CHINA*: Local laboratory results may be used for treatment decisions; however, central laboratory samples should also be drawn per protocol and sent to the central laboratory unless otherwise approved by the sponsor.)
  - Central and local labs may be collected up to 48 hours prior to study treatment.
  - Holidays and weekends should be taken into account when scheduling these blood draws.
  - Additional assessments may be done centrally or locally to monitor AEs or as clinically indicated.
- 14. <u>Coagulation</u> (PT, PTT and INR): Coagulation tests should be done at Screening and during study treatment period if clinically indicated. Local or central lab results may be used to confirm eligibility. Ongoing evaluation should be continued for subjects who are receiving therapeutic anticoagulation according to local standard of care. See [Section 5.4.3 Laboratory Assessments].
- 15. Serum Pregnancy Test: Serum pregnancy tests will be collected for female subjects of childbearing potential only. Serum pregnancy tests collected at Screening, during study treatment period and if clinically indicated or per local requirements. Serum pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. (Note: For Screening, subjects with elevated serum βHCG and a demonstrated non-pregnant status through additional testing are eligible.) Local or central laboratory results may be used to confirm eligibility.


16. <u>Urine Pregnancy Test</u>: Urine pregnancy tests will be collected for female subjects of childbearing potential only. Local urine pregnancy tests to be performed during the treatment period every 3 weeks on day 1 of each cycle and at the zolbetuximab/placebo Study Treatment Discontinuation and 30-day Safety Follow-up Visits. Urine pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. Additional urine pregnancy testing for up to 9 months after the final study treatment administration may be conducted based on local requirements.

- 17. <u>HRQoL and HRU questionnaires</u>: eCOA questionnaires should be completed by the subject at Screening (except for HRU), on day 1 of each cycle (or up to 48 hours) before any antiemetic or drug treatment and before the disease status is discussed with the subject using the electronic tablet device provided. When completion by the subject is not possible, the questionnaires may be administered to the subject by site personnel using the electronic tablet device. For subjects with low literacy, situations where translations are unavailable or other circumstances preventing the screening questionnaires to be completed, please contact the sponsor for further guidance.
- 18. Study Treatment Discontinuation Visit (End of Study Treatment): The Study Treatment Discontinuation Visit will take place ≤ 7 days following the decision to discontinue study treatment (zolbetuximab/placebo and CAPOX [both components]). If zolbetuximab/placebo and CAPOX (both components) are discontinued on a different day, subjects will have separate Study Treatment Discontinuation Visits following each treatment's discontinuation. Laboratory tests must be sent to the central laboratory for analysis. HRQoL and HRU questionnaires are not required at CAPOX treatment discontinuation visit. A combined visit can be completed if zolbetuximab/placebo are discontinued on the same day. If necessary during a crisis, this visit can be completed remotely for safety assessments and the required laboratory samples should be collected as soon as the crisis permits.
- 19. 30-day Safety Follow-up Visit: A 30-day Safety Follow-up Visit should occur 30 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 30-day Safety Follow-up Visit should occur 30 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. HRQoL and HRU questionnaires are not required at CAPOX 30-day safety follow up visit. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day and HRQoL and HRU questionnaires should be completed for a combined visit. If necessary during a crisis, this visit can be completed remotely for safety assessments and the required laboratory samples should be collected as soon as the crisis permits.
- 20. 90-day Safety Follow-up Visits: A 90-day Safety Follow-up Visit should occur 90 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 90-day Safety Follow-up Visit should occur 90 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. HRQoL and HRU questionnaires are not required at CAPOX 90-day safety follow up visit. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day and HRQoL and HRU questionnaires should be completed for a combined visit.
- 21. Post-treatment Follow-up: if a subject discontinues all study treatments (zolbetuximab/placebo and both components of CAPOX) prior to IRC-confirmed radiological disease progression, the subject will enter the Post-treatment Follow-up Period and continue to undergo imaging assessments every 9 weeks (±7 days) (or every 12 weeks [±7 days] if subjects has been on study over 54 weeks) until radiologic disease progression (i.e., PFS) or the subject starts subsequent anticancer treatment, whichever occurs earlier. If study treatments (zolbetuximab/placebo and both components of CAPOX) are discontinued due to PD, the subject will enter the Long-term and Survival Follow-up Period.
- 22. Long-term and Survival Follow-up Period: Following disease progression on first-line treatment or start of subsequent anticancer treatment, subjects will be followed in the Long-term and Survival Follow-up Period per institutional guidelines, but not less than every 12 weeks. Radiologic imaging will be done per standard of care and read locally until PFS2 is documented. Survival Follow-up Period will continue until death (from any cause). All post-progression details including subsequent anticancer treatment and date and site of progression will be recorded on the eCRF. Subject contact by phone or other remote methods is sufficient during Long-term and Survival Follow-up.

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

- 23. <u>Pharmacokinetics</u>: Serum samples for zolbetuximab/placebo will be taken at the below time points and sent to the central laboratory. The date and time of each blood sample collection will be recorded to the nearest minute.
  - o Cycle 1 Day 1: End of zolbetuximab/placebo infusion
  - o Cycle 2 Day 1: Predose
  - o Cycle 3 Day 1: End of zolbetuximab/placebo infusion
  - o Predose on Day 1 of Cycles 5, 9, 13 and 17
  - o Zolbetuximab/placebo 30-Day Safety Follow-up visit
  - Zolbetuximab/placebo 90-Day Safety Follow-up visit
  - o Unscheduled pharmacokinetic blood samples may be taken at any time during the study to evaluate drug exposure following a safety event

### Pharmacokinetic Sampling Window:

- o Predose: within 60 minutes prior to dosing
- o End of Infusion: within 10 minutes after the end of the infusion
- 24. ADA: Blood samples (Serum) for ADA will be taken at the below time points and sent to the central laboratory.
  - o Cycle 1 Day 1: Predose
  - o Cycle 2 Day 1: Predose
  - o Predose on Day 1 of Cycles 5, 9, 13 and 17
  - o Zolbetuximab/placebo 30-Day Safety Follow-up visit
  - o Zolbetuximab/placebo 90-Day Safety Follow-up visit

ADA Sampling Window: Predose: within 60 minutes prior to dosing

- 25. <u>Genetic Immune Polymorphism</u>: To be collected per local policy. Whole blood sample taken at C1D1 will be sent to the central laboratory. Samples may be collected up to 48 hours prior to study treatment. (*UNIQUE TO CHINA*: Genomic biomarker testing will not be performed on samples from subjects in China.)
- 26. Exploratory Biomarker (Serum and Plasma): To be collected per local policy. Samples should be taken at the below time points and sent to the central laboratory:
  - o Cycle 1 Day 1: Predose
  - o Cycle 2 Day 1: Predose
  - o Cycle 3 Day 1: Predose
  - o Cycle 4 Day 1: Predose
  - o Cycle 5 Day 1: Predose
  - o Cycle 6 Day 1: Predose
  - o Cycle 8 Day 1: Predose
  - o Zolbetuximab/placebo Study Treatment Discontinuation Visit

Exploratory Biomarker samples may be collected up to 48 hours prior to study treatment.

(UNIQUE TO CHINA: Exploratory biomarker testing will not be performed on samples from subjects in China.)

27. Optional PGx: For subjects who signed a separate ICF, an optional whole blood sample for PGx for exploratory biomarker analysis may be collected up to 48 hours prior to first study drug administration. Sample collection is optional and only collected as allowed per local policy. (UNIQUE TO CHINA: Genomic testing will not be performed on samples from subjects in China.)


- 28. Optional Post-Progression Tumor Sample: For subjects who signed a separate ICF, an optional post-progression tumor sample for exploratory biomarker analysis may be collected following IRC confirmation of disease progression and prior to initiation of subsequent anticancer therapy. Sample collection is optional and only collected as allowed per local policy. (UNIQUE TO CHINA: Optional post-progression tumor sample is not applicable for China.)
- 29. Concomitant medications will be collected from the time of full main informed consent through 90 days following the last dose of study treatment.
- 30. <u>AEs/SAEs</u>: AEs and SAEs (regardless of causality) will be collected from the time of full main informed consent through 90 days following the last dose of study treatment. See [Section 5.5.5 Reporting of Serious Adverse Events].
- 31. With implementation of Protocol Version 7.0, please refer to [Table 11] for the Protocol Version 7.0 and later Schedule of Assessments.

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

#### **IMP SUPPLY**

If any of the conditions outlined above in the Participants Procedures Assessment are met, one or all of the following mitigating strategies will be employed, as needed, to ensure continuity of IMP supply to the participants:

• Increase stock of IMP on site to reduce number of shipments required, if site space will allow, as cold storage space is needed.

#### **DATA COLLECTION REQUIREMENTS**

Additional data may be collected in order to indicate how participation in the study may have been affected by a crisis and to accommodate data collection resulting from alternate measures implemented to manage the conduct of the study and participant safety.

• Critical assessments for safety and efficacy based on study endpoints to be identified as missing or altered (performed virtually, at alternative locations, out of window, or other modifications) due to the crisis.

# 13 PROTOCOL VERSION 7.0 (SUBSTANTIAL AMENDMENT 6) AND LATER: FLOW CHART AND SCHEDULE OF ASSESSMENTS

a. Protocol Version 7.0 (Substantial Amendment 6): Flow Chart



CAPOX: capecitabine and oxaliplatin; CLDN: Claudin; HER2: human epidermal growth factor receptor 2

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

Table 11 Protocol Version 7.0 (Substantial Amendment 6) and Later: Schedule of Assessments

| | Study Treatme | nt Period (Each Cycle = app | proximately 21 Days) | 1 | Follow-up Period | |
|---|---|---|---|---|---|---|
| VISIT† | | Cycle 9+ Zolbetuximab/Placebo + Capecitabine (at investigator discretion | | Study Treatment<br>Discontinuation Visit <sup>13</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>14</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>15</sup> |
| Day | 1 | 2-14 | 15-21 | | | |
| Visit Window (calendar days) | +7 | (no visit) | (no visit) | +7 | ±7 | ±7 |
| Treatments | | | | • | • | |
| Antiemetic Pretreatment <sup>1</sup> | X | | | | | |
| Zolbetuximab/Placebo <sup>2</sup> | X | | | | | |
| Post-infusion Observation Period <sup>3</sup> | X | | | | | |
| Oxaliplatin CAPOX <sup>4</sup> | | | | | | |
| Capecitabine | X | X | | | | |
| Safety Assessments | | | | | | |
| Physical Examination <sup>5</sup> | X | | | X | X | |
| Weight <sup>5</sup> | X | | | X | X | |
| Vital Signs <sup>6</sup> | X | | | X | X | |
| ECOG Performance Status <sup>5</sup> | X | | | X | | |
| 12-lead ECG <sup>7</sup> | | ally indicated and/or per local | | If clinically | | |
| Image Assessment <sup>8</sup> | Every | 9 weeks ±7 days from C1D1 | l for the first 54 weeks and | then every 12 weeks | ±7 days thereafter | |
| Laboratory Tests | | | | | | |
| Biochemistry <sup>9</sup> | X | | | X | X | |
| TSH and Free T49 | | If clinically indicated | | X | | |
| Hematology <sup>9</sup> | X | | | X | X | |
| Coagulation Parameters (PT, PTT and INR) <sup>10</sup> | | If clinically indicated | | | | |
| Urinalysis <sup>9</sup> | | | inically indicated | | | |
| Serum Pregnancy Test <sup>11</sup> | | ally indicated and/or per local | l requirements | | | |
| Urine Pregnancy Test <sup>12</sup> | X | | | X | X | |
| Cytokine/Chemokine and/or Tryptase | | If clinically indicated | | | | |
| Table continued on next page | | | | | _ | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


| | Study Treatmen | t Period (Each Cycle = appı | oximately 21 Days) | I | ollow-up Period | |
|---|---|---|---|---|---|---|
| VISIT† | | Cycle 9+ Zolbetuximab/Placebo + Capecitabine (at investigator discretion) | | Study Treatment<br>Discontinuation Visit <sup>13</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>14</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>15</sup> |
| Day | 1 | 2-14 | 15-21 | | | |
| Visit Window (calendar days) | +7 | (no visit) | (no visit) | +7 | ±7 | ±7 |
| Sampling | | | | | | |
| Pharmacokinetics of Zolbetuximab (Serum) <sup>16</sup> | X | | | | | |
| Antidrug-Antibodies (ADA) for Immunogenicity <sup>17</sup> | X | | | | | |
| Post-progression Tumor Sample (optional) <sup>18</sup> | | | | X | | |
| Concomitant Medication <sup>19</sup> | X | | · | X | X | $X^{21}$ |
| AE/SAE <sup>20</sup> | X | | | X | X | $X^{21}$ |

ADA: antidrug antibody; AE: adverse event; βhCG: beta human chorionic gonadotropin; C1D1: Cycle 1 Day 1; CAPOX: capecitabine and oxaliplatin; CT: computerized tomography; ECG: electrocardiogram; ECOG: Eastern Cooperative Oncology Group; ICF: informed consent form: INR: international normalized ratio; IRC: independent review committee; IRR: infusion-related reaction; IRT: interactive response technology; IV: intravenous; MRI: magnetic resonance imaging; OS: overall survival; PD: progressive disease; PFS: progression free survival; PFS2: progression free survival following subsequent anticancer treatment; PT: prothrombin time; PTT: partial thromboplastin time; RECIST: Response Evaluation Criteria In Solid Tumors; SAE: serious adverse event; T4: thyroxine; TSH: thyroid stimulating hormone

†Local and/or regional protocols or precautions for COVID-19 management should be followed as applicable.

1. <u>Antiemetic Pretreatment</u>: Antiemetic premedication (prophylactic antiemetics) should be administered prior to each study treatment. IV antiemetic premedication should be initiated prior to treatment, or oral antiemetic premedication should be initiated at a <u>minimum of 30 minutes</u> prior to treatment. Antiemetic premedication should be given according to institutional standard of care, published guidelines and the respective product package insert(s). For further details, see [Section 5.1.1.2 Antiemetics].


2. <u>Zolbetuximab/placebo</u> will be administered as a minimum 2-hour intravenous infusion every 3 weeks starting on C1D1. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information. Zolbetuximab/placebo should be administered prior to CAPOX. For further details, see [Section 5.1.1.1 Zolbetuximab/Placebo].

- 3. Post-infusion Observation Period: Following the first dose of zolbetuximab/placebo on C1D1, the subject must be observed for 2 hours post zolbetuximab/placebo infusion. The post-infusion observation period can be conducted during the CAPOX administration. If any ≥ grade 2 AEs are observed during infusion or during the post-infusion observation period, subsequent zolbetuximab/placebo infusion times should be extended and subjects should continue to be observed for 2 hours post zolbetuximab/placebo infusion. If the subject does not develop any grade ≥ 2 AEs, the subject should be observed for 1 hour post-infusion for their subsequent zolbetuximab/placebo infusions. The subject should be instructed to notify site personnel if they develop any AEs during this observation time period. In the event of an IRR with features of anaphylaxis (regardless of grade) or grade 3 or 4 IRR, blood samples for cytokine/chemokine panel and serum total tryptase level (levels typically peak within 3 hours after the onset of symptoms) should be collected once the subject has stabilized, for shipment to the central laboratory. See Observation Period following zolbetuximab/placebo infusion [Section 5.4.2] for further details.
- 4. <u>CAPOX</u> is a combination of oxaliplatin intravenous infusion and capecitabine tablets and will be administered starting at C1D1 for up to 8 treatments. See [Section 5.1.1.3].
- 5. <u>Physical Exam</u>: should include height (at Screening only), <u>weight</u> and <u>ECOG performance status</u>. For all cycles, the physical examination, weight and ECOG performance status assessments can be completed up to 48 hours prior to zolbetuximab/placebo administration. Targeted (symptom driven) physical exams should be conducted every 3 weeks on day 1 of each cycle. For further details, see [Section 5.4.4 Physical Examination]
- 6. <u>Vital signs</u> (pulse, blood pressure, temperature) should be taken during every visit at the following time points (see [Section 5.4.1 Vital Signs]):
  - o Predose at every visit
  - o If the subject did not develop any ≥ grade 2 AEs during the C1D1 zolbetuximab/placebo infusion or Post-infusion Observation Period, the site may do the following for subsequent zolbetuximab/placebo infusions:
    - The post-infusion observation period can be 1 hour for subsequent visits after C1D1
    - The vital signs can be assessed every 60 minutes for subsequent visits after C1D1
  - Every 60 (±10) minutes post zolbetuximab/placebo infusion during the Post-infusion Observation Period (for 1 or 2 hours. See footnote 7)
  - o Unscheduled if clinically indicated
- 7. <u>ECGs</u>: ECGs will be locally assessed. When collected on the same day, ECG should be collected prior to pharmacokinetic samples. For further details, see [Section 5.4.5 Electrocardiogram]. A single ECG will be performed at the following time points:
  - o Up to 48 hours prior to every oxaliplatin infusion (before any antiemetic treatment administration)
  - o Up to 6 hours following completion of every oxaliplatin infusion
  - o Zolbetuximab/placebo Discontinuation Visit (if clinically indicated)
  - o Zolbetuximab/placebo 30-day Follow-up Visit (if clinically indicated)
  - o If clinically indicated or per local requirements


8. Imaging Assessments: Effective with implementation of Protocol Version 7.0 (Substantial Amendment 6), radiologic imaging will be evaluated locally. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), radiographic imaging was evaluated centrally by IRC [Table 1]. Radiologic imaging will be evaluated every 9 weeks (± 7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (± 7 days) thereafter until subject develops radiological disease progression per RECIST 1.1 confirmed locally or by IRC or starts other systemic anticancer treatment, whichever comes earlier. Imaging schedule should be maintained regardless of treatment delay. Imaging will include CT scans with contrast of the thorax, abdomen, and pelvis. If CT scan with contrast is medically not feasible, MRI may be used for imaging. Bone scans (or focal X-ray) or brain imaging should be performed if metastatic disease in bone or brain is suspected, respectively. The same mode of imaging should be utilized throughout the study unless medical necessity requires a change. See [Section 5.3 Efficacy Assessments]. Refer to Imaging Acquisition Guidelines for further detail on scan modality and contrast options.

- 9. <u>Laboratory Assessments</u>: See [Section 5.4.3 Laboratory Assessments] for list of laboratory assessments. Laboratory tests must be sent to the local laboratory for analysis. For screening/eligibility laboratory assessments, see footnote number 1.
  - <u>Laboratory test results (local) will be reviewed by the investigator prior to any study treatment</u>. Clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician.
  - Local labs may be collected up to 48 hours prior to study treatment.
  - Holidays and weekends should be taken into account when scheduling these sample collections.
  - Additional assessments may be done centrally or locally to monitor AEs or as clinically indicated.
- 10. <u>Coagulation</u> (PT, PTT and INR): Coagulation tests should be done during study treatment period if clinically indicated. Ongoing evaluation should be continued for subjects who are receiving therapeutic anticoagulation according to local standard of care. See [Section 5.4.3 Laboratory Assessments].
- 11. <u>Serum Pregnancy Test</u>: Serum pregnancy tests will be collected for female subjects of childbearing potential only. Serum pregnancy tests collected at Screening, during study treatment period and if clinically indicated or per local requirements. Serum pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration.
- 12. <u>Urine Pregnancy Test</u>: Urine pregnancy tests will be collected for female subjects of childbearing potential only. Local urine pregnancy tests to be performed during the treatment period every 3 weeks on day 1 of each cycle and at the zolbetuximab/placebo Study Treatment Discontinuation and 30-day Safety Follow-up Visits. Urine pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. Additional urine pregnancy testing for up to 9 months after the final study treatment administration may be conducted based on local requirements.
- 13. Study Treatment Discontinuation Visit (End of Study Treatment): The Study Treatment Discontinuation Visit will take place ≤ 7 days following the decision to discontinue study treatment (zolbetuximab/placebo and CAPOX [both components]). If zolbetuximab/placebo and CAPOX (both components) are discontinued on a different day, subjects will have separate Study Treatment Discontinuation Visits following each treatment's discontinuation. Laboratory tests must be sent to the local laboratory for analysis. A combined visit can be completed if zolbetuximab/placebo are discontinued on the same day. The Study Treatment Discontinuation Visit is not required if the participant has transitioned to commercially available zolbetuximab and/or CAPOX. Safety reporting should continue as per post-marketing requirements in this case.
- 14. 30-day Safety Follow-up Visit: A 30-day Safety Follow-up Visit should occur 30 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 30-day Safety Follow-up Visit should occur 30 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day. The 30-Day Safety Follow-up visit is not required if the participant has transitioned to commercially available zolbetuximab and/or CAPOX. Safety reporting should continue as per post-marketing requirements in this case.


15. <u>90-day Safety Follow-up Visits</u>: A 90-day Safety Follow-up Visit should occur 90 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 90-day Safety Follow-up Visit should occur 90 days after the last dose of CAPOX (both components) and may be conducted by phone. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day. The 90-Day Safety Follow-up visit is not required if the participant has transitioned to commercially available zolbetuximab and/or CAPOX. Safety reporting should continue as per post-marketing requirements in this case.

- 16. <u>Pharmacokinetics</u>: Serum samples for zolbetuximab/placebo will be taken at the below time points and sent to the central laboratory. The date and time of each blood sample collection will be recorded to the nearest minute.
  - o Predose on Day 1 of Cycles 9, 13 and 17
  - o Unscheduled pharmacokinetic blood samples may be taken at any time during the study to evaluate drug exposure following a safety event

Pharmacokinetic Sampling Window:

- o Predose: within 60 minutes prior to dosing
- o End of Infusion: within 10 minutes after the end of the infusion
- 17. ADA: Blood samples (Serum) for ADA will be taken at the below time points and sent to the central laboratory.
  - o Predose on Day 1 of Cycles 9, 13 and 17
  - ADA Sampling Window: Predose: within 60 minutes prior to dosing
- 18. Optional Post-Progression Tumor Sample: For subjects who signed a separate ICF, an optional post-progression tumor sample for exploratory biomarker analysis may be collected following local confirmation or IRC confirmation of disease progression and prior to initiation of subsequent anticancer therapy. Sample collection is optional and only collected as allowed per local policy. (UNIQUE TO CHINA: Optional post-progression tumor sample is not applicable for China.)
- 19. Concomitant medications will be collected from the time of full main informed consent through 90 days following the last dose of study treatment.
- 20. <u>AEs/SAEs</u>: AEs and SAEs (regardless of causality) will be collected from the time of full main informed consent through 90 days following the last dose of study treatment. See [Section 5.5.5 Reporting of Serious Adverse Events].
- 21. Collection by phone.

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

Table 12 Protocol Version 7.0 (Substantial Amendment 6) and Later: Alternate Schedule of Assessments in Response to a Crisis

| | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>13</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>14</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>15</sup> |
|---|---|---|---|---|---|
| | | | Stı<br>Dis | 30-I<br>Visi | 90-D<br>Visit |
| 1 | 2-14 | 15-21 | | | |
| X | | | | | |
| X | | | | | |
| X | | | | | |
| X | х | | | | |
| X | | | | | |
| X | | | _ | | |
| X | | X X | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | | | Critical T | imepoint† | | |
|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>13</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>14</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>15</sup> |
| Cycle Day | | 1 | 2-14 | 15-21 | | | |
| Vital Signs <sup>6</sup> | If a cycle is administered at a local facility for SoC regimen administration, SoC can be applied. Missed assessments at Study Treatment Discontinuation Visit and 30-Day Safety Follow-up visit are acceptable if there are no associated active AEs. Vital sign frequency during post observation period can be decreased. | х | | | | | |
| ECOG Performance Status <sup>5</sup> | Not required at Study Treatment Discontinuation visit; ECOG Performance Status may be assessed and captured via phone contact. | X | | | | | |
| 12-lead ECG <sup>7</sup> | ECGs allowed up to 4 days prior to treatment visits after C1D1 and can be done locally but must be reviewed prior to dosing; if dosing visits are conducted at local facility, SoC ECG monitoring would be acceptable; if capecitabine only is dispensed and ECG is not able to be performed, this is acceptable; Study Treatment Discontinuation Visit and 30-Day Safety Follow-up Visit required only if clinically indicated. | | indicated and/orequirements | or per local | | If clinically indicated | |
| Image Assessment <sup>8</sup> | At select visits, efficacy assessment using radiological examinations are required. Imaging assessment should be done locally. If investigational site read is not an option, the investigator should discuss the case with the local institution radiologist. The local site imaging report is required. | Every 9 w | eeks ±7 days f | | or the first 54 v | weeks and then | every 12 |
| Laboratory Tests | | | | | | | |
| Biochemistry <sup>9</sup> | Sample may be collected up to 4 days prior to treatment visit; collection of samples at local facility acceptable if results can be made available to investigative site. | X | | | X | X | |
| TSH and Free T49 | If this testing is unable to be performed, this is acceptable | If cl | inically indicat | ted | | | |
| Hematology <sup>9</sup> | Sample may be collected up to 4 days prior to treatment visit; collection of samples at local facility acceptable if results can be made available to investigative site. | X | | | X | X | |
| Table continued on next page | | | | | | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

| | | Critical Timepoint† | | | | | |
|---|---|---|---|---|---|---|---|
| Critical Assessment†† | Alternate Approach(es) | Cycle 9+ | | Study Treatment<br>Discontinuation Visit <sup>13</sup> | 30-Day Safety Follow-up<br>Visit(s) <sup>14</sup> | 90-Day Safety Follow-up<br>Visit(s) <sup>15</sup> | |
| Cycle Day | | 1 | 2-14 | 15-21 | | | |
| Coagulation Parameters (PT, PTT and INR) <sup>10</sup> | None as protocol allows SoC if clinically indicated. If the subject is not on a concomitant medication that affects these parameters, it is acceptable if these are not done. | If clinically indicated | | | | | |
| Urinalysis <sup>9</sup> | Sample may be collected up to 4 days prior to treatment visit; collection at local facility. | X | | | | | |
| Serum Pregnancy Test <sup>11</sup> | Collection at local facility. | If clinically indicated and/or per local requirements | | | | | |
| Urine Pregnancy Test <sup>12</sup> | Collection at local facility. | X | | | X | X | |
| Sampling | | | | | | | |
| Pharmacokinetics of Zolbetuximab (Serum) <sup>16</sup> | Samples at predose/End of Infusion will be collected if subject receives treatment at investigative site. If central lab cannot receive samples, samples can be stored at sites in -70°C freezer until shipping is accepted again. Follow-up samples will be collected if subject visits the investigative site. | X | | | | | |
| Antidrug-Antibodies (ADA) for<br>Immunogenicity <sup>17</sup> | If subject is dosed or visits investigative site, ADA samples should be collected. Samples cannot be collected at local facility. Sample collection prioritized if clinically indicated. If central lab cannot receive samples, samples can be stored at sites in -70°C freezer until shipping is accepted again. | X | | | | | |
| Post-progression Tumor Sample (optional) <sup>18</sup> | In general, biomarker samples are collected on zolbetuximab treatment days and do not require a unique visit to the study site. If samples can be collected but central labs cannot receive samples, samples can be stored at sites until shipping is accepted again. | | | | Х | | |
| Concomitant Medication <sup>19</sup> | Remote/Virtual/Telemedicine "Visits" allowed for non-dosing visits. Please refer to protocol schedule of assessments. | X | | | X | X | $X^{21}$ |
| AE/SAE <sup>20</sup> | Remote/Virtual/Telemedicine "Visits" allowed for non-dosing visits. Please refer to protocol schedule of assessments. | X | | | X | X | $X^{21}$ |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


ADA: antidrug antibody; AE: adverse event; βhCG: beta human chorionic gonadotropin; C1D1: Cycle 1 Day 1; CAPOX: capecitabine and oxaliplatin; CT: computerized tomography; ECG: electrocardiogram; ECOG: Eastern Cooperative Oncology Group; ICF: informed consent form: INR: international normalized ratio; IRC: independent review committee; IRR: infusion-related reaction; IRT: interactive response technology; IV: intravenous; MRI: magnetic resonance imaging; OS: overall survival; PD: progressive disease; PFS: progression free survival; PFS2: progression free survival following subsequent anticancer treatment; PT: prothrombin time; PTT: partial thromboplastin time; RECIST: Response Evaluation Criteria In Solid Tumors; SAE: serious adverse event; SoC: standard of care; T4: thyroxine; TSH: thyroid stimulating hormone

†In case subjects are unable to be evaluated in person on Day 1 of each cycle, the site will contact the subject by phone for a safety assessment at the time the next visit would be due. ††Additional non-protocol-specific testing may be required per local regulations. Local and/or regional protocols or precautions for COVID-19 management should be followed as applicable.

\*+7 calendar day visit window does not apply to C1D1.

- 1. <u>Antiemetic Pretreatment</u>: Antiemetic premedication (prophylactic antiemetics) should be administered prior to each study treatment. IV antiemetic premedication should be initiated prior to treatment, or oral antiemetic premedication should be initiated at a <u>minimum of 30 minutes</u> prior to treatment. Antiemetic premedication should be given according to institutional standard of care, published guidelines and the respective product package insert(s). For further details, see [Section 5.1.1.2 Antiemetics].
- 2. <u>Zolbetuximab/placebo</u> will be administered as a minimum 2-hour intravenous infusion every 3 weeks starting on C1D1. Please refer to Pharmacy Manual and Infusion Guidelines for more detailed information. Zolbetuximab/placebo should be administered prior to CAPOX. For further details, see [Section 5.1.1.1 Zolbetuximab/Placebo].
- 3. Post-infusion Observation Period: Following the first dose of zolbetuximab/placebo on C1D1, the subject must be observed for 2 hours post-zolbetuximab/placebo infusion. The post-infusion observation period can be conducted during the CAPOX administration. If any ≥ grade 2 AEs are observed during infusion or during the post-infusion observation period, subsequent zolbetuximab/placebo infusion times should be extended and subjects should continue to be observed for 2 hours post zolbetuximab/placebo infusion. If the subject does not develop any grade ≥ 2 AEs, the subject should be observed for 1 hour post-infusion for their subsequent zolbetuximab/placebo infusions. The subject should be instructed to notify site personnel if they develop any AEs during this observation time period. In the event of an IRR with features of anaphylaxis (regardless of grade) or grade 3 or 4 IRR, blood samples for cytokine/chemokine panel and serum total tryptase level (levels typically peak within 3 hours after the onset of symptoms) should be collected once the subject has stabilized. See Observation Period following zolbetuximab/placebo infusion [Section 5.4.2] for further details.
- 4. <u>CAPOX</u> is a combination of oxaliplatin intravenous infusion and capecitabine tablets and will be administered starting at C1D1 for up to 8 treatments. See [Section 5.1.1.3].
- 5. <u>Physical Exam</u>: should include height (at Screening only), <u>weight</u> and <u>ECOG performance status</u>. A full physical exam is required at Screening. The physical exam only needs to be repeated on C1D1 if clinically significant changes from screening are observed (in the opinion of the investigator). For all cycles, the physical examination, weight and ECOG performance status assessments can be completed up to 48 hours prior to zolbetuximab/placebo administration. Targeted (symptom driven) physical exams should be conducted every 3 weeks on day 1 of each cycle. For further details, see [Section 5.4.4 Physical Examination]
- 6. Vital signs (pulse, blood pressure, temperature) should be taken during every visit at the following time points (see [Section 5.4.1 Vital Signs]):
  - o Predose at every visit
  - o C1D1: Every 30 (±10) minutes during zolbetuximab/placebo infusion
  - o If the subject did not develop any ≥ grade 2 AEs during the C1D1 zolbetuximab/placebo infusion or Post-infusion Observation Period, the site may do the following for subsequent zolbetuximab/placebo infusions:
    - The post-infusion observation period can be 1 hour for subsequent visits after C1D1
    - The vital signs can be assessed every 60 minutes for subsequent visits after C1D1
  - o Every 60 (±10) minutes post zolbetuximab/placebo infusion during the Post-infusion Observation Period (for 1 or 2 hours. See footnote 7)
  - Unscheduled if clinically indicated

Footnotes continued on next page

06 Dec 2024 Astellas 


7. <u>ECGs</u>: ECGs will be locally assessed. When collected on the same day, ECG should be collected prior to pharmacokinetic samples. For further details, see [Section 5.4.5 Electrocardiogram]. A single ECG will be performed at the following time points:

- o Screening
- o Up to 48 hours prior to every oxaliplatin infusion (before any antiemetic treatment administration)
- o Up to 6 hours following completion of every oxaliplatin infusion
- o Zolbetuximab/placebo Discontinuation Visit (if clinically indicated)
- o Zolbetuximab/placebo 30-day Follow-up Visit (if clinically indicated)
- o If clinically indicated or per local requirements
- 8. <u>Imaging Assessments</u>: Effective with implementation of Protocol Version 7.0 (Substantial Amendment 5), radiologic imaging will be evaluated locally. Under Protocol Version 6.1 or earlier (e.g., Original Protocol Version 1 through 6.1), radiologic imaging was evaluated centrally by IRC [Table 1]. Radiologic imaging will be every 9 weeks (± 7 days) counting from C1D1 for the first 54 weeks and then every 12 weeks (± 7 days) thereafter until subject develops radiological disease progression per RECIST 1.1 by local or IRC or starts other systemic anticancer treatment, whichever comes earlier. Imaging schedule should be maintained regardless of treatment delay. Imaging will include CT scans with contrast of the thorax, abdomen, and pelvis. If CT scan with contrast is medically not feasible, MRI may be used for imaging. Bone scans (or focal X-ray) or brain imaging should be performed if metastatic disease in bone or brain is suspected, respectively. The same mode of imaging should be utilized throughout the study unless medical necessity requires a change. See [Section 5.3 Efficacy Assessments]. Refer to Imaging Acquisition Guidelines for further detail on scan modality and contrast options.
- 9. <u>Laboratory Assessments</u>: See [Section 5.4.3 Laboratory Assessments] for list of laboratory assessments. Laboratory tests must be sent to the local laboratory for analysis. For screening/eligibility laboratory assessments, see footnote number 1.
  - <u>Laboratory test results (local) will be reviewed by the investigator prior to any study treatment</u>. Clinical significance of out-of-range laboratory findings is to be determined and documented by the investigator/sub-investigator who is a qualified physician.
  - Local labs may be collected up to 48 hours prior to study treatment.
  - Holidays and weekends should be taken into account when scheduling these blood draws.
  - Additional assessments may be done locally to monitor AEs or as clinically indicated.
- 10. <u>Coagulation</u> (PT, PTT and INR): Coagulation tests should be done at Screening and during study treatment period if clinically indicated. Local or central lab results may be used to confirm eligibility. Ongoing evaluation should be continued for subjects who are receiving therapeutic anticoagulation according to local standard of care. See [Section 5.4.3 Laboratory Assessments].
- 11. <u>Serum Pregnancy Test</u>: Serum pregnancy tests will be collected for female subjects of childbearing potential only. Serum pregnancy tests collected at Screening, during study treatment period and if clinically indicated or per local requirements. Serum pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. (Note: For Screening, subjects with elevated serum βHCG and a demonstrated non-pregnant status through additional testing are eligible.)


12. <u>Urine Pregnancy Test</u>: Urine pregnancy tests will be collected for female subjects of childbearing potential only. Local urine pregnancy tests to be performed during the treatment period every 3 weeks on day 1 of each cycle and at the zolbetuximab/placebo Study Treatment Discontinuation and 30-day Safety Follow-up Visits. Urine pregnancy test can be completed up to 48 hours prior to zolbetuximab/placebo administration. Additional urine pregnancy testing for up to 9 months after the final study treatment administration may be conducted based on local requirements.

- 13. Study Treatment Discontinuation Visit (End of Study Treatment): The Study Treatment Discontinuation Visit will take place ≤ 7 days following the decision to discontinue study treatment (zolbetuximab/placebo and CAPOX [both components]). If zolbetuximab/placebo and CAPOX (both components) are discontinued on a different day, subjects will have separate Study Treatment Discontinuation Visits following each treatment's discontinuation. A combined visit can be completed if zolbetuximab/placebo are discontinued on the same day. If necessary during a crisis, this visit can be completed remotely for safety assessments and the required laboratory samples should be collected as soon as the crisis permits. The Study Treatment Discontinuation Visit is not required if the participant has transitioned to commercially available zolbetuximab and/or CAPOX. Safety reporting should continue as per post-marketing requirements in this case.
- 14. 30-day Safety Follow-up Visit: A 30-day Safety Follow-up Visit should occur 30 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 30-day Safety Follow-up Visit should occur 30 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day. If necessary during a crisis, this visit can be completed remotely for safety assessments and the required laboratory samples should be collected as soon as the crisis permits. The 30-Day Safety Follow-up visit is not required if the participant has transitioned to commercially available zolbetuximab and/or CAPOX. Safety reporting should continue as per post-marketing requirements in this case.
- 15. <u>90-day Safety Follow-up Visits</u>: A 90-day Safety Follow-up Visit should occur 90 days after the last dose of zolbetuximab/placebo and will include the assessments as shown in the Schedule of Assessments above. A 90-day Safety Follow-up Visit should occur 90 days after the last dose of CAPOX (both components) and may be conducted by phone if the subject is unable to visit the site and will require contact for AE/SAE collection only. A combined visit can be completed if zolbetuximab/placebo and both components of CAPOX are discontinued on the same day. The 90-Day Safety Follow-up visit is not required if the participant has transitioned to commercially available zolbetuximab and/or CAPOX. Safety reporting should continue as per post-marketing requirements in this case.
- 16. <u>Pharmacokinetics</u>: Serum samples for zolbetuximab/placebo will be taken at the below time points and sent to the central laboratory. The date and time of each blood sample collection will be recorded to the nearest minute.
  - o Predose on Day 1 of Cycles 9, 13 and 17
  - o Unscheduled pharmacokinetic blood samples may be taken at any time during the study to evaluate drug exposure following a safety event

Pharmacokinetic Sampling Window:

- o Predose: within 60 minutes prior to dosing
- o End of Infusion: within 10 minutes after the end of the infusion
- 17. ADA: Blood samples (Serum) for ADA will be taken at the below time points and sent to the central laboratory.
  - o Predose on Day 1 of Cycles 9, 13 and 17
  - ADA Sampling Window: Predose: within 60 minutes prior to dosing
- 18. Optional Post-Progression Tumor Sample: For subjects who signed a separate ICF, an optional post-progression tumor sample for exploratory biomarker analysis may be collected following local or IRC confirmation of disease progression and prior to initiation of subsequent anticancer therapy. Sample collection is optional and only collected as allowed per local policy. (UNIQUE TO CHINA: Optional post-progression tumor sample is not applicable for China.)
- 19. Concomitant medications will be collected from the time of full main informed consent through 90 days following the last dose of study treatment.


- 20. <u>AEs/SAEs</u>: AEs and SAEs (regardless of causality) will be collected from the time of full main informed consent through 90 days following the last dose of study treatment. See [Section 5.5.5 Reporting of Serious Adverse Events].
- 21. Collection by phone.

**Sponsor: APGD**EUCT 2024-511648-16-00; EudraCT number 2018-000519-26

### 14 COORDINATING INVESTIGATOR'S SIGNATURE

A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus CAPOX Compared with Placebo Plus CAPOX as First-line Treatment of Subjects with Claudin (CLDN)18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma

ISN/Protocol 8951-CL-0302

**Version 8.0 Incorporating Substantial Amendment 7** 

06 Dec 2024

| I have read all pages of this clinical study protocol for which Astellas is the sponsor. I agree that it contains all the information required to conduct this study. Coordinating Investigator: | | |
|---|---|---|
| - | artment/affiliation, name of institution> | Date (DD Mmm YYYY) |
| Printed Name: | | |
| Address: | | |
| _ | | |

EUCT 2024-511648-16-00; EudraCT number 2018-000519-26


## 15 SPONSOR'S SIGNATURES

Required sponsor signatures as required by ICH GCP 4.5.1 are located in the first attachment.

| Attachment 1 | Electronic Sponsor Signatures |
|--------------|-------------------------------|
|--------------|-------------------------------|

Global Protocol Format V12.1